## FRED HUTCHINSON CANCER RESEARCH CENTER UNIVERSITY OF WASHINGTON SCHOOL OF MEDICINE SEATTLE CHILDREN'S

Current Version: 1/13/2016 Previous Version: 12/25/2014

Nonmyeloablative Conditioning with Pre- and Post-Transplant Rituximab followed by Related or Unrelated Donor Hematopoietic Cell Transplantation for Patients with Advanced Chronic Lymphocytic Leukemia: A Multi-Center Trial

Principal Investigators: Fred Hutchinson Cancer Research Center

| Mohamed L. Sorror, MD | orror, MD Associate Member, FHCRC, Associate Professor of | |
|---|---|---|
| | Medicine, UW | |
| David G. Maloney, MD | Member, FHCRC, Professor of Medicine, UW, | 667-5616 |
| Brenda M. Sandmaier, MD | Member, FHCRC, Professor of Medicine, UW, | 667-4961 |
| Stanley Riddell, MD | Member, FHCRC, Professor of Medicine, UW | 667-5249 |
| Mary E.D. Flowers, MD | Member, FHCRC, Professor of Medicine, UW | 667-5115 |
| Rainer Storb, MD | Member, FHCRC, Professor of Medicine UW | 667-4407 |

Statistician: Barry Storer, Ph.D., Affiliated Associate Professor of Biostatistics, UW,

Member, FHCRC (667-6533).

**Research Nurse:** Michelle Bouvier, RN (206) 667-6993, pager (206) 995-7658

Emergency (24 hour) Phone: (206) 598-8902 Fax: (206) 598-4034

| Additional Performance Sites Rigshospitalet | <u>Investigators</u> Niels Andersen, MD | Emergency Phone Numbers<br>+45 35 45 1134 |
|---|---|---|
| City Hlth & Sci - Torino | Benedetto Bruno, MD | 011-39-0339-1129064 |
| Veterans Affairs Puget Sound<br>Health Care System | Thomas Chauncey M.D., PhD | (206) 762-1010 for the oncologist on- |
| Mayo Clinic | William Hogan, MD | (507) 284-2511 |

#### 1. Introduction

Chronic lymphocytic leukemia (CLL) is a proliferative disorder of functionally abnormal lymphocytes. CLL is grouped with a spectrum of diseases known as low-grade lymphoproliferative disorders, CLL is the most common form of leukemia (25% of all cases) in western countries, and 95% of all cases are of B-cell phenotype. [1,2] Median age at diagnosis is 70 years, and only 10-15% of patients are younger than 50 years. [3] Despite some therapeutic progress, standard treatment is not curative for CLL. This, together with the advanced age of most patients and the relatively indolent course of the disease for some patients, makes symptom palliation a reasonable treatment goal. Therefore, chlorambucil or fludarabine are usually given for CLL patients who have anemia, thrombocytopenia, hepatosplenomegaly, and/or lymphadenopathy. Even though fludarabine was shown to result in higher response rates and longer progression free survival (PFS) compared to single-agent or combination chemotherapy, overall survival (OS) was not improved. [4-6] The use of fludarabine-rituximab or fludarabinecyclophosphamide-rituximab combinations may improve PFS and appears to improve OS based on historical controls[7,8]. Despite these advances, most patients who live long enough eventually fail fludarabine therapy, and about 20% of CLL patients have primary refractoriness (defined by failing to meet NCI Working Group Criteria for complete or partial responses: see Appendix H). Fludarabine-refractory CLL patients have a poor prognosis with median survival of 12 months. [9,10] Re-treatment with fludarabine or other nucleoside analogues such as cladribine or pentostatin, combination chemotherapy with or without fludarabine, and new biological agents such as Rituximab and Campath-1H has not demonstrably improved PFS. [9,11-17]

HCT using myeloablative conditioning has been increasingly used to treat young patients with CLL who have early stage disease and limited prior treatment. [18] Autologous high-dose HCT for CLL has shown long-term remissions and transplant-related mortality (TRM) of less than 10%. However, this treatment option was associated with high relapse rates reaching 56%[19]. Allogeneic HCT with high-dose conditioning has the theoretic advantage of graft-versus-leukemia (GVL) effects, and has resulted in tumor eradication and lower relapse rates compared to autologous HCT. However, TRM is higher than after autologous HCT by 20-40%. Unrelated-donor HCT has not been widely used for treatment of CLL because of the higher TRM as compared to related-donor HCT[20-22]. Hence, there has been no standard curative therapy for patients with fludarabine-refractory CLL. The Cancer Therapy Evaluation Program (CTEP) at the National Institute of Health (NIH) has recommended clinical trials for patients who have failed fludarabine treatment.

Allogeneic HCT after nonmyeloablative conditioning with fludarabine and low dose total body irradiation (TBI) and postgrafting immunosuppression with cyclosporine (CSP) and mycophenolate mofetil (MMF) was developed in an attempt to eradicate hematologic malignancies by GVL effects while avoiding morbidities and mortalities associated with myeloablative HCT. This approach using unrelated donor grafts has resulted in an encouraging OS and PFS rates of 67% at 2 years in 16 patients with fludarabine-refractory CLL. [23] Our updated results with longer follow-up show OS and PFS of 50% and 39%, respectively, at 5-years, which exceed any conventional salvage therapy for patients with fludarabine-refractory CLL. [24] However, disease relapse remain a cause of treatment failure with 5-years rate of 38%. NRM was the other cause of treatment failure (23% at 5-years), which resulted mainly from GVHD and infections. Outcomes were comparable between related and unrelated recipients.

The current protocol will attempt to better define safety and efficacy of allogeneic HCT after nonmyeloablative conditioning as salvage therapy for high-risk CLL patients. We propose to add the chimeric monoclonal anti-CD20 antibody Rituximab once immediately prior and three times in the weeks following the current non-myeloablative conditioning regimen. Our main goal is to reduce disease relapse. We will collect pharmacokinetic data to better define the optimal dosing of Rituximab and its impact on response. In addition, we will attempt to identify the recipient/donor pairs that benefit the most from Rituximab. This will be done by assessing recipient and donor polymorphisms of the FCγRIIIa receptor, which have been shown in some series to affect responsiveness to Rituximab.

#### 2. Background

#### A. Diagnosis, epidemiology, staging and prognosis of CLL

CLL is characterized by a progressive accumulation of atypical monoclonal lymphocytes in the bone marrow, peripheral blood and other organs. CLL is part of a spectrum of diseases grouped as low-grade lymphoproliferative disorders. It is the most common form of leukemia in western countries and constitute 25% of all cases. [1] The current annual incidence estimates vary from approximately 8100 to 12,500 new cases in the United States, [25,26] with annual CLL-related deaths of 4500. [27] The National Cancer Institute-sponsored Working Group (NCI-WG) on CLL had revised their guidelines for diagnosis of CLL. [28] All patients must meet all the following criteria to be diagnosed as CLL:

- An absolute peripheral lymphocytosis greater than 5,000 mature-appearing lymphocytes/μl.
- One or more B-cell markers (CD19, CD20, CD23) plus CD5 by flow cytometry.
- Mature lymphocytes with less than 55% cells being atypical lymphocytes, prolymphocytes or lymphoblasts.
- A normal to hypercellular bone marrow aspirate with ≥ 30% of the nucleated cells being of lymphoid origin.

Patients with CLL are staged utilizing either the Rai or Binet systems. Both systems discriminate CLL based on the sites of disease and/or degree of cytopenias induced by leukemic marrow replacement after exclusion of autoimmune etiologies. While, the Binet classification divides CLL patients into three stages as noted in, the Rai classification originally defined five stages of CLL (See Appendix R). However, in 1987, a modified Rai system was developed creating three prognostic risk categories (low, intermediate, and high risk) equivalent to the three stages of the Binet system. Factors predictive of poor prognosis in CLL patients include older age, male gender, a diffuse bone marrow pattern, a lymphocyte doubling time of less than one year, serum levels of B2-microglobulin greater than 4.0 mg/L, serum thymidine kinase levels greater than 7.0 U/L, and higher serum soluble CD23 levels. [29-32] Chromosomal analysis can also be used to assign risk. Patients with a normal karyotype, or isolated 13q14 deletions have a benign course. [33] However, 17p13 or 11q23 deletions (10-15% of patients) are associated with very poor prognosis. [34,35]

CLL has been categorized into two prognostic subsets based on the immunoglobulin variable-heavy chain (IgV<sub>H</sub>) mutational status. It was found that Binet stage A CLL patients with somatically unmutated IgV<sub>H</sub> genes have a median survival of 8 years compared to 25 years in patients with mutated genes. [36,37] Further, the two IgV<sub>H</sub> subsets are distinct and do not metamorphose from one into the other. Although surface CD38 expression was originally suggested as a surrogate assay for V gene mutations, [36] it appears that there is a 30% discordance between the assays. [38] Furthermore, CD38 expression was found to change in 25% of cases during the course of the disease, and therefore was not a useful prognostic indicator. [38] More recently, zeta-chain-associated protein 70 (ZAP-70), a kinase linked to T-cell receptor activation, was shown to be as excellent surrogate marker for the V gene mutational status with a sensitivity and specificity of 91% and 100%, respectively. [39] Unlike CD38, ZAP-70 surface expression does not change over time. [39] Given the difficulty in performing IgV<sub>H</sub> sequencing in a routine diagnostic laboratory, ZAP-70 detection with flow cytometry can be utilized efficiently in determining the prognosis of CLL patients or ensuring molecular complete remission (CR) after clinical trials.

#### **B.** Fludarabine-refractory CLL

Fludarabine has been considered frontline therapy for symptomatic CLL. Three large phase III trials of fludarabine in symptomatic untreated CLL patients have shown a higher response rate with prolongation of PFS compared to chlorambucil or combination chemotherapy. [5,6,40] There was no survival advantage in any of these studies likely due to crossover to fludarabine in the other arms. All surviving eventually failed fludarabine therapy, while approximately 20% of patients were refractory to primary therapy. Patients with fludarabine-refractory CLL have a very poor prognosis with a median survival of one year and less than 5% have responded to retreatment with single-agent fludarabine. [9,41,42] These patients have had limited treatment options, and most investigators encourage their participation in clinical trials. [43-45] Several

clinical trials have been performed on patients with fludarabine-refractory CLL using other nucleoside analogs like cladribine or pentostatin, combination chemotherapy, and monoclonal antibodies such as Rituximab or Campath-1H with limited improvement in disease-free survival and OS. In the current protocol, fludarabine-refractory CLL will be defined by failure to meet NCI-WG Criteria (Appendix H) for complete or partial response after a regimen containing fludarabine (or other nucleoside analogue) or relapse /progression within 12 months after completion of a regimen containing fludarabine (or other nucleoside analogue such as pentostatin or cladribine).

The best clinical outcomes for patients with fludarabinerefractory CLL were associated with the use of Campath-



**Figure 1.** OS curve for patients with fludarabine-refractory CLL treated with Campath-1H.

1H. [14,17,46] Campath-1H is a humanized anti-CD52 monoclonal antibody that has been approved by the United States Food and Drug administration for treatment of fludarabine-refractory CLL (reviewed in [47]). Ninety-three CLL patients who were refractory to fludarabine were given Campath-1H in a prospective phase II trial involving 21 centers worldwide. The overall response rate was 33% however, only 2% achieved CR. Median time to progression was

4.7 months and median survival was 16 months. OS was approximately 45% at 18 months (Figure 1). [14] Since this was the best reported outcome for salvage therapy for fludarabine-refractory CLL patients, we will use this outcome as the gold standard for comparison in the current protocol. Campath-1H caused substantial toxicities that included infusion-related fevers and chills, infections in 55% of patients (25 of 93 patients had grade III-IV infections), and hematological toxicity (21% had grade IV neutropenia). Updated results in 152 fludarabine-refractory CLL patients who received CAMPATH-H1 showed 42.5% overall response rate and CR rate of 5%.[17] This update included 29 patients with T-cell prolymphocytic leukemia (T-PLL) who showed lower overall response rate of 24%, but 14% were in CR. CMV disease occurred in 4 patients and 5 patients died from infections. Duration of response and OS rate were not available in this update.

Rituximab which is a chimeric human-mouse monoclonal antibody directed against the CD20 antigen present on B cells, has been investigated in the treatment of fludarabine-refractory CLL. A trial of thrice-weekly dosing of rituximab in 33 patients with CLL/small lymphocytic lymphoma (SLL), 52% of whom were fludarabine-refractory, the overall response rate among the fludarabine-refractory subset was 41% with a median response duration of 6 months. [11] A dose-escalation study of 40 patients with CLL showed that only 20% of fludarabine-refractory patients achieved PR and none CR. In a multiple parameter analysis, sensitivity to fludarabine was the only factor that correlated significantly with response to rituximab[12], a finding that reflects the limited activity of rituximab as a single agent for treating fludarabine-refractory CLL patients.

Combination chemotherapy with nucleoside analogs has not resulted in better outcomes than that of Campath-1H. Twenty-eight patients with fludarabine-refractory CLL were treated with a combination of cyclophosphamide and fludarabine[9]. Overall response rate was 39% with 3% of patients achieving CR. Median survival was 12 months with OS rate of 30% at 18 months. Thirteen patients with fludarabine-refractory CLL or SLL were treated with pentostatin plus cyclophosphamide resulting in an overall response rate of 77% with only one patient achieving CR, but responses were transient and median survival was only 16 months[15]. Cladribine has shown modest clinical activity and considerable toxicity. In one study, cladribine was given alone to treat 28 fludarabine-refractory CLL patients who had modest fludarabine or chemotherapy exposure and lacked pre-treatment neutropenia and thrombocytopenia. Despite this selection, Overall response rate was 32% without achieving CR with median PFS of 9 months. Grades III-IV toxicities were frequent and included infections (43%), neutropenia (75%), and thrombocytopenia (68%)[13]. Another trial explored a combination of cladribine and cyclophosphamide in 16 purine analog-refractory patients. The overall response rate was 25% and only one patient achieved CR. Toxicities were significant with myelosuppression being the dose limiting toxicity[16]. A combination of fludarabine, cyclophosphamide, and rituximab was used to treat 102 CLL patients of whom 27 were refractory to fludarabine[48]. Overall response rate among the fludarabine-refractory patients was 59% with CR rate of 7%. Survival data were not reported in this study

#### C. Autologous HCT for CLL

Autologous HCT has been offered only to selected groups of patients with CLL. The main criteria of eligibility for autologous HCT were documented chemosensitivity, minimal tumor burden (typically requiring several cycles of cytoreductive chemotherapy), and successful collection of enough hematopoietic progenitor cells. Best results have been achieved in patients undergoing autologous HCT earlier in their disease course and in those with fewer previous treatments or relapses. [49] Concerns about studies investigating autologous HCT for CLL include 1) the limited applicability due to the judicious selection of patients likely to benefit from the approach, 2) the high probability of disease relapse, and 3) the long-term risk of treatmentrelated secondary malignancies (reviewed in[50]). Failure to respond to pretransplant debulking chemotherapy has been one of the difficulties with autologous HCT. [51] In a series of 20 CLL patients, 10 patients did not meet the eligibility criteria either because of chemotherapy resistance (n=5, 4 died from progression), mortality from chemotherapy complications (n=2), or failure to mobilize adequate numbers of C34+cells (n=3). [52] Others have described poor hematopoietic cell collection due to advanced disease stage[49,53], or from prior marrow toxic chemotherapy including fludarabine and chlorambucil[54,55]. Available purging methods were found to either have no impact on survival[56] or increase the risk of life threatening infections[57], thereby causing morbidity and mortality[58].

Two large studies using autologous HCT for CLL, one from the European Group for Blood and Marrow Transplantation (EBMT) and one from the International Project for CLL are summarized in Table 1.

Table 1. Autologous HCT for CLL

| | EBMT[59]<br>(n=482) | International project for CLL[19] (n=124) |
|---|---|---|
| Age, median (range), years | 50 (22-66) | 49 (22-64) |
| Median interval from diagnosis to HCT (range), months | 26 (4-215) | 36 (5-218) |
| Prior regimens | 50% received <3 regimens | * |
| Prior fludarabine exposure | 26% | * |
| Chemo-sensitive disease at time of HCT | 85% (CR=31%) | 73% |
| Overall disease response | (n=239) 87% (CR=78%) | * |
| TRM | 11% at 3-years | 6% at 3 months |
| Relapse | 41% at 3-years | 58% at 5 years |
| DFS | * | 32% at 5 years |
| OS | 79% at 3-years, no plateau | 63% at 5 years |
| Factors predicting better outcome | Early HCT (<36 months<br>from diagnosis), low number<br>of prior regimens, and being<br>in CR at HCT | Early stage (Rai 0), short<br>interval between diagnosis<br>and HCT (<36 months0, low<br>marrow involvement, and <1<br>prior regimens |

#### \* Not reported

The German CLL Study group treated 65 patients, median age of 49 years, with TBI/cyclophosphamide followed by transplantation of immunomagnetically purged autologous stem cells[60]. Median interval from diagnosis to HCT was 14 months, and 94% of patients were chemotherapy naïve. Protocol failures before HCT occurred in 25% of patients either because they were not in remission (n=7), had poor mobilization (n=3), and/or protocol violations (n=4). One-year DFS was 95% by clinical and 69% by molecular criteria. The same authors have shown that persistence of the leukemic clone was found among 24 of 30 studied patients (80%) by sensitive Taqman CDR3 amplification for clone-specific primers {Dreger P, von Neuhoff, et al. 2000 23081 /id}. The German CLL Study concluded that autologous HCT does not appear to cure CLL even if performed early.

The Fred Hutchinson Cancer Research Center (FHCRC) has enrolled 7 patients under protocol 962 for autologous HCT. All had advanced stage CLL and had failed primary therapy. Their median age was 57 years. Only 5 patients were able to receive their HCT. Two patients died after HCT, one from respiratory failure secondary to acute pneumonitis with pseudomonas septicemia 4 months after HCT and the other after receiving a second HCT for secondary AML 39 months after the initial HCT. Three patients are alive, 2 of whom have relapsed 50 and 52 months after HCT, and one of whom developed Hodgkin's disease 69 months after HCT.

In summary, autologous HCT has remained restricted to younger patients without heavy prior chemotherapy regimens and with early stage chemo-responsive disease with fewer numbers of prior regimens. Although autologous HCT resulted in relatively low TRM, has not been shown to eradicate CLL on the molecular level. Therefore, patients had remained at risk of relapse, and there has been no plateau in DFS or OS. Autologous HCT has never been studied in patients with fludarabine-refractory CLL.

#### D. Allogeneic HCT for CLL

Allogeneic HCT for CLL has been characterized by high TRM and low relapse incidence. The risk for TRM has been higher for older patients and those who have received unrelated donor grafts. Most reported studies using myeloablative allogeneic HCT for CLL focused on younger patients with good performance status and limited numbers of preceding chemotherapy regimens.

Despite the low relapse rate, survival after allo-HCT has been lower than after autologous HCT mainly because of high TRM up to 50% even in experienced centers[61]. The majority of allotransplants have used related donors, and the experience with unrelated donors is limited (reviewed in [62]).

Table 2 summarizes data reported from 4 large studies investigating the role of allogeneic myeloablative HCT from related or unrelated donor for treatment of CLL.

Table 2. Allogeneic myeloablative HCT for CLL

| Tuote 2. Timogenere | International | Nebraska and | EDMT[50] | CLL working |
|---|---|---|---|---|
| | | | EBMT[59] | CLL working |
| | project for | Tennessee[63] | (n=209) | group-NMDP[64] |
| | CLL[19] | (n=23) | | (n=40) |
| | (n=48) | | | |
| Donor | | | | |
| Related | 100% | 87% | 96% | 0% |
| Unrelated | 0% | 13% | 4% | 100% |
| Age, Median | 43 (28-60) | 46 (29-60) | 47 (22-64) | 44 (26-57) |
| (range), years | | | | |
| Interval between | 26 (5-148) | 19 (4-160) | 45 (5-198) | 45 (8-121) |
| diagnosis and | | | | |
| HCT, median | | | | |
| (range), months | | | | |
| Number of | * | Median (range): | 73% received | Median (range): |
| chemotherapy | | 2 (1-6) | <3 regimens | 3 (0-5) |
| regimens | | = (1 0) | 5 1 5 5 111 5 115 | |
| Chemotherapy | 57% refractory | 61% refractory | 56% chemo- | 50% chemo- |
| sensitivity | 3770 Terractory | 0170 Terractory | responsive | refractory |
| Fludarabine | * | 65% received | 21% received | |
| | · | | | 80% received prior |
| exposure | * | prior FLU | prior FLU | FLU |
| Type of | ক | 70% VP/CY/TBI | 64% TBI-based | 92% TBI-based |
| conditioning | | and 26% CY/TBI | | **** |
| Acute GVHD | * | II-IV=52% | II-IV=40% | III-IV=28% |
| Chronic GVHD | * | 68% | 40% | 35% extensive |
| Disease response | 67% CR | 87% CR | 78% CR | 64% CR |
| TRM | 31% at 3 | 35% | 40% at 3 years | * |
| | months | | | |
| Relapse | * | * | 25% at 3 years | 13% at 3 years |
| DFS | 50% at 3 years | 61% at a median | * | 44% at 3 years |
| | j | follow up of 26 | | |
| | | months | | |
| OS | 56% at 3 years | * | 55% at 3 years | 41% at 3 years |
| Factors predicting | Phase of disease | * | Prior exposure | CR at HCT and |
| outcome | predicted | | to FLU is | Karnofsky score of |
| | survival while | | associated with | 90% predicted |
| | chemo- | | better outcome | better survival |
| | sensitivity | | | octor survivur |
| | predicted | | | |
| | relapse | | | |
| | rciapse | | | |

<sup>\*</sup>Not reported

Twenty-six patients with advanced stage and/or refractory CLL have undergone allogeneic stem cell transplantation from HLA-matched related donors at the FHCRC between 1980 and 1999. Patients were a median of 49 (range 14-59) years old. Twenty-one had B-cell CLL, one had T-

CLL and four patients did not undergo phenotyping. One patient had Richter's transformation and one patient evolved to prolymphocytic leukemia prior to transplant. Nineteen patients had received fludarabine with a median of 4 different regimens prior to HSCT. All patients had persistent disease at the time of transplant; 19 were Rai stage IV, 3 were stage III, 2 were stage II, and 2 were Rai stage 0. Patients received conditioning with busulfan (14 mg/kg) and CY (150 mg/kg) or CY/TBI (10-16 Gy). One patient underwent conditioning with etoposide 60 mg/kg, CY 100 mg/kg and 12 Gy TBI. Patients received HSCT from HLA-matched, sibling donors (n=22), syngeneic donors (n=3) or DRB1 mismatched sibling (n=1). Twenty-two patients engrafted. VOD occurred in 12 patients and renal failure occurred in 6 patients. Fourteen patients had GVHD  $\geq$  grade 2 requiring therapy. Thirteen patients (50%) achieved CR by bone marrow morphology, and six of seven evaluable patients achieved CR by flow cytometry. Eighteen patients (69%) have died at a median follow-up of 139 days (range 16-1906 days) from multiorgan failure (n=6), infection (n=5), GVHD + infection (n=2), Relapse (n=2), other/unknown (n=3). Eight patients survive at a median of 39 (range 9.5-101) months. The 5-year actuarial survival is 31% for all patients, and 56% for patients receiving conditioning with TBI after 1992 (n=14).

Five patients with advanced stage and/or refractory CLL (n=4) or CLL transformed to PLL (n=1) were given unrelated HCT between 1990 and 2000 at FHCRC. Median age was 46 (range 35-49) years and median interval between diagnosis and HCT was 22 (range 12-55) months. Patients were conditioned with cyclophosphamide/TBI (13.2Gy). After HCT, three patients had grade II and one grade III acute GVHD. Chronic extensive GVHD developed in 3 patients. Overall 4 patients died, one patient achieved CR, but died from multiorgan failure, one died from complications of a second HCT given for rejection of the first graft, one died from renal failure associated with progressive disease, and one from pneumonia with persistent disease. One patient who was in CR at time of HCT, is alive in CR at 1091 days after HCT.

In summary, conventional allogeneic HCT, while potentially curative as evidenced by the low relapse rates, was associated with a high TRM ranging from 31% to 50% (reviewed in [62]), even in patients less than 50 years of age. Unrelated donor HCT carries even higher risk of TRM with low survival advantage.

#### E. Reduced-dose regimens for allogeneic HCT

The use of nonmyeloablative regimens are appealing as treatment for patients with CLL for several reasons. First there are data that graft-versus-leukemia (GVL) effects appear to be effective in treating patients with CLL. The reduced toxicity of the nonablative conditioning was anticipated to result in lower TRM as compared to conventional conditioning. Third CLL patients are generally older than usual age where ablative HCT is offered.

The experience with reduced intensity transplants for CLL has been limited. Two large studies using reduced intensity conditioning and HCT for CLL, one from the Cooperative German Transplant Study Group[65] and one from the EBMT representing 29 European centers[66] are summarized in Table.3.

Table 3. Allogeneic reduced-intensity HCT for CLL

| Table 3. Allogeneic reduced-inten | | TD) (T) ( T) 566 |
|---|---|---|
| | Cooperative German | EBMT (n=77) [66] |
| | Transplant Study Group | |
| | (n=30) [65] | |
| Donor | | |
| Related | 50% | 82% |
| Unrelated | 50% | 18% |
| Age, Median (range), years | 50 (12-63) | 54 (30-66) |
| Interval between diagnosis and | 48 (12-510) | 49 (8-146) |
| HCT, median (range), months | | |
| Number of chemotherapy | 3 (0-8) | 3 (0-8) |
| regimens, median (range) | , , , | |
| Disease status at HCT | | |
| Responsive (CR/PR) | 46% | 65% |
| Refractory (SD/PD) | 46% | 35% |
| Fludarabine exposure | 33% fludarabine-refractory | 82% previous exposure, no |
| | | report on refractoriness |
| Type of conditioning | Fludarabine/ busulfan/ rabbit | 65% low dose TBI or |
| | anti-thymocyte globulin | cyclophosphamide-based |
| | | 35% fludarabine/busulphan |
| | | or high dose melphalan |
| | | combinations |
| Acute GVHD | | |
| Grade II-IV | 56% | 34% |
| Grade III-IV | 20% | 16% |
| Chronic GVHD | | |
| Limited | 54% | 58% limited+extensive |
| Extensive | 21% | |
| Disease response (CR+PR) | (40+53%) | (69%+22%) |
| TRM | | |
| All patients | 15% at 2 years | 18% at 1-year |
| Unrelated donor | 28% at 2 years | ĺ |
| recipients | ĺ | |
| Relapse | * | 31% at 2-years |
| PFS | 67% | 56% at 2-years |
| OS | 72% | 72% at 2-years |
| *N-4 1 | , = , \$ | , = , 0 at = j tazz |

<sup>\*</sup>Not reported

# **F. Our preliminary results of nonmyeloablative conditioning and allogeneic HCT for CLL** Based on preclinical studies in a canine model, [67] we developed a nonmyeloablative conditioning regimen for hematopoietic cell transplantation (HCT) for patients with hematological malignancies. The regimen was first used in patients receiving HCT from HLA-

SD indicates stable disease; and PD, progressive disease

matched related donors[68] and from January 2000, for patients given HCT from HLA-matched unrelated donors. [69,70]

In 2005, we reported our encouraging early results of allogeneic hematopoietic cell transplantation (HCT) after nonmyeloablative conditioning in 64 patients who had advanced chronic lymphocytic leukemia (CLL). Patients were given HCT from related (n = 44) or unrelated (n = 20) donors. Patients had multiple risk factors: median age was 56 years; median interval between diagnosis and HCT was 4.4 years; CCI scores of ≥1 for pretransplantation comorbidities were present in 48% of patients; chemotherapy resistance to pretransplantation salvage treatment was present in 53% of patients and untreated relapse occurred in 11% of patients; there was a median of four prior treatment regimens; and disease refractoriness to at least one regimen was present in all but two patients (97%). Thirty patients (47%) were refractory to one regimen, 23 patients (36%) were refractory to two regimens, and nine patients (14%) were refractory to ≥three regimens. Eighty-eight percent of patients were refractory to fludarabine, 25% of patients were refractory to rituximab, 30% of patients were refractory to alkylating agents, and 22% of patients were refractory to other miscellaneous regimens. In addition, patients had multiple adverse disease burden characteristics: bulky lymphadenopathy (lymph node

diameter  $\geq 5$  cm, 28%), splenomegaly (47%), CD5/CD9 coexpression of CD38 more than 30% (58%), beta<sub>2</sub>-microglobulin more than 2.5  $\mu$ g/mL (53%),  $\geq$ 50% marrow infiltration with CLL cells (52%), and unfavorable cytogenetics (39%). No significant differences in adverse disease burden characteristics were present between related and unrelated recipients. After HCT, Sixty-one of 64 patients had sustained engraftment, whereas three patients rejected their grafts. The incidences of grades 2, 3, and 4 acute and chronic graft-versus-host disease were 39%, 14%, 2%, and 50%, respectively. Three patients who underwent transplantation in complete remission (CR) remained in CR. The overall response rate among 61 patients with measurable disease was 67% (50% CR). whereas 5% had stable disease. All patients with morphologic CR who were tested by polymerase chain reaction (n = 11) achieved negative molecular results, and one of these patients subsequently experienced disease relapse. The 2-year incidence of relapse/progression was 26%, whereas the 2year relapse and nonrelapse mortalities were



Figure 2. Cumulative incidences of nonrelapse mortality (NRM), relapse-related mortality, overall survival (OS), and disease-free survival (DFS) for (A) related and (B) unrelated recipients.

18% and 22%, respectively. Two-year rates of overall and disease-free survivals were 60% and 52%, respectively. Unrelated HCT resulted in higher CR and lower relapse rates than related HCT. Two-year OS and DFS of related compared with unrelated recipients were 56% v 75% (P = .33) and 44% v 75% (P = .15), respectively (Figure 2).

Recently, Here, we have extended the follow-up to a median of 5 years and have included data on an additional 18 patients. Grafts were from related (n = 52) or unrelated (n = 30) donors. Complete remission (CR) and partial remission were achieved in 55% and 15% of patients,

respectively. Higher CR rates were noted after unrelated HCT (67% v 48%). The 5-year incidences of nonrelapse mortality (NRM), progression/relapse, overall survival, and progression-free survival were 23%, 38%, 50%, and 39%, respectively. Among 25 patients initially reported in CR, 8% relapsed and 8% died as a result of NRM, whereas 84% have remained alive and in CR. Among 14 responding patients who were tested and who had molecular eradication of their disease, two died as a result of NRM, two relapsed, and 10 have remained negative. The 5-year prevalence of patients alive after discontinuation of all immunosuppressive medications was 38% (35% for

Durelated Related Resolution of chronic GVHD Res

os

p = 0.57

**Figure 3.** CLL: OS based on donor type and resolution of GVHD following allogeneic HCT.

related and 44% for unrelated recipients, Figure 3); the median performance status in each group was 100% and 90%, respectively. Lymphadenopathy > or = 5 cm, but not cytogenetic abnormalities at HCT, predicted relapse. In a risk-stratification model, patients who had

lymphadenopathy less than 5 cm and no comorbidities had a 5-year OS of 71%.

Outcomes of patients with favorable (normal or 13q deletion) versus unfavorable (all others) cytogenetic abnormalities were comparable (Figure 4). Seven patients had 17p deletion, of whom 4 (57%) are alive and in CR, 1 died with NRM while in CR, and 2 died from relapse.

In summary, Nonmyeloablative HCT resulted in a median survival of 5 years for patients who had fludarabine-refractory CLL with sustained remissions and in the continued resolution of chronic graft-versushost disease in surviving patients. The approach appeared feasible with acceptable NRM, high rates of disease responses, and a good evidence of GVL effect. Outcomes of related and unrelated recipients were similar, providing the rationale to combine both grafts in this protocol. However, disease relapse remained as a cause of treatment failure with 5-years rate of 26%. NRM was the other cause of treatment failure, 24% at 5-years, and it resulted mainly from GVHD and its complications and infections. We thought to further improve our results by adding peri-transplant Rituximab with the main goal of more robust disease-



Figure 4. Comparable 5-year relapse and PFS rates among CLL patients with unfavorable (17p deletion, 11q deletion, trisomy 12, and complex) versus favorable (normal and 13q deletion) cytogenetic abnormalities following nonmyeloablative allogeneic HCT.

control and a secondary goal of limiting GVHD and its complications.

#### G. Update on results of CLL patients with poor prognosis

Recently, investigators from MD Anderson Cancer Center have presented at the American Society of Clinical Oncology 2007 Meeting results of 77 patients with CLL who have failed initial treatment with combination chemo-immunotherapy comprising fludarabine, cyclophosphamide, and rituximab (FCR). Ten of those patients have not required therapy while 67 patients received first salvage therapy with a variety of regimens. Overall response rate was 39% and CR rate was 17%. Median survival after the first salvage therapy was 30 months (28 deaths) and was shorter for patients with PR or refractory disease (10 months). Of interest, 13 patients who failed the first salvage therapy went to receive allogeneic HCT after reduced intensity regimens. Of those 13 patients, 3 died early, one relapsed, 2 in PR, and 7 in CR. Survival at 3 years is 76%. The authors concluded that patients who failed to obtain CR or nodular PR after FCR or first salvage therapy should be considered for allogeneic HCT. <sup>52</sup>

Alternatively, patients with advanced CLL and 17p deletion genomic feature have a very poor prognosis even after intensive chemotherapy. The hierarchical model of Dohner and colleagues identified the prevalence of this genomic aberration to be of 7%. Patients with 17p deletion had only 0.75 year treatment-free interval and 2.7 years median survival from time of diagnosis. Recently, investigators from Germany have shown that patients with 17 p deletion had statistically significantly shorter median PFS (11 versus 24 months, p=0.002) and median OS (15.9 months versus not reached, p<0.001) compared to patients without 17p deletion following fludarabine-based regimens (Figure 5). Similar findings were also reported by investigators of the US Intergroup Phase III Trial E2997, where patients with 17p deletion had median PFS of 0.9 years after initial therapy with fludarabine  $\pm$  cyclophosphamide. Further, investigators from MD Anderson Cancer Center have shown at the American Society of Hematology 2007 Meeting that 17p deletion  $\pm$ 0 other genomic aberrations was the strongest independent predictor for

shorter survivals and poor response to the combination FCR

as an initial therapy for CLL.<sup>56</sup>

Updated results suggest that patients who fail FCR combination chemotherapy at any time point and patients with "de novo" or acquired 17p deletion cytogenetic abnormality, who received induction chemotherapy should be enrolled in nonmyeloablative protocols.

### H. Peri-transplant Rituximab to improve early disease control and reduce relapse risk

The cell-surface antigen CD20 is a 297-amino acid transmembrane phosphoprotein that is expressed on more than 90% of mature B-cell leukemias and lymphomas. [71] Rituximab is a chimeric anti-CD20 monoclonal antibody, which has been shown to be active against CLL either as a

1.0 9 8 7 6 5 4 3 2 1.1 0.0 0 6 12 18 24 30 36 42 48 54 60 66 OS in Months

Figure 5. Kaplan-Meier survival for CLL patients (n=375) with versus without 17p deletion following initial treatment with fludarabine ± cyclophosphamide.

single agent[72]or in combination with chemotherapy. [73]. The proposed mechanisms for the cytotoxic action of rituximab include complement-dependent cytotoxicity, [71] antibody-

dependent cellular cytotoxicity, [71] and signaling-induced apoptosis [74,75] in addition to synergistic effects with chemotherapeutic agents [71] and radiation therapy. [76]

#### Theory:

The antitumor effects of NM HCT are substantial, but disease progression occurs in a substantial fraction of patients. In our earlier results with nonmyeloablative HCT for patients (n=64) with advanced CLL, we found that the median time to early progression was 3.3 months, while median time to the first sign of disease eradication, complete resolution of cytogenetic abnormalities, by GVL was 3 months. Patients with progressive disease frequently have a larger tumor burden prior to transplant and fail to develop T cell responses to CLL, suggesting that tumor antigens are not efficiently presented or reactive T cells are tolerized by the high tumor burden. Based on these findings, we could hypothesize that improvement of disease control could be achieved by 1) additional treatment in the early few weeks after HCT and 2) earlier and/or stronger generation of GVL effects. Rituximab given days before and after HCT could hypothetically meet these two objectives. Rituximab through antibody-dependent cytotoxicity could prevent disease progression in the early interval after HCT[71]. Further, investigators found that anti-CD20 antibodies, by induction of apoptosis, could promote uptake and cross presentation of cell-derived peptides by antigen-presenting dendritic cells. [77] In these lines, Rituximab could allow cross-priming and generation of specific donor-derived cytotoxic T cells resulting in earlier "switch-on" of GVL effects. [78,79]

#### *Tolerability:*

Rituximab, alone or in combination with various chemotherapy regimens, was generally well tolerated in clinical trials in patients with advanced-stage indolent or aggressive B-cell NHL or B-cell CLL. The most common types of adverse events in these trials were infusion-related reactions, hematological adverse events and infections. Infusion-related reactions that occur in the majority of patients, most within 2 hours of the first infusion, are generally mild to moderate flu-like symptoms that usually resolve upon slowing or stopping the infusion, and become less frequent with subsequent infusions. Severe (grade 3/4) reactions, including severe cytokine release syndrome, occur in 10% of patients and may also require supportive care (e.g. analgesic, antihistamine, oxygen, intravenous fluids, bronchodilators, vasopressors and/or corticosteroids). The true incidence of rituximab-related infections has not been determined, but nonrandomized trial data showed a 31% overall (19% bacterial, 10% viral) and 2-4% incidence of severe infectious events. (Biogen Idec Inc., Genentech Inc. Rituxan® (Rituximab): prescribing information. 2006 Feb 28; and Roche Registration Limited. MabThera 100mg (concentrate for solution for infusion): summary of product characteristics[online]. Available from URL: www.rocheuk.com [Accessed 2006 Mar 10]). Overall, treatment with rituximab, in combination with fludarabine or as part of the FCR regimen, was well tolerated by patients with B-cell CLL in phase II trials[80-82], Incidences of severe neutropenia and infections were comparable to those seen with fludarabine-based regimens[81]. Myelosuppression was considered predominantly chemotherapy, rather than rituximab related. [80-82]

#### Pharmacokinetics:

Some facts are known from the intravenous administration of Rituximab in patients with B-cell malignancies:

1) The drug serum concentration is directly proportional to the administered dose and to the clinical response [71]. However, they are inversely correlated to the absolute level of circulating peripheral B cells and the tumor bulk measurements at baseline. [83] 2) Repeated administration results in accumulation of the drug due to reduction in the population of both normal and malignant CD20-positive B cells and the reduction or saturation of CD20-binding sites[71]. 3) There is wide interindividual variability reflecting the variable tumor responsiveness and burden among patients with B-cell malignancies. 4) Clinically relevant drug concentrations were detectable by ELISA in the serum of these patients up to 6 months after treatment [71]. 5)



Fig. 6 Rituximab ELISA. The mean of triplicate assays was 41.1 +/- 5.5  $\mu$ g/ml and 11.8 +/- 0.7  $\mu$ g/ml for 2 spiked samples of 40.0 and 10.0  $\mu$ g/ml.

Rituximab serum concentrations were significantly lower in patients with B-cell CLL. [84] This is probably due to the presence of the soluble CD20 antigens, found in patients with CLL, that act as a 'sink' for rituximab, increasing clearance and reducing delivery of the drug to malignant B cells.

Very limited information is available though on pharmacokinetics of Rituximab in the settings of allogeneic HCT. We aim to study these pharmacokinetics in the current patient population and ask questions about serum concentrations and correlations to drug dose and clinical responses at different time points after HCT. There is no commercial assay available to determine serum concentrations of rituximab. The Maloney lab has developed a murine anti-idiotype (anti-Id) monoclonal antibody (18C9) which binds specifically to rituximab, to the murine parent antibody used to construct rituximab, and to Fab' fragments of these antibodies and which does not cross-react with other human IgG1 antibodies or human serum (Fig. 6). The 18C9 anti-Id was used to develop an ELISA to measure serum rituximab concentrations. This assay can quantify rituximab levels in fresh, refrigerated or frozen human serum to <1  $\mu$ g/ml. We will use this assay to measure rituximab levels in patients before and after allogeneic HCT; we will correlate serum levels with response and relapse rates, and evaluate the effectiveness of our dosing regimen in consistently achieving trough serum rituximab levels of >25  $\mu$ g/mL based on a reported correlation of trough levels >25  $\mu$ g/mL with disease response [83].

#### Genetic determinants of responsiveness to Rituximab

Polymorphisms of the Fc $\gamma$ RIIIa receptor predominantly expressed on NK cells, have been shown to affect the antitumor activity of Rituximab in some but not all studies. [85-87] The Fc  $\gamma$ RIIIa of individuals that are homozygous for valine at position 158 (158V/V) has a higher affinity for human IgG1 than Fc $\gamma$ RIIIa that are homozygous for F (158F/F), and confers greater antibody dependent cell mediated cytotoxicity in vitro. [85] Patients with 158V/V have better and more durable responses to Rituximab than patients with 158F/F, while 158 V/F heterozygotes have a variable response. Maloney lab has developed a method to genotype FC  $\gamma$ RIIIa by PCR and

single-strand conformation polymorphism (SSCP). A region of exon 4 of FC  $\gamma$ RIIIa was amplified by PCR and the 125 bp product verified on a 2% agarose gel and by sequencing (**Fig 7A**). The PCR products were denatured and then electrophoresed through pre-cast 20% TBE in

Xcell II Mini-Cell gel electrophoresis unit in 1% TBE buffer to separate the different strands (**Fig. 7**). This is a sensitive method to identify Fc γRIII polymorphisms from small amounts of DNA isolated from patient or donor cells. A similar method has been developed to detect the



**Figure** 7: (A) PCR amplification of FC $\gamma$ RIIIa exon 4 from 3 patients, (B) SSCP analysis of the 3 samples, V/V, V/F, and F/F. Data from D. Maloney.

position 131 (histidine/arginine) polymorphism in the Fc receptor CD32, which has also been correlated with Rituximab response in some studies. [85] This method will be used to determine the genotype of these polymorphisms in hematopoietic cells pre and post NM HCT.

Patients with FcR polymorphisms that provide high affinity binding for human IgG1 had higher response rates or longer duration of remission following Rituximab therapy in some studies. This has not been evaluated in the context of allogeneic HCT, where the FcR status may change pre and posttransplant. We hypothesize that CD16 158 (VV) and CD32 131(HH) will be associated with increased efficacy and better outcome. It is unknown whether donor or recipient Fc  $\gamma$ RIII genotype will be more relevant for the efficacy of Rituximab in NM HCT.

#### **GVHD**

Cumulative incidence of extensive chronic GVHD in our 82 CLL patients was 50%. We will study in this protocol whether the addition of Rituximab would reduce chronic GVHD rates in comparison to our historical CLL patients given nonmyeloablative HCT. This is based on several reports indicating efficacy of Rituximab in treating refractory chronic GVHD. [88-92] Responses have been limited to cutaneous and musculoskeletal features[88-90] with few exceptions. [93] The precise role of B cells in chronic GVHD and the mechanism of benefit from rituximab remain controversial. Autoantibodies have been implicated in the pathogenesis of chronic GVHD by some groups [94], and rituximab may function by suppressing their production [89]. Alternately, rituximab-mediated B-cell depletion may modulate T-cell alloreactivity, as in other autoimmune diseases [95]. Given the clinical benefit in established chronic GVHD, administration of rituximab in the early post-transplant period may have a prophylactic effect, reducing the incidence or severity of chronic GVHD.

#### I. Assessment of Pretransplant Comorbidities

Charlson Comorbidity Index (CCI) is a well-known simple index to score comorbidities which was developed to provide prediction of risks of survival after treatment of chronic medical illnesses.[96] The Seattle team used this index in 2004 to score pretransplant comorbidities among patients diagnosed with hematological malignancies and offered HCT. The CCI was helpful in predicting risks of non-relapse mortality and survival[97,98]. However, the CCI showed a limited ability in capturing comorbidities among the transplanted population. Therefore, the same authors investigated the possibility of modifying the original CCI to better

capture comorbidities among transplanted patients.[99] They tried to a) better define previously identified comorbidities utilizing pretransplant laboratory data, b) investigate additional HCT-related comorbidities, and c) establish comorbidity scores that were suited for HCT. This resulted in developing a new HCT-specific comorbidity index (HCT-CI), which captured comorbidities among 62% of patients with scores >0 compared to 12% captured by the original CCI.[99] Additionally, the new index was superior to the old CCI in prediction of survival (likelihood ratio of 23.7 versus 7.1 and *c* statistics of 0.661 versus 0.561, *P*=<0.0001, respectively). Recently, the HCT-CI was shown to be an important prognostic and risk-assessment factor in comparing outcomes of patients diagnosed with CLL and given myeloablative versus nonmyeloablative HCT. [100]

#### 3. Proposal

We intend to study whether allogeneic HCT after nonmyeloablative conditioning and peri-HCT Rituximab is effective therapy for CLL. We intend to demonstrate this by comparing survival of patients transplanted under this protocol to that achieved in the historical controls after treatment with CAMPATH.

#### 4. Objectives

#### A. Primary objective

1. Determine whether nonmyeloablative conditioning and allogeneic HCT improves survival at 18 months for patients with fludarabine-refractory, FCR-failed, or del 17p CLL over that of historical controls (45% at 18 months) given CAMPATH-1H.[14]

#### B. Secondary objectives

- 1. Estimate the overall response rate (CR + PR) by standard morphologic, flow cytometric, and molecular techniques.
- 2. Assess the rate of relapse/progression.
- 3. Define incidences of RRT and infections within the first 100 days and the incidence of TRM within the first year.
- 4. Estimate incidences of grade II-III and III-IV acute GVHD and chronic GVHD.
- 5. Assess the impacts of Rituximab
  - a. Determine whether the addition of Rituximab to the nonmyeloablative conditioning and allogeneic HCT improves survival at 18 months over our historical data (57% at 18 months).

- b. Determine the incidence of serious adverse events with the addition of Rituximab in comparison to historical data of unrelated nonmyeloablative HCT.
- c. Evaluate the pharmacokinetics of Rituximab.
- d. Evaluate B-cell and T-cell immune reconstitution in comparison to historical data of unrelated nonmyeloablative HCT.
- e. Describe donor and host polymorphisms of the FCγRIIIa receptor and CD32 and evaluate their impact on disease response and relapse.

#### 6. Graft-versus-leukemia analysis

- a. Investigating mechanism of disease resistance in relapsed/non-responding patients
- b. Isolation of donor cytotoxic T lymphocytes specific for host minor histocompatibility antigens

#### 5. Patient Selection

#### A. Inclusions:

- 1. Patients with a diagnosis of CLL (or small lymphocytic lymphoma) or Diagnosis of CLL that progresses to prolymphocytic leukemia (PLL).
- 2. Patients with B-Cell CLL or PLL who:
  - a. Failed to meet NCI Working Group criteria<sup>2</sup> (Appendix H) for complete or partial response after 2 cycles of therapy with a regimen containing fludarabine (or another nucleoside analog, e.g. 2-CDA, pentostatin) or with disease relapse within 12 months after completing therapy with a fludarabine (or another nucleoside analog) containing regimen.
  - b. Failed FCR or PCR combination chemotherapy at any time point.
  - c. Patients with novo or acquired "17p deletion" cytogenetic abnormality. Patients should have received induction treatment but could be transplanted in 1<sup>st</sup> CR.
- 3. Patients who have suitable HLA-matched related or unrelated donors willing to receive G-CSF, undergo leukapheresis to collect PBMC, and to donate stem cells.
- 4. Patients who are older than 18 years old.

#### B. Exclusions:

- 1. Infection with HIV.
- 2. Active diagnosis of CNS involvement with CLL. For LP requirement, see Appendix N.
- 3. Patients unwilling to use contraceptive techniques before and for 12 months after HCT
- 4. Pregnant women or females who are breastfeeding.
- 5. The addition of cytotoxic agents for "cytoreduction" with the exception of tyrosine kinase inhibitors (such as imatinib mesylate), cytokine therapy, hydroxyurea, low dose cytarabine, chlorambucil, or rituxan will not be allowed within three weeks of the initiation of conditioning.

- 6. Active bacterial or fungal infections unresponsive to medical therapy.
- 7. Performance status:
  - a. Karnofsky score < 60 (see **Appendix B**) for adult patients
- 8. Severe organ dysfunction:
  - a. Cardiovascular:
    - i. Cardiac ejection fraction < 40%. Ejection fraction is required if age > 50 years or there is a history of prior transplant, anthracycline exposure or history of cardiac disease
    - ii. Poorly controlled hypertension despite multiple antihypertensives.

#### b. Pulmonary:

- i. DLCO < 40%, TLC <40%, FEV1 <40% and/or requiring continuous supplementary oxygen, or severe deficits in pulmonary function testing as defined by pulmonary consultant service.
- ii. The FHCRC PI of the study must approve of enrollment of all patients with pulmonary nodules.

#### c. Hepatic:

Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension. Patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, hepatic damage with bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin >3 mg/dl, or symptomatic biliary disease.

- 9. Patients with active non-hematologic malignancies (except non-melanoma skin cancers). This exclusion does not apply to patients with non-hematologic malignancies that do not require therapy.
- 10. Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a >20% risk of disease recurrence.
  - This exclusion does not apply to patients with non-hematologic malignancies that do not require therapy.

#### 6. Donor Selection

#### A. Inclusions

#### 1. Related donors

When more than one potential donor exists, priority should be given to donors based on HLA identity > CMV seronegativity > ABO compatibility > sex matching. Eligibility guidelines for donor PBMC apheresis based on immunization status are shown in Appendix A.

- a. <u>Donor who is HLA phenotypically or genotypically identical at the allele level at HLA-A, -B, -C, -DRB1, and -DQB1.</u>
- b. Donor must consent to G-CSF administration and leukapheresis.
- c. Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian).
- d. Only G-CSF mobilized PBMC only will be permitted as a HSC source on this protocol.

#### 2. Unrelated donors

- **a.** FHCRC matching allowed will be Grades 1.0 to 2.1 (Appendix O): Unrelated donors who are prospectively:
  - Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing;
  - ii) *Only a single allele disparity* will be allowed for HLA-A, B, or C as defined by high resolution typing (see **Appendix O for other donor selection details**).
- **b.** Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment. This determination is based on the standard practice of the individual institution. The recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT. If the PRA shows >10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained. The donor should be excluded if any of the cytotoxic cross match assays are positive. For those patients with an HLA Class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results. A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion.
- c. Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A\*0101 and the donor is A\*0102, and this type of mismatch is not allowed.
- **d.** Only G-CSF mobilized PBMC will be permitted as a HSC source on this protocol.

#### **B.** Exclusions

- 1. Age < 12 years
- 2. Identical twin
- 3. Pregnancy
- 4. Infection with HIV
- 5. Inability to achieve adequate venous access
- 6. Known allergy to filgrastim (G-CSF)
- 7. Current serious systemic illness

#### 7. Informed Consent

#### Patient

A conference conducted by the outpatient, attending physician will be held with the patient and family to discuss this study and alternative treatments available for treatment of advanced CLL. The goals of the study, requirement for data collection, and requirement for release of medical records will be discussed with the patient. All potential risks associated with the use of fludarabine, low dose TBI, Rituximab, immunosuppressive drugs, HCT, and disease progression/recurrence will be discussed as objectively as possible. Discussion of potential complications should include graft rejection, GVHD, infections, and death. It should be explained that patients offered this protocol have advanced malignancy with life expectancy of about 10 months with conventional treatments, and are at high risk of early transplant mortality with conventional allogeneic HCT and high relapse rate after an autologous transplant. It should also be explained to the patient that our preliminary results showed no difference in outcomes after related or unrelated donor nonmyeloablative allogeneic HCT.

Informed consent from the patient will be obtained using a form approved by the Institutional Review Board (IRB) of the Fred Hutchinson Cancer Research Center and the local IRB if the patient is treated in a collaborating institution. The patient is also required to sign a HIPPA consent form.

#### Donor

For the family member stem cell donor, the procedure for collecting peripheral blood mononuclear cells and toxicities of G-CSF will be explained. The donor should be counseled as to the risks of treatment with G-CSF and be informed that leukapheresis at several time points may be necessary. Informed consent from the patient and donor will be obtained using forms approved by the Institutional Review Board of the Fred Hutchinson Cancer Research Center. All patients enrolled at collaborating centers will engage in institution-specific informed consent conferences after completion of the pre-transplant evaluation. Informed consent from the donor and patient will be obtained using a form approved by the Institutional Review Board for each treatment center.

Informed consent from the unrelated donor will be obtained according to NMDP regulations.

#### 8. Protocol Registration

<u>A. FHCRC patients</u>: Eligible patients will be assigned to the protocol by the Clinical Coordinator who will register the patient with the Registration Office (206-667-4728) between 8:30 am and 4:00 pm, Monday through Friday. After hours, the Registration Office can be reached by paging (206) 995-7437.

<u>B. Collaborating institutions</u>: Eligible patients will be identified by the principal investigator of the collaborating institution who will register the patient with the FHCRC Registration Office. Registration will include completion of the eligibility checklist and demographic form (Appendix L). This form and a copy of the signed informed consent will be faxed to the Trial Coordinator (206-667-5378). Questions regarding eligibility or protocol information should be directed to the Principal Investigators, Mohamed Sorror, M.D. (206-667-2765) or David Maloney, M.D. (206-667-5616).

#### 9. Plan of Treatment

#### A. Outline of treatment plan

The plan for treatment is shown below in Figure 8 and described in Table 4.

#### B. HCT

Patients will undergo HCT as soon as eligibility requirements are met and donor leukapheresis, for related recipients, is scheduled (in practice approximately 7-21 days after the arrival conference). For unrelated recipients, HC source will be G-PBMC collected as per NMDP or other regulatory protocol. Two (12 liters) leukaphereses will be obtained on consecutive days, and collections will be infused together on day "0".

Patients will only be admitted as medically necessary for control of transplant complications or for the infusion of HCT.

For unrelated recipients, standard cryopreservation of 10% of the G-PBMC will take place for DLI.

#### C. Cytoreduction

Cytoreduction and /or radiation therapy may be given by the referring physician or the attending physician as determined on clinical grounds or to meet eligibility requirements of the protocol for patients with advanced malignancy or to reduce tumor bulk. Cytoreduction can be performed with any appropriate therapy for CLL. The choice of therapy will depend on prior regimens and the current disease status and may be selected at the discretion of the attending physician and/or the referring physician. However, no intensive chemotherapy can be given within three weeks (or the interval in which a cycle of standard chemotherapy would be administered in a non-transplant setting) prior to initiating the nonmyeloablative transplant conditioning (see exclusion criteria page 19). The need for this therapy should be discussed with the principal investigator. The referring oncologist may be asked to administer this therapy. Alemtuzumab should be given only >60 days before allogeneic HCT to avoid its lingering immunosuppressive effect on the donor graft.

**Definition of Preceding Chemotherapy and Biologic Modifiers:** For the purposes of this protocol, preceding chemotherapy is defined as any exposure to systemic chemotherapy. Exceptions to this definition include cytokine therapy, low dose cytarabine, chlorambucil, or rituxan.

#### D. Conditioning regimen

Conditioning will begin four days prior to stem cell infusion.

- i. On days –4 to –2 patients will receive fludarabine intravenously at a dose of 30 mg/m²/day.
- ii. On day -3, patients will receive rituximab intravenously at a dose of 375 mg/m<sup>2</sup>.
  - Follow SCCA general oncology guidelines for infusion of drug
  - Follow SCCA general oncology guidelines for rituximab pre-meds and prn reactions
- iii.On day 0, 200cGy of TBI will be administered at 6-10 cGy/min from a linear accelerator. TBI will be administered between 10:00 a.m. and 2:00 p.m. to avoid proximity to the start of immunosuppression.
- iv. G-PBMC from an HLA-matched donor, will be infused on day 0, following TBI.
- v. Patients will receive rituximab intravenously at a dose of 375 mg/m² at three time points after stem cell transplantation. These time points are set up at days 10+, 24+, and 38+. However, if there are clinical reasons that prohibit giving Rituximab at one of these specified time points the dose can be delayed to a maximum of 5 days. Following doses should be attempted to be given at the scheduled time points. If doses need to be delayed more than 5 days from the specified time points, then patient should only get the next scheduled dose Day 38+ dose can be delayed up to 100 days after HCT.

**Table 4. Conditioning Schema and Immunosuppression Schedule** 

| | | _ | unic | ••• | onantioni | <del></del> 5 ~ ∙ | | | | -osupp | Coston | ~ circuatio | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day number | -4 | -3 | -2 | -1 | 0 | +1 | +10 | +24 | +27 | +38 | +40 | +56 | +96 | +100 | +180 |
| Fludarabine | X | X | X | | | | | | | | | | | | |
| TBI | | | | | 200 cGy | | | | | | | | | | |
| Rituximab | | X | | | | | X <sup>A</sup> | X <sup>A</sup> | | X <sup>A</sup> | | | | | |
| Stem cell infusion | | | | | Infusion | | | | | | | | | | |
| Related recipients | | | | | | | | | | | | | | | |
| CSP | | Start | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | | $\rightarrow$ | $\rightarrow$ | Taper <sup>B</sup> | $\rightarrow$ | $\rightarrow$ | Stop |
| MMF | | | | | Start <sup>C</sup> | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | Stop | | | | | | |

<sup>&</sup>lt;sup>A</sup>These are recommended time points that can be delayed for a maximum of 5 days for clinical reasons.

Unrelated recipients

| em emen ree | en cuicu recipients | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CSP | | Start | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | Taper <sup>C</sup> | Stop |
| MMF | | | | | Start <sup>D</sup> | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | $\rightarrow$ | Taper <sup>D</sup> | $\rightarrow$ | Stop | | |

<sup>&</sup>lt;sup>C</sup>Taper will be a ~8% dose reduction per week x 11 weeks.

#### E. Immunosuppression

- Postgrafting immunosuppression with CSP and MMF will be used to permit engraftment and provide GVHD prophylaxis.
- Day –3. Commence CSP at 5.0 mg/kg PO Q12 hrs, continue to day +56 for related and day +100 for unrelated recipients, then taper to day +180. CSP should be routinely taken at 9:00 a.m. and 9:00 p.m.
- Day 0: **After** HCT on day 0, MMF will be given based on adjusted body weight, at 15 mg/kg PO, 4-6 hours after HCT is complete.
  - For related recipients MMF to be given at 15 mg/kg PO Q12 hrs, continue to day +27, then stop abruptly.
  - For unrelated recipients MMF to be given at 15 mg/kg PO Q8 hrs, continue to day +40, then start to taper to day +96

CSP and MMF treatment and taper schedules are described below and depicted in Table 4.

<sup>&</sup>lt;sup>B</sup>Taper will be a ∼6% dose reduction per week x 17 weeks.

<sup>&</sup>lt;sup>C</sup>The first dose of MMF is to be given 4-6 hours after the stem cell infusion.

<sup>&</sup>lt;sup>D</sup>The first dose of MMF is to be given 4-6 hours after the stem cell infusion

Figure 8. Diagram of treatment plan



If T-Cell (CD3) chimerism is >50% on day +28, then repeat only on days +84 and +365. If T-Cell (CD3) chimerism is  $\le 50\%$  on day +28, then repeat on days +56, +84, +180, & +365.

Granulocyte (CD33) chimerism on day +84 only.

Natural killer (NK) cell (CD56+) chimerism will be obtained on day 28.

Bone Marrow chimerism will be obtained on days +84 & +365

#### (See Patient Post-Transplant Evaluation for more details)

#### 1. CSP

- a. CSP Administration Plan
  - i. Starting dose: CSP (Neoral is preferred) is given orally based on adjusted body weight at 5.0 mg/kg Q12 hrs PO from starting day -3. Doses should be adjusted to maintain high therapeutic CSP levels as discussed below.
  - ii. If there is no evidence of GVHD, *for related recipients:* a CSP taper will be initiated on day +56. CSP will be tapered so that patients will be off of CSP by day +180 (approximately 6% decrease every seven days). *For unrelated recipients:* a CSP is to be tapered from day +100 at 8% of the pre-taper therapeutic dose per week to be discontinued at the end of 11

weeks (day +180). The referring physician, who will receive explicit instructions and guidelines for detecting and managing GVHD, will manage this.

iii. If there is evidence of chronic GVHD, then the standard recommendations for chronic GVHD with CSP/prednisone will be followed.

iv. If there is evidence of CLL disease progression, please see section K.

#### b. Guidelines for CSP Dose Adjustment and Monitoring

- i. Blood pressure, renal function (serum creatinine, BUN), electrolytes and magnesium need to be followed at least three times per week during the first month, twice weekly until day +100, then once per week until CSP is stopped, unless clinical circumstances suggest the need for more frequent evaluations.
- ii. CSP, whole blood "trough" levels (i.e., just prior to the next dose) will be evaluated on day 0 and twice weekly post-transplant until the initiation of the taper and adjusted if necessary to maintain blood levels that target upper end of therapeutic range (see Table A) during the 28 days.

Table A: CSP Dose Adjustment

| able A. CSI Dose Aujustment | CSP Level to Target Using LC-MS/MS Method | CSP Level to Target Using<br>Immunoassay Method |
|---|---|---|
| Day "0"- Day +28<br>Whole blood "trough" (11-12 hrs<br>from prior dose) | 400 ng/ml | 500 ng/ml<br>(upper end therapeutic range for<br>this method) |
| After Day +28 | 120 - 360 ng/ml | 150 - 450 ng/ml |
| Levels >480 mg/ml by LC-MS/MS Method • with or without CSP toxicity • decrease GFR \geq 50% • increase creatinine 2x baseline due to CSP | 25% dose reduction | N/A |
| Levels >600 mg/ml by Immunoassay Method • with or without CSP toxicity • Decrease GFR >50% • increase creatinine 2x baseline due to CSP | N/A | 25% dose reduction |
| Patients on Hemodialysis | 320 ng/ml | 400 ng/ml |

- iii. CSP Monitoring: CSP determinations should be performed on a twice weekly basis for the first month and then weekly until day +56 *for related* and day +100 *for unrelated recipients* unless high levels are detected (i.e., >600ng/ml), or toxicity is suspected in which case more frequent monitoring will be performed as clinically indicated. Routine monitoring of CSP will not be required for patients on a CSP taper after day + 140 unless clinically indicated.
- iv. CSP Dose Adjustment: Initial high Cyclosporine (CSP) doses are required based on the pre clinical nonmyeloablative canine studies, which used an equivalent dose to establish an allograft. After day +28, CSP levels typical for related or unrelated HCT will be targeted. Dose reduction should only be made if CSP toxicity is present, and/or levels exceed values provided in Table A. There are two methods for calculating CSP levels. Table A provides desired levels for specific methods. To avoid inadequate immune suppression, dose reductions should be conservative. Therapeutic levels of CSP should be maintained.
- v. After day +28, typical serum CSP transplant levels for related or unrelated HCT between 120 and 360 will be targeted.

vi. Dose reductions should only be made if CSP toxicity is present or levels exceed 480 ng/ml - 600ng/ml depending on method (see Table A), in the absence of toxicity. Dose reductions for high levels without toxicity should be conservative e.g. 25%, to avoid inadequate immunosuppression.

vii. If there is nausea and vomiting at anytime during CSP treatment the drug should be given intravenously at the dose that was used to obtain a therapeutic level. **Oral to IV conversion:** 

Oral CSP dose  $\div$  2.5 = IV dose

Oral Sandimmune may be substituted for oral Neoral.

viii. Patients requiring hemodialysis should be have CSP levels maintained in the high therapeutic range (Table A).

ix. Drugs that may affect CSP levels are:

| <b>Decrease CSP levels</b> | Increase CSP lev | els | <b>Enhance Potential for</b> |
|---|---|---|---|
| | | | Nephrotoxicity |
| Phenytoin | Erythromycin | Diltiazem | Aminoglycosides |
| Phenobarbital | Alcohol | Doxycycline | Loop diuretics (furosemide) |
| Carbamazepine | Ketoconazole | Verapamil | Amphotericin formulations |
| Primidone | Acetazolamide | Nifedipine | |
| Rifampicin | Fluconazole* | Nicardipine | |
| Nafcillin | Colchicine | Azithromycin | |
| Octreotide | Itraconazole* | Imipenem | |
| Sulfonamides | Fluoroquinolones | | |
| Trimethoprim | Voriconazole | | |
| Metoclopramide | Caspofungin | | |
| ste . | Clarithromycin | | |

<sup>\*</sup>Discontinuation of fluconazole or itraconazole may lower CSP levels, and if used for antifungal prophylaxis, then changes in these drugs should be avoided during the first 2 months posttransplant.

#### 2. MMF

a. <u>Initiating MMF therapy</u>: *For related recipients:* Oral administration of MMF will be at a daily total dose of 30 mg/kg/day based on adjusted body weight (15 mg/kg/d every 12)

*For unrelated recipients:* Oral administration of MMF will be at 15 mg/kg Q8 hours (45mg/kg/day), based on adjusted body weight.

- b. The first dose will be on the evening of day 0 (i.e. first dose to follow 4-6 hours after stem cell infusion).
- c. Doses will be rounded to the nearest 250 mg (capsules are 250 mg).
- d. If there is nausea and vomiting at any time preventing the oral administration of MMF, MMF should be administered intravenously at 15 mg/kg Q8 hours.
- e. <u>Stoppage/Tapering of MMF</u>: *For related recipients*, MMF will be given until day +27 post-transplant and then stopped without tapering in the absence of GVHD that requires therapy (e.g. steroids). If treatment for GVHD is required prior to day +27, MMF will be continued at full dose until a steroid taper begins.

For unrelated recipients, MMF will be given based on adjusted body weight daily at 15 mg/kg Q8 hrs until day +40 post transplant and then tapered by 12%/week to be discontinued after day +96, in the absence of GVHD requiring therapy.

- f. Guidelines for MMF dose adjustment for drug toxicity: If in the clinical judgment of the investigator and/or attending physician the observed toxicity is related to MMF administration, a dose adjustment will occur. The discontinuation of MMF at any point should be discussed with the Study PI and should be documented in the permanent medical record and all Case Report Forms (CRF). Based on previous organ transplant studies, dose adjustments are likely to occur because of hematopoietic or rarely gastro-intestinal adverse effects.
  - i. Neutropenia: A thorough evaluation of neutropenia should occur including peripheral blood chimerism studies, marrow aspiration and review of marrow suppressive medications (e.g. bactrim). G-CSF may be started at 5μg/kg subcutaneously qd to facilitate neutrophil recovery for patients with ANC <750/ul 21 days after HCT. Dose adjustments of MMF will only be made for severe neutropenia that develops or persists after day 21 post-transplant (ANC < 100/μl for > 5 days) that is refractory to G-CSF treatment independent of any other toxicity. In this case dose reductions could be made and should be conservative (20-25%). MMF should only be discontinued temporarily. The MMF should be restarted at 20% reduced dose when the underlying toxicity subsides. Any planned dose adjustments for hematologic toxicity **must** be discussed with the principal investigator.
  - ii. Gastrointestinal toxicity: In the event of gastrointestinal toxicity that requires medical intervention including medication for control of persistent vomiting or diarrhea and is considered to be due to MMF, a 20% dose reduction will occur first and if there is no

improvement, MMF will be reduced a further 20%. For severe G.I. toxicity related to MMF, then MMF may be stopped. Patients should be evaluated by a Gastroenterology consultant to determine the need for dose adjustments for this indication.

#### F. Collection and infusion of donor G-PBMC

#### 1. G-CSF Administration to Donors:

For related recipients: From day -4 to day -0, all PBSC donors will receive G-CSF, at a dose of 16  $\mu$ g/kg/day, for 5 consecutive days (Table 5). G-CSF will be administered by a subcutaneous daily injection. The schedule of G-CSF administration and PBSC collections can only be ascertained once day 0 is identified. Once a treatment regimen schedule has been fixed and the schedule of G-CSF administration and PBSC collections made this has to be confirmed with the personnel in the apheresis room. Day 0 should be fixed on a Tuesday-Thursday.

For unrelated recipients: Timing of G-PBMC collection is prearranged through the NMDP. Day 0 should be fixed on a Monday-Thursday when possible. G-CSF will be administered by subcutaneous injection to the unrelated donor starting 5 days prior to the day of HCT (see Table 5) as per NMDP protocol. Donors will receive approximately 10 μg/kg of G-CSF each day of mobilization. A 12 liter apheresis will be obtained on day −1 and possibly on day 0 for a total of 12 to 24 liters of apheresis collection that will be infused on day 0.

**Table 5. Treatment Schema for donor** 

| Day | -5 | -4 | -3 | -2 | -1 | 0 |
|---------------------|----|----|----|----|----|---|
| G-CSF (10-16 ug/kg) | X | X | X | X | X | |
| G-PBMC collection | | | | | X | X |

#### 2. <u>G-PBMC Collection</u>:

For related recipients: donors will preferably undergo vein-to-vein collections or may receive an appropriate catheter inserted on or before day of apheresis. Two 12-liter leukaphereses on consecutive days will be obtained, and cells will be infused together on day 0. First, PBSCs will be collected in the afternoon of day -1, stored in the refrigerator at 4°C overnight. A second collection will be performed the following afternoon and both collections will be transfused on day 0. If  $< 5 \times 10^6$  CD34+ cells/kg are collected an additional day of collection will be performed. If PBSCs cannot be collected by a vein-to-vein technique, a percutaneous Mahurkar catheter will be inserted. General procedures will include the use of a standard apheresis machine (COBE Spectra, Lakewood Colo.), and processing up to 16 liters of whole blood during the collection

For unrelated recipients: G-PBMC scheduling and collection is arranged through the NMDP. The schedule of GCSF administration and collection of PBMC is

determined as per NMDP protocol. The physician responsible for HC collection will obtain informed consent from the donor.

3. <u>HCT infusion</u>: All patients will receive unmodified G-PBMC infusion on day 0 of the treatment regimen (Refer to institutional practice guidelines for methods of infusion).

#### G. ABO incompatibility

All patients with ABO incompatibility should be evaluated and treated according to the standard practice of the individual institution. Recommendations are provided in Appendix C. It should be noted that two cases of recipient hemolysis have been documented in patients with minor ABO mismatch with their donor. The suspected cause is donor anti-host hemagglutinin production from "passenger lymphocytes" in the donor G-PBMC that may expand posttransplant[101]. Therefore, these patients should be monitored and treated aggressively when there is any evidence of hemolysis.

#### H. Post-transplant growth factors

Patients are not eligible to receive post-transplant growth factors such as G-CSF during the first 21 days. Growth factors should not be given unless severe persistent neutropenia develops or persists past day 21 post-transplant (ANC <500/ $\mu$ l).

#### I. Infection prophylaxis

Patients should receive prophylaxis for PCP, VZV, HSV, CMV and candida according to the standard practice of the individual institution for a conventional allogeneic HCT. Recommended infectious prophylaxis is provided in Appendix D. Standard CMV monitoring and prophylaxis should commence at the time of initial transplant and should continue until 1 year post HSCT. Recommendations for monitoring and evaluation of infectious complications are specified in Appendix D. In case of low donor chimerism or disease progression that necessitates transfer of DLI to the patient, modifications in infection prophylaxis will be made according to that protocol.

#### J. Chimerism

#### 1. Definition

For the purposes of this protocol, definitions will be:

- a. Mixed chimerism will be defined as the detection of donor T cells (CD3+) and granulocytes (CD 33+), as a proportion of the total T cell and granulocyte population, respectively, of greater than 5% and less than 95% in the peripheral blood.
- b. Full donor chimerism is defined as > 95% donor CD3+ T cells. Mixed or full donor chimerism will be evidence of donor engraftment

- c. *Increasing donor chimerism* is defined as an absolute increase of 20% of donor CD3+ T cells over the previous chimerism evaluation.
- d. *Low donor chimerism* is defined as < 40% CD3+ T cells after HCT. Low donor chimerism should always be confirmed with repeat peripheral blood T cell and granulocyte chimerism analysis.
- e. Decreasing donor chimerism is defined as an absolute decrease of  $\geq$  20% of CD3+ T cell chimerism over the previous month.

A DNA-based assay that compares the profile of amplified fragment length polymorphisms (ampFLP) (or FISH studies or VNTR) of the patient and donor will be used to quantitate chimerism of sorted peripheral blood T-cells (CD3+) and granulocytes (CD 33+). The same assay should be used in a given patient for repeated studies of chimerism. This DNA-based analysis will also be performed on the whole nuclear cell fraction from marrow aspirates.

#### 2. Evaluation

Patients will have peripheral blood and whole bone marrow evaluations for chimerism at various time points through one year post transplant. If the patient has not obtained > 95% donor chimerism in CD+3 by one year continue to evaluate through 5 years post transplant as clinically necessary. Peripheral blood will be sorted to evaluate T-cell (CD+3), granulocyte (CD+33), **and/or** NK cell (CD56) compartments. (See Patient Post Transplant Evaluation section for instructions and exceptions).

#### 3. Continuation of immunosuppression

- a. In case of low or decreasing donor chimerism. Immunosuppression should be continued or reinitiated at full dose until the low donor chimerism is corrected or the patient may be eligible for another protocol for DLI according to institutional practice.
- b. Patients who reject their graft may be eligible for a second allogeneic transplant on other protocols.
- 4. Definition of mixed donor/host chimerism, engraftment, graft failure and rejection. For the purposes of this protocol, mixed chimerism will be defined as the detection of donor T cells (CD3+) and granulocytes (CD 33+), as a proportion of the total T cell and granulocyte population, respectively, of greater than 5% and less than 95% in the peripheral blood. Full donor chimerism is defined as > 95% donor CD3+ T cells. Mixed or full donor chimerism will be evidence of donor engraftment. Increasing donor chimerism is defined as an absolute increase of 20% of CD3+ T cells over the previous chimerism evaluation. Decreasing donor chimerism is defined as an absolute decrease of 20% of CD3+ T cell chimerism over the previous month. Low donor chimerism is defined as < 40% CD3+ T cells after HCT. Low donor chimerism

should always be confirmed with repeat peripheral blood T cell and granulocyte chimerism analysis. A DNA-based assay that compares the profile of amplified fragment length polymorphisms (ampFLP) (or FISH studies or VNTR) of the patient and donor will be used to quantitate chimerism of sorted peripheral blood T-cells (CD3+) and granulocytes (CD 33+). The same assay should be used in a given patient for repeated studies of chimerism. This DNA based analysis will also be performed on the whole nucleated cell fraction from marrow aspirates. Therapeutic decisions (i.e. DLI) will be made based on the results of sorted T-cell studies of peripheral blood. For the purposes of this protocol, rejection is defined as the inability to detect or loss of detection of greater than 5% donor T cells (CD3+) as a proportion of the total T cell population, respectively, after nonmyeloablative HCT. Also for the purposes of this protocol, graft failure is defined as grade IV thrombocytopenia and/or neutropenia after day 21 that continue, uninterrupted, for >3 weeks and is refractory to transfusions and growth factor support, respectively.

#### K. Management of disease progression

In case of disease progression and >40% T-cell donor chimerism. Evidence of substantial disease progression (as defined in Appendix H) will be an indication for therapeutic intervention. In part, this will be dependent on where a patient is relative to the standard tapering schedule. If the attending physician believes that the patient requires very aggressive therapy, the case will be presented to the institutions' patient review committee. Otherwise, priority should be given to rapid reduction of immunosuppression, option (i) below. Therapeutic options include:

- 1. Early discontinuation of immunosuppression (prior to day +28 for related and day +100 for unrelated recipients). This should be considered the first therapeutic maneuver. If there is no GVHD, MMF is to be stopped if still being taken, and CSP tapered over 2 weeks. Bone marrow aspirate and blood chimerism studies will be performed when off immunosuppression after 2 weeks. If disease continues to progress 2 weeks after stoppage of all immunosuppression, <20% increase in donor chimerism and there is no GVHD, patients will be considered as treatment failure. The patient may then be eligible for DLI treatment according to institutional practice.
- 2. Early discontinuation of immunosuppression (between days +28 and +180 for related and days +100 and +180 for unrelated recipients). If there is no

- GVHD, CSP is to be stopped. Bone marrow aspirate and blood chimerism studies will be performed when off immunosuppression after 4 weeks. If disease continues to progress 2 weeks after stoppage of all immunosuppression, T cell chimerism has not significantly increased (<20% increase) and there is no GVHD, patients will be considered as treatment failure. The patient may then be eligible for DLI treatment or according to institutional practice.
- 3. <u>Intercurrent treatment with chemotherapy or radiation</u>. Conventional chemotherapy or radiation therapy should be considered in the setting of life threatening disease progression. Patients in this situation would be considered treatment failures. After therapy is completed, the patient may then be eligible for DLI treatment or according to institutional practice.
- 4. <u>Conventional allogeneic HCT.</u> This option should be discussed with the institutions' patient review committee and the principal investigator. Patients who undergo conventional allogeneic HCT will be removed from the protocol at that time.

#### 10. Patient and Donor Evaluations

- A. Patient Pretransplant Baseline Evaluation
  - 1. History: A complete history with full details of the patient's prior treatment and response
  - 2. Assessment of patient pretransplant comorbidities and scoring them using the HCT-Comorbidity Index (HCT-CI; see Appendix Q).
  - 3. Careful physical exam with determination of Karnofsky score (Appendix B).
  - 4. Complete blood count (CBC), serum sodium, potassium, chloride, CO<sub>2</sub>, creatinine, BUN, uric acid, calcium, magnesium, phosphate, total bilirubin, alkaline phosphatase, AST, ALT, ABO/Rh typing, hepatitis screen, CMV, VZV, HSV and toxoplasma serology, and anti-HIV serology.
  - 5. Chest X-ray (CXR), PA and lateral views.
  - 6. Pulmonary function tests with corrected DLCO.
  - 7. MUGA scan or echocardiogram to evaluate cardiac ejection fraction for patients > 50 years of age, or history of cardiac disease or prior transplant or anthracycline exposure.

#### Additionally, see Table 6 for further pre-transplant evaluations.

Table 6: Disease-Specific Pre-Transplant Evaluations

Note: Bone marrow aspirates and biopsies are recommended to be **bilateral** and to be collected within **30 days** of treatment. See Tables 7, 8 and 9 for post-transplant evaluations and additional lab instructions.

| Specimen / Test / Imaging | Clinical /<br>Research | Comment |
|---|---|---|
| Bone marrow aspirate | | |
| Pathology | Clinical | |
| Flow Cytometry | Clinical | |
| Cytogenetics | Clinical | |
| FISH for clonal abnormalities | Clinical | |
| Bone marrow biopsy | | |
| Pathology | Clinical | |
| Peripheral Blood | | |
| Storage for chimerism analysis | Clinical | |
| Quantitative Ig levels | Clinical | |
| β-2 microglobulin | Clinical | |
| LDH | Clinical | |
| ZAP – 70 by flow cytometry– *see comment | Clinical | *for patients not in CR |
| Rituxan trough levels – *see comment | Research - | *Should be done immediately prior |
| Kituxan trough levels – see comment | Maloney Lab | to the Day -3 dose |
| Imaging | | |
| CT of chest, abdomen, pelvis (neck if indicated) | Clinical | |
## **Pre-conditioning/Pre-transplant** Research Studies **only** for FHCRC patients who have signed **Consent D**;

- 1. Send 40cc heparinized blood and one 10ml red top tube to the Maloney Lab (206-667-4284; FHCRC D1-331) for cryopreservation of tumor cells. Label the samples "Protocol 1840." These cells will be used as a possible source of leukemia against which the efficacy of killer T cells could be evaluated. The option of leukapheresis for sample acquisition will be discussed with the patient and Attending Physician.
- 2. Leukapheresis may be done in order to collect a large volume of mononuclear cells. Leukapheresis will be performed using the apheresis machines at the Seattle Cancer Care Alliance and will be done prior to the start of transplant conditioning.

#### B. Patient Post-transplant Evaluation

1. See Table 7 for disease specific post-transplant evaluation on Day +28, 56, 84, etc. This is a recommended evaluation schedule.

#### Additionally, include the following for all diseases:

- 2. CBC three times a week, or more often if clinically indicated, from day 0 until day +28, and twice weekly until 2 months post-transplant or later if clinically indicated.
- 3. Electrolyte panel and renal and hepatic function 3 times per week until day +28 and then weekly.
- 4. Evaluate at Day +84

GVHD evaluation guidelines:

- a. History and physical exam with attention to the evaluation of chronic GVHD (Appendix G)
- b. Complete blood count, serum IgG, and serum total bilirubin, alkaline phosphatase, ALT, and AST
- c. Skin biopsy
- d. Schirmer's tear test
- e. Pulmonary function test
- f. Oral exam
- g. Dietician assessment
- h. Gynecological assessment (adult female)

See Section 11 for diagnosis and treatment guidelines for acute and chronic GVHD.

5. Patients should be assessed for the need of IVIG monitoring and replacement therapy per Institutional Guidelines

**Table 7: Post-Transplant Evaluation (**See text for pre-transplant evaluations)

This is a recommended evaluation schedule. Note that research draws are for FHCRC patients only. See Table 8 for peripheral blood research studies. See Table 9 for additional lab instructions.

| Disease | Specimen/ Test/ Imaging | Clinical/ | Comment | | Days | | | Ye | Annual x | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Research | | 28 | 56 | 84 | 180 | 1 | 1.5 | 5 years |
| CLL | | | transplant if patient is in CR, bone | marrow | is recomn | nended o | nly as clir | ically ind | icated. | |
| | Chimerism | Clinical | | | | X | | X | | |
| | Pathology | Clinical | | X | X | X | X | X | X | X |
| | Flow cytometry | Clinical | | X | X | X | X | X | X | X |
| | Cytogenetics | Clinical | *If abnormal pre-transplant | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see comment |
| | FISH | Clinical | *If abnormal pre-transplant | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see comment |
| | BM biopsy – unilateral* Afte | | ransplant if patient is in CR, bone n | narrow is | recomme | nded onl | y as clinic | ally indic | ated. | |
| | Pathology | Clinical | | | | X | X | X | X | X |
| | Peripheral blood | T | | T | ı | ı | T | ı | | |
| | Chimerism (CD3+) | Clinical | *Days 56 and 180 only if <50%<br>on day 28 | X | *see<br>comment | X | *see<br>comment | X | | |
| | Chimerism (CD33+) | Clinical | | | | X | | | | |
| | Chimerism (NK CD56+) | Clinical | Optional for outside institutions | X | | | | | | |
| | Flow cytometry | Clinical | *If abnormal pre-transplant<br>AND bone marrow not done | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see comment |
| | Quantitative Ig Levels | Clinical | *If abnormal pre-transplant | | | *see<br>comment | *see<br>comment | *see<br>comment | *see<br>comment | *see comment |
| | B2 microglobulin | Clinical | *If abnormal pre-transplant | | | *see<br>comment | | | | |
| | LDH | Clinical | | | | X | X | X | X | X |
| | Additional research studies | Research –<br>Maloney Lab | | S | ee Table 8 | 3 for addit | ional perip | heral blood | l research s | tudies |
| | Imaging | | | | | | | | | |
| | CT of chest, abdomen, pelvis (neck if indicated) | Clinical | * Needed on Day 56 only if abnormal pre-transplant | | *see<br>comment | X | X | X | X | x |
| | <b>GVHD</b> evaluation | Clinical | | | | X | | | | |

**Table 8: Peripheral blood research studies** 

| Disease | Specimen | Research | Comment | | Days | | | | | Years | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 10 | 24 | 35 | 38 | 49 | 60 | 63 | 80 | 84 | 110 | 140 | 180 | 1 | 1.5 |
| CLL | T cell response | Research – | Only for pts. who have | | | | | | | | | X | | | X | X | |
| | studies | Maloney Lab | signed Consent D | | | | | | | | | | | | | | |
| | Polymorphism | Research – | For all Patients | | | | | | | | | x** | | | | | |
| | studies | Maloney Lab | For all Fatients | | | | | | | | | | | | | | |
| | Rituxan trough | Research – | For all Patients | X | X | | X | | | | | | | | | | |
| | levels* | Maloney Lab | For all Fatients | | | | | | | | | | | | | | |
| | Rituxan | Research – | For all Patients | | | | | | X | | | X | | | X | X | |
| | pharmacokinetics | Maloney Lab | roi an Patients | | | | | | | | | | | | | | |

<sup>\*</sup>Rituxan trough level on Day +10, Day +24, and Day +38 should be done immediately prior to rituximab dose \*\* Polymorphism studies is included with the T-cell response draw, no extra blood will be drawn

#### Additional information for research studies is as follows:

The blood obtained from the T cell response studies will be used as a source of donor T cells that recognize recipient minor histocompatibility or leukemia associated antigens. Briefly, mononuclear cells (PBMC) will be separated from the blood and aliquots will be cryopreserved. Aliquots of the posttransplant PBMC will be stimulated in vitro with irradiated (3300 rads) recipient PBMC and leukemia cells that were cryopreserved pretransplant (Section 10). The pretransplant recipient PBMC may be activated with CD40L prior to irradiation and use as stimulator cells. Cultures will be restimulated at weekly intervals, supplemented with IL-2 (10-20 U/ml), and assayed for cytolytic and proliferative responses against recipient PHA induced T cell blasts, EBV-LCL, CLL and fibroblasts and against donor target cells generated from the donor PBMC. Independent aliquots of cultures exhibiting responses to recipient CLL but not donor cells will be depleted of CD4<sup>+</sup> or CD8<sup>+</sup> T cells to determine the subset of cells mediating cytolytic activity. CD8<sup>+</sup> and CD4<sup>+</sup> T cells from T cell lines that are reactive with the patient CLL will be cloned by limiting dilution and the T cell clones will be further analyzed for specificity and function.

CD3<sup>+</sup> CD8<sup>+</sup> T cell clones will be tested for cytolytic activity against <sup>51</sup>Cr labeled donor and recipient B-LCL, PHA-induced T cell blasts, skin fibroblasts, and recipient CLL. T cell clones that lyse recipient hematopoietic cells but not dermal fibroblasts or donor hematopoietic cells (<5% lysis at E/T of 5:1) will be characterized for the class I MHC restricting allele using a panel of B-LCL from donors that are partially matched at HLA with the recipient. T cell clones specific for minor histocompatibility antigens expressed by CLL and presented by common class I alleles (e.g. HLA A0101, A0201, A0301, A1101, A2402, B0702, B0801, B3501, B4001, and B4402) will be preferentially selected for gene discovery using cDNA expression cloning or genetic linkage analysis.

The blood obtained for the polymorphism studies will be used to determine polymorphisms of FCyRIIIa and CD32 in comparison to pre-transplant polymorphisms.

### **Table 9: Additional Lab Instructions**

Note: All bone marrow tests are done on aspirate unless specifically identified as biopsy. Off-site providers may use local facilities for the tests. All research studies are for FHCRC patients only.

Volumes represent desired amounts.

| Specimen /<br>Test | Type | Instructions | Lab Name | Contact Information |
|---|---|---|---|---|
| one marrow | | | | |
| Chimerism | Clinical | 1-3mL bone marrow in green-top tube | Clinical Immunogenetics<br>Lab | Seattle Cancer Care Alliance (206) 288-7700 |
| Pathology (aspirate) | Clinical | 2mL bone marrow in EDTA formalin | SCCA Pathology Lab | Seattle Cancer Care Alliance (206) 288-1355 |
| Pathology (biopsy) | Clinical | 1cm bone marrow in formalin <b>OR</b> mounted in paraffin | SCCA Pathology Lab | Seattle Cancer Care Alliance (206) 288-1355 |
| Flow Cytometry | Clinical | 2mL bone marrow in green-top tube | UW Hematopathology Lab | Seattle Cancer Care Alliance (206) 288-7060 |
| Cytogenetics | Clinical | 3mL bone marrow in green-top tube | SCCA Cytogenetics Lab | Seattle Cancer Care Alliance (206) 288-1390 |
| FISH | Clinical | 2mL bone marrow in green-top tube | SCCA Cytogenetics Lab | Seattle Cancer Care Alliance (206) 288-1390 |
| eripheral blood | | | | |
| Chimerism<br>(CD3+), (CD33+)<br>NK(CD56+) | Clinical | 10mL blood in green-<br>top tube for Flow<br>sorting then to CIL | UW Hematopathology Lab,<br>routed to Clinical<br>Immunogenetics Lab | Mailstop G7-800 825 Eastlake Ave,<br>East Seattle, WA 98109<br>(206) 288-7060 |
| Flow Cytometry | Clinical | 10mL blood in green-<br>top tube<br>Label "protocol 1840) | UW Hematopathology Lab | Seattle Cancer Care Alliance (206) 288-7060 |
| Quantitative Ig<br>Levels | Clinical | 3mL blood in red-top tube | SCCA Alliance Lab | Seattle Cancer Care Alliance (206) 288-2057 |
| β-2 Microglobulin | Clinical | 3mL blood in red-top tube | UW Department of<br>Laboratory Medicine | University of Washington (800) 713-5198 |
| LDH | Clinical | 3mL blood in red-top tube | SCCA Alliance Lab | Seattle Cancer Care Alliance (206) 288-2057 |
| ZAP – 70 by Flow cytometry | Clinical | 5mL blood in green-<br>top tube | UW Hematopathology Lab | Mailstop G7-800 825 Eastlake Ave,<br>East Seattle, WA 98109<br>(206) 288-7060 |
| T cell response studies | Research | Pretransplant: 10mL<br>blood in red-top tube<br>and if Consent D is<br>signed: 40 mL in<br>green-top tube<br>Label "protocol 1840" | Maloney Lab | FHCRC D1-331<br>(206) 667-4260 |
| T cell response studies | Research | Posttransplant: 10mL<br>blood in red-top tube<br>and if Consent D is<br>signed: 30 mL in | Maloney Lab | FHCRC D1-331<br>(206) 667-4260 |

| Sp | pecimen / | Type | Instructions | Lab Name | Contact Information |
|---|---|---|---|---|---|
| | Test | | | | |
| | | | green-top tube<br>Label "protocol 1840" | | |
| Poly<br>studi | ymorphism<br>lies | Research | 10mL blood in green-<br>top tube (only if no T-<br>cell response drawn) | Maloney Lab | FHCRC D1-331<br>(206) 667-4260 |
| | ıxan trough | Research | 10mL blood in red-top | Maloney Lab | FHCRC D1-331 |
| leve | els | | tube | | (206) 667-4260 |
| Ritu | ıxan | Research | 10mL blood in red-top | Maloney Lab | FHCRC D1-331 |
| phar | rmacokinetics | | tube | | (206) 667-4260 |

Outside institutions may use VNTR analysis (sex- matched transplants) or sex chromosome FISH-analysis (sex-mismatched transplants) for PB chimerism analysis.

#### C. Donor Evaluation

- 1. Unrelated donors will undergo evaluation for allogeneic hematopoietic cell donation at the collection center by NMDP standard. The attending physician of the collection center will review the results of the donor evaluation.
- 2. A blood sample (10cc heparinized blood) from related and unrelated donors should be sent to the Maloney lab for determination of patient FCγRIIIa and CD32 polymorphisms prior to HCT.

#### 11. Drugs and toxicities

Detailed treatment-related adverse events will be reported using the adapted NCI Common Toxicity Criteria (Appendix P).

#### <u>A. TBI</u>

TBI will be given in one 200 cGy fraction from linear accelerator at a rate of 6 - 10 cGy/min. Dosimetry calculations are performed by the radiation therapist. At the dosage of TBI used in this protocol, patients have not experienced the adverse effects associated with myeloablative TBI such as fever, alopecia, parotitis, diarrhea, reversible skin pigmentation, and mucositis. Late effects are unknown but may include cataract formation, growth retardation, pulmonary damage, and carcinogenesis.

#### B. CSP

See section 9.E.1 for information about administration and dosage adjustments. Side effects are generally reversible and may include renal insufficiency and failure, hypomagnesemia, paresthesias, tremor, seizures, visual disturbances, paresis, disorientation, depression, confusion, somnolence, coma, nausea, hypertension, hemolytic-uremic syndrome, hyperglycemia, gynecomastia, and hypertrichosis.

#### C. MMF

Mycophenolate mofetil (MMF): is supplied in 250mg hard gelatin capsules. Capsules

may be stored at room temperature.

- 1. Precautions: MMF has not extensively been studied in patients after HSC transplantation. Previous clinical studies in patients after kidney transplantation suggested that the principal adverse reactions associated with the administration of MMF include leukopenia, sepsis, vomiting and diarrhea. Patients will be monitored for the development of these complications.
- 2. Adverse Events: Studies in solid organ transplant recipients suggest that MMF may be associated with vomiting, diarrhea, anemia, leukocytopenia and infection. In the setting of marrow transplantation, however, several etiologic factors may contribute to above mentioned symptoms. MMF has an increased incidence of digestive system adverse events, including GI tract ulceration, and hemorrhage (3% of patients receiving MMF). GI tract perforations have rarely been observed. Most patients in these studies were also on other drugs known to be associated with these complications. Up to 2% of patients receiving MMF for prevention of rejection developed severe neutropenia (ANC <500). The development of neutropenia may be related to MMF itself, concomitant medications, viral infections or some combination of these causes. MMF dose adjustments will be made if clinically indicated if, in the opinion of the attending physician, no other cause is thought to be causative for the abnormality. These adjustments should be discussed with the principal investigator. Dose administration and adjustments are described in Section 9.E.2.

#### D. Fludarabine

The dose of fludarabine used in this protocol is nonmyeloablative, but does cause significant immunosuppression. Fludarabine can lower the white blood cell count, in particular the CD4+ T-cells. The immunosuppression observed with the use of fludarabine increases the risk of infection, which can be life threatening.

#### E. Rituximab (rituxan)

Chemistry and Mechanism of Action. The rituximab antibody is a genetically engineered chimeric murine/human monoclonal antibody directed against the CD20 antigen found on the surface of normal and malignant B lymphocytes. The antibody is an IgG1 kappa immunoglobulin containing murine light- and heavy-chain variable region sequences and human constant region sequences. Rituximab is composed of two heavy chains of 451 amino acids and two light chains of 213 amino acids (based on cDNA analysis) and has an approximate molecular weight of 145 kD. Rituximab has a binding affinity for the CD20 antigen of approximately 8.0 nM.

Stability and Storage: Rituximab solutions for infusion are stable at 2° to 8° C (36° to 46° F) for 24 hours and at room temperature for an additional 12 hours. Rituximab vials should be protected from direct sunlight.

<u>Adverse Events</u>. The predominate toxicity of Rituximab is infusion related fever, chills, rigors, hypotension during the initial infusion. Premedication with acetaminophen and diphenhydramine may decrease the severity of the infusion complex. In the event of an

infusion reaction, the infusion should be slowed or stopped until the symptoms resolve or are successfully treated. The infusion should be restarted at one half the previous rate. Rapid depletion of B-lymphocytes may produce tumor lysis syndrome. Rituximab administration must be followed precisely. Patients on antihypertensive medications, or with prior history of cardiac arrhythmias may require additional clinical monitoring. Other adverse events of lowering of white blood cell or platelet counts, abnormal heart rhythms and/or congestive heart failure have also occurred. Rituximab treatment may involve risks to the embryo or fetus that are unknown and both women and men should practice contraception. Since Rituximab has only recently been approved by the FDA for use in the treatment of lymphoma, there is no long term information regarding toxicity. Very rarely, in about 1 per 1000 patients treated, severe reactions resulting in death have been associated with Rituximab infusion.

#### F. GVHD

For related recipients: In our phase I/II trials, grade II-IV acute GVHD associated with primary engraftment occurred in 49% of 192 evaluable patients, and the addition of fludarabine did not influence the incidence of grade II-IV or III-IV acute GVHD. Clinical extensive chronic GVHD occurred in 74 (67%) of 110 evaluable patients. Two of the first 10 evaluable patients receiving an HLA matched sibling donor transplant after conditioning with fludarabine and TBI on Protocol #1533 died of grade IV acute GVHD following discontinuation of CSP at day +56. Fifteen of 21 evaluable patients on Protocol #1533 had to restart immunosuppression after tapering off of CSP for clinically acute GVHD. The median day post-transplant for patients restarting immunosuppression for clinically acute GVHD was day +85 (range 65 to 107). These results prompted revision of the protocol (Protocol #1596) with extension of CSP to day +56 followed by a CSP taper that is adjusted based on the risk of relapse.

For unrelated recipients: After nonmyeloablative HCT from 10/10 HLA-antigen matched unrelated donors, the incidences of grades II, III and IV acute GVHD in patients who received G-PBMC grafts were 42%, 9% and 2% in protocol 1463 (with MMF q12hrs), and 39%, 10%, 2% in protocol 1641 (with MMF q8hrs) respectively. Acute GVHD has been readily controlled in most patients with high dose corticosteroids. Psoralen activated ultraviolet light (PUVA) has been required on occasion. Chronic extensive GVHD has occurred in 40 and 45% of patients in protocols 1463 and 1641, respectively.

#### 1. Diagnosis:

- a. On the day of GVHD evaluation, the diagnosis of acute or chronic GVHD will be made based on clinical criteria (Appendix F and G). Skin involvement will be assessed by biopsy and percentage of involved body surface area will be recorded in the medical record and CRF. GI symptoms suspicious for GVHD will be evaluated by biopsy as indicated.
- b. If manifestations of GVHD satisfy criteria for acute GVHD (Appendix F) and are not pathognomonic for chronic GVHD (Appendix G), for purposes of documentation and treatment, GVHD will be considered acute. The day post-transplant will not be used to discriminate acute from chronic GVHD. This

recommendation is based on the observation<sup>77</sup>[102] that the onset of acute GVHD can be delayed after nonmyeloablative conditioning.

c. If manifestations of GVHD are pathognomonic of chronic GVHD (Appendix G), for purposes of documentation and treatment, GVHD will be considered chronic even if concurrent manifestations satisfy criteria for acute GVHD (Appendix F).

#### 2. Recommended Treatment:

- a. Patients developing acute GVHD  $\geq$  grade II while on CSP taper or off immunosuppression:
  - i. CSP 5.0 mg/kg PO Q12 hrs. If there is concern of GI absorption use IV route (1.5 mg/kg Q12hrs).
  - ii. Prednisone (2 mg/kg/day) may be added at diagnosis or if the GVHD manifestations are mild when there is no response after 72 hours or if there is progression of GVHD during the 24 hours after the start of CSP. Patients who respond to steroids after 10 to 14 days of treatment, should begin a 6 week steroid taper See below section 2.b. for MMF and CSP taper recommendations.
  - iii. Patients may also be eligible for institutional trials of GVHD therapy.
- b. Patients who develop acute GVHD  $\geq$  grade II prior to day +56 for related and prior to day +100 for unrelated recipients:

#### Related recipients:

- i. Patients who develop acute GVHD  $\geq$  grade II prior to day +28 should receive prednisone (2 mg/kg/day) or intravenous equivalent. MMF should not be discontinued on day +28. If nausea and/or vomiting prevent the oral administration of MMF, MMF should be administered intravenously at 15 mg/kg q8hrs. Patients who respond to steroids after 10 to 14 days of treatment, should begin a 6 week steroid taper. MMF may be discontinued without taper, once prednisone has been tapered to a dose of 0.5 mg/kg/day.
- ii. Patients who develop acute GVHD ≥ grade II after day +27 should receive prednisone (2 mg/kg/day) or intravenous equivalent. MMF need not be restarted.
- iii. Patients may also be eligible for institutional trials of GVHD therapy.

#### **Unrelated recipients**:

i. Patients who develop acute GVHD ≥ grade II prior to day +40 should receive prednisone (2 mg/kg/day) or intravenous equivalent.

Patients who respond to steroids after 10 to 14 days of treatment, should begin a 6 week steroid taper. When steroids are tapered to 0.5 mg/kg p.o. q.d then an MMF taper should be initiated. In the absence of a GVHD flare, the MMF and prednisone tapers should continue until completion. The suggested sequence for tapering MMF and CSP is as follows: taper MMF over 1-2 months, then taper the Cyclosporine such that the completion of the taper is NOT prior to Day + 180 post transplant. If nausea and/or vomiting prevent the oral administration of MMF, MMF should be administered intravenously at 15 mg/kg TID.

- ii. Patients who develop acute GVHD ≥ grade II after day +90 should receive prednisone (2 mg/kg/day) or intravenous equivalent. MMF need not be restarted.
- iii. Patients may also be eligible for institutional trials of GVHD therapy.
- c. Patients with clinical extensive chronic GVHD: CSP 5.0 mg/kg PO Q12hrs and prednisone 1 mg/kg qd or eligible protocols at the time. The patient should receive antibiotic prophylaxis with daily double strength Bactrim.
- d. Patients off immunosuppression who develop concurrent manifestations of GVHD that satisfy criteria for ≥ grade II acute GVHD (e.g. erythematous rash, diarrhea, hyperbilirubinemia) **and** are pathognomonic of clinical extensive chronic GVHD (e.g. lichenoid oral changes, ocular sicca, scleroderma, bronchiolitis obliterans, contractures), should receive prolonged immunosuppressive therapy similar to that for chronic extensive GVHD.

#### G. Myelosuppression

Grade IV myelosuppression will be defined as a decrease in ANC to  $\leq 500/\mu L$  and/or platelet count to  $\leq 20,000/u L$ . If myelosuppression occurs, a bone marrow aspirate and biopsy should be performed in the proper clinical circumstances to exclude disease progression or graft rejection. Samples should be sent for chimerism analysis by a DNA-based assay that compares the profile of amplified fragment length polymorphisms (ampFLP) (or FISH studies or VNTR). Myelosuppression may occur in this patient population for a number of reasons such as direct toxic effect of drugs, rejection, or relapse.

Patients with myelosuppression may be managed as follows:

- 1. <u>Suspected MMF toxicity</u>: refer to sections **9.E.2.f** <u>Guidelines for MMF dose adjustment</u> for management recommendations.
- 2. <u>Suspected ganciclovir toxicity</u>: consider changing to foscarnet.

- 3. Patients who are > 21 days after HCT with a hypoplastic marrow and an ANC of ≤750/uL may receive G-CSF 5µg/kg/day S.C.
- 4. Thrombocytopenic patients will receive platelet transfusion as per standard care.

#### 12. Toxicity Reporting Guidelines

Detailed treatment-related adverse events will be reported using the adapted NCI Common Toxicity Criteria (Appendix P).

#### 13. Records

Clinical records will be maintained as confidentially as possible by all collaborating institutions. Collection of Case Report Forms (CRF) at standard intervals is the primary method of collecting data from collaborating centers. Clinical Statistics at FHCRC maintains a patient database to allow storage and retrieval of patient data collected from a wide variety of sources. The principal investigator will ensure that data collected conform to all established guidelines for coding collection, key entry and verification. These data are then entered into a secure dedicated database operated by a data manager. Any publication or presentation will refer to patients by a unique patient number and not by name to assure patient confidentiality. The licensed medical records department, affiliated with the institution where the patient receives medical care, maintains all original inpatient and outpatient chart documents.

At the FHCRC, patient research files are kept in a locked room. They are maintained by the FHCRC data collection staff that is supervised by an A.R.T. Access is restricted to personnel authorized by the Division of Clinical Research.

#### Collection of Survival and Disease Response Data

Centers enrolling patients will complete case report forms within 120 days of HCT that detail events occurring within the 100 days after HCT (Appendix M). The case report form provides detailed descriptions of the transplantation procedure, disease response, and complications. Detailed treatment-related adverse events will be reported using the NCI Common Toxicity Criteria (Appendix P). The coordinating center will contact subjects when they return to the HCT center for routine HCT follow-up at 3, 6, 12 and 24 months to ascertain the patient's disease status and survival. Referring physicians are required to report the date and cause of death within 48 hours of occurrence. Supporting medical records must be available upon request to substantiate data on the case report forms. Death information including date and cause will be reviewed from these medical records, and will be confirmed by death certificate.

#### 14. Statistical Consideration and Criteria of Termination of Study

The primary objective of this protocol is to estimate survival using allogeneic HCT from related or unrelated donors after nonmyeloablative conditioning and peri-transplant Rituximab in patients with advanced CLL, and to gain a preliminary indication as to whether survival is improved compared to treatment with conventional salvage therapies. The primary endpoint will be survival at 18 months. The 18 months time point is chosen because prior experience with HCT indicates that survival

reaches a relative plateau by that time, and thus offers an endpoint that can be evaluated somewhat more rapidly than 2 year survival. The estimated 18 months survival with standard treatment (Campath-1H) from historical patients is approximately 0.45. This treatment approach will be deemed promising for further study if we can achieve reasonable confidence that survival exceeds 0.45. Reasonable confidence will be taken to mean that the lower limit of a one-sided 90% confidence interval for the true survival fraction at 18 months is greater than 0.45.

Protocol 1840 has enrolled 14 patients so far before the current changes. We anticipate enrolling eighty new patients in eight years from the data when peri-transplant Rituximab was added to the inclusion criteria. The total targeted accrual for the protocol will be 94 but only the last 80 patients will be evaluated for the study objectives.

Eighty new patients will be evaluated; thus the above criterion will be met if 43 or more of 80 patients are alive at 18 months, then we will be at least 90% confident that the true survival rate exceeds 0.45. We assume based on our prior studies that we will achieve 100% ascertainment of this endpoint in these closely followed patients. The probability of such a favorable outcome is 89%, if the true survival fraction at 18 months is 60% and 63% if the true fraction is 55%. Our current experience with non-myeloablative HCT from unrelated donor in CLL indicates that this is a reasonable expectation.

A secondary objective of this protocol is to test the hypothesis that pre- and post-transplant rituximab will reduce the incidence of chronic GVHD. Therefore, the incidence of chronic GVHD in the study population will be compared to that seen in our published historical controls receiving non-myeloablative allogeneic HCT without rituximab. Enrollment of a total of 80 new patients will yield 90% power to detect an absolute decrease of 15% in the risk of chronic GVHD ( $45\% \rightarrow 30\%$ ), and 64% power to detect a 10% absolute risk reduction for chronic GVHD ( $45\% \rightarrow 35\%$ ), at the 1-sided 0.1 level of significance.

#### Criteria for Termination of Study

This will be a single stage trial of a single cohort of 80 patients. However, safety stopping rules will be imposed for acute grade IV GHVD at anytime that precludes the diagnosis of chronic GVHD, and transplant-related mortality at 200 days. If sufficient evidence exists to suggest that the true rate of transplant related mortality at day 200 exceeds 0.30, or the true rate of grade IV acute GVHD exceeds 0.10, then the protocol will be terminated. Sufficient evidence will be taken to be any observed rate for which the lower limit of a one-sided 80% confidence interval exceeds the target rate.

Therefore, **stopping rules** will be imposed for:

- Transplant-related mortality at day 200 > 30%
- Grade IV acute GVHD >10% at anytime that precludes the diagnosis of chronic GVHD

These rules will be evaluated after every tenth patient is evaluable for the endpoint in question. Operationally, this will occur:

- Transplant-related mortality (by day 200. 30% threshold): 3/5, 5/10, 7/15, 9/20, 10/25, 12/30, 14/35, 15/40, 19/50, 22/60, 25/70, 28/80
- Grade IV acute GVHD (10% threshold) at anytime that precludes the diagnosis of chronic GVHD: 2/5, 3/10, 3/15, 4/20, 5/25, 5/30, 6/35, 7/40, 8/50, 9/60, 10/70, 11/80.

These stopping criteria are listed in Table 10. Patients may continue to be enrolled pending the evaluation of these stopping rules after every tenth patient, but the outcome in subsequent patients cannot be used to override a stopping rule triggered in an earlier number. The operating characteristics of these stopping rules are given in Table 11.

Table 10. Criteria for stopping trial based on day 200 evaluation

| Number of patients enrolled | Number of Patients with<br>Grade IV GVHD | Number of Patients<br>Experiencing day-200 TRM |
|---|---|---|
| 10 | 3 | 5 |
| 20 | 4 | 9 |
| 30 | 5 | 12 |
| 40 | 7 | 15 |
| 50 | 8 | 19 |
| 60 | 9 | 22 |
| 70 | 10 | 25 |
| 80 | 11 | 28 |

Table 11. Operating characteristics of stopping rules

| | Day 200 TRM | | | acute GVHD at and acute GVHD at an acute GVHD at acute GVHD | • |
|---|---|---|---|---|---|
| True rate of event | Probability of stopping* | Average N at stopping* | True rate of event | Probability of stopping* | Average N at stopping* |
| 0.35 | 70% | 46 | 0.15 | 77% | 44 |
| 0.40 | 91% | 32 | 0.20 | 96% | 28 |
| 0.45 | 98% | 23 | 0.25 | >99% | 19 |

#### 15. Targeted Planned Enrollment Table

Table 12 shows the anticipated distribution of subjects based on data from the US Census Bureau and the age-adjusted incidence of CLL in populations in the United States from SEER.

**Table 12. Targeted Planned Enrollment Table** 

| TARGETED / PLANNED ENROLLMENT: Number of Subjects | | |
|---|---|---|
| Sex / Gender | | |
| Females | Males | Total |
| 1 | 2 | 3 |
| 32 | 45 | 77 |
| 33 | 47 | 80 |
| | 1 | |
| | 1 | 1 |
| 1 | 1 | 2 |
| 1 | 1 | 2 |
| 31 | 44 | 75 |
| 33 | 47 | 80 |
| | Females 1 32 33 1 1 1 1 31 | Sex / Gender |

<sup>\*</sup>The "Ethnic Category Total of All Subjects" must be equal to the "Racial Categories Total of All Subjects". This is the targeted planned enrollment after adding peri-transplant rituximab and allowing grafts from related or unrelated HLA-matched donors).

#### 16. Data Safety Monitoring Board and Adverse Events Reporting

#### A. Monitoring the progress of trials and the safety of participants

This protocol is a multi-institutional clinical trial that is monitored by the principal investigators (PI), Drs. Sorror and Dr. Maloney, with oversight by Dr. Sandmaier, and Dr. Storb, a Data Safety and Monitoring Board (DSMB), the Protocol and Data Monitoring Committee (PDMC) and the Institutional Review Board (IRB). The PI reviews outcome data with the protocol mentors for each local individual patient on a weekly basis at a minimum of 3 months after HCT and the updated data are presented at Mixed Chimerism Meetings that includes peer review by co-investigators.

Adverse events are reported to the trial coordinator, one of the study nurses, or directly to the PI. The trial coordinators at collaborating centers or the local PIs will fax an official report of a serious adverse event to the coordinating center (FHCRC) within ten days. The serious adverse event report is reviewed by Dr. Sorror and Dr. Maloney. If the serious adverse event meets the FHCRC and/or NCI criteria for reporting then an official signed report is submitted to the FHCRC Institutional Review Office (IRO). All deaths, regardless of the cause, are reported to the IRB. This protocol has a dedicated independent DSMB responsible for monitoring patient safety on this clinical trial. The DSMB meets twice a year and all outcome data is reviewed including all adverse events reported to the coordinating center (FHCRC) along with those officially reported to the FHCRC IRO. The DSMB confirms whether or not the trial has met any stopping rules and reviews any patient safety problems necessitating discontinuation of the trial. A report from the DSMB is submitted to the FHCRC IRB as well as the trial coordinators/local PIs of this protocol. Furthermore, the FHCRC also has a PDMC that reviews the progress of the protocol with respect to the monitoring plan at the time of each annual renewal. An initial IRB review and approval will occur before any patients are enrolled in the trial and an annual IRB review and approval also is required. The DSMB will discontinue the review of outcomes when this protocol is closed to accrual.

With respect to safety, all patients are monitored for the development of GVHD, myelosuppression, infections, and organ-specific toxicities. All patients, regardless of diagnosis, will be considered in the safety analysis. Because of the older age profile of the patients, complications of HCT, GVHD and infections, may be less well tolerated than patients on other protocols. These events will be closely monitored and severity of GVHD graded. Formal stopping rules for TRM, defined as death before day 100 not related to progression of disease, will be closely monitored and stopping rules are provided above in **section 14** Statistical Consideration and Criteria Termination of Study. This endpoint encompasses serious problems associated with the potential complications of severe GVHD, infections, and rejection.

Flow of information concerning clinical trial participants originates with the clinicians and nurses in the clinic or referring clinicians at other institutions and is transmitted to the Trial coordinator. At the FHCRC, health care providers and rotating attending physicians assess patients and record their observations regarding toxicity and response outcomes in the medical record. This documentation is extracted by the study nurse within 140 days +/- after HCT via chart review and collection of copies of source documents and entered into a hard copy or electronic Case Report Form (CRF). Drs. Sorror and Maloney will review the official CRF and primary source documents. When the CRFs are verified, they are signed by PI. Thus, multiple health care providers provide independent

observations and participate in monitoring this trial. Drs. Sorror or Maloney may be a clinician for some patients entered on this trial. However, assessments are the sum total of the primary health care provider (fellow or physician assistant), floor or outpatient nurse and the PI or other attending clinician involved with the patient averting possible conflict of interest having the PI as the attending clinician for protocol patients. In addition, direct oversight from other PIs including Dr. Sandmaier and Dr Storb, will further minimize potential conflict of interest inherent in the PI serving as primary study monitor. If determination of adverse events is controversial, coinvestigators will convene on an ad hoc basis as necessary to review the primary data and render a decision.

This protocol is a multi-institutional protocol and all collaborating centers sign an agreement with the FHCRC stating that data generated from patients from the protocol will be reported accurately in a timely manner to the FHCRC. All centers have an IRB that review the protocol and that the local PIs contact when an adverse event on the protocol occurs. Most of the centers have internal auditing mechanisms that assure accurate assessment of clinical outcomes. Clinical outcome data are summarized and transmitted from collaborating centers as CRFs. When possible, primary source documents regarding patient outcomes are collected with patients' names removed and replaced by Unique Patient Numbers (UPNs). The CRFs are generated from the collaborating centers at defined time points (100 days, 6 months, and yearly). The local PI will review the official CRF and primary source documents. When the CRFs are verified, they are signed by the local PI and the data are entered into a central database managed by the Trial Coordinator.

#### B. Plans for assuring compliance with requirements for reporting adverse events

The adverse event reporting in this multi-institution clinical trial will follow the FHCRC Guidelines for serious adverse event (SAE) reporting. The FHCRC guidelines have been expanded to give further details on what events meet expedited reporting requirements for consistency in SAE reporting across the centers. Definitions of particular events that require reporting are in Appendix P. These guidelines (attached in Appendix I.) detail the expedited reporting requirements. definitions of particular events. The trial coordinators at collaborating centers or the local PIs will fax an official report of an SAE to the coordinating center (FHCRC) within ten days. The SAE report is reviewed by Dr. Maloney and Dr. Sorror. If the SAE meets the FHCRC criteria for expedited reporting then an official signed report is submitted to the FHCRC Institutional Review Office (IRO) within 10 days. All deaths, regardless of the cause, are reported to the IRB. For patients being cared for at the FHCRC, health care providers communicate with the PI, trial coordinator or research nurses as events occur triggering subsequent reporting. For patients not being cared for at FHCRC the outside facilities communicate with the PI, trial coordinator, or research nurse for these reporting purposes. All other deaths and expected serious adverse events are reported to the IRB at the time of annual renewal and at the biannual mixed chimerism meeting. The PI for a study is responsible for this reporting and the IRO assures adverse event reporting on an annual basis. The PI in the annual application for grant continuation will summarize reports of toxicities. Furthermore, an additional safeguard for adverse event analysis and reporting in this protocol is provided by stopping rules. All collaborating PIs have fulfilled all NIH requirements for training in human subjects' protection.

C. Plans for assuring that any action resulting in a temporary or permanent suspension of an NCI-funded clinical trial is reported to the NCI grant program director responsible for the grant

This clinical research trial uses commercial agents and there is no associated Investigational New Drug (IND) or Investigational Device Exemption (IDE). Any temporary or permanent suspension, as determined by the PI, IRB, or PDMC, of this clinical research trial will be reported to the NCI grant program director by the PI.

#### D. Plans for assuring data accuracy and protocol compliance

Collaborating sites send signed consents, eligibility forms, and CRFs with source documents demonstrating eligibility, treatment, and serious adverse events (if applicable) to the study staff. These are reviewed for eligibility, adherence to the protocol, accuracy, and completeness by the study staff. Queries are sent to the collaborating investigators if CRFs are inaccurate or incomplete.

The study is monitored under the FHCRC Monitoring Plan. The FHCRC Data and Safety Monitoring Plan details the full scope and extent of monitoring and provides for immediate action in the event of the discovery of major deviations.

#### References

1. Hager EB, Mannick JA, Thomas ED, Ferrebee JW. Dogs that survive "lethal" exposures to radiation. Radiat Res 14: 192-205, 1961.

**Reference ID: 44** 

- 2. Mannick JA, Lochte HL, Jr., Thomas ED, Ferrebee JW. In vitro and in vivo assessment of the viability of dog marrow after storage. Blood 15: 517-524, 1960.

  Reference ID: 43
- 3. Dreger P, Montserrat E. Autologous and allogeneic stem cell transplantation for chronic lymphocytic leukemia (Review). Leukemia 16: 985-992, 2002. **Reference ID:** 24477
- 4. Rai KR, Peterson BL, Appelbaum FR, Kolitz J, Elias L, Sheperd L, Hines J, Threatte GA, Larson RA, Cheson BD, Schiffer CA. Fludarabine compared with chlorambucil as primary therapy for chronic lymphocytic leukemia. N Engl J Med 343: 1750-1757, 2000.

Reference ID: 17998

- 5. Mannick JA, Lochte HL, Jr., Ashley CA, Thomas ED, Ferrebee JW. A functioning kidney homotransplant in the dog. Surgery 46: 821-828, 1959.

  Reference ID: 31
- 6. Thomas ED, Collins JA, Kasakura S, Ferrebee JW. Lethally irradiated dogs given infusions of fetal and adult hematopoietic tissue. Transplantation 1: 514-520, 1963.

  Reference ID: 64
- 7. Byrd JC, Rai K, Peterson BL, Appelbaum FR, Morrison VA, Kolitz JE, Shepherd L, Hines JD, Schiffer CA, Larson RA. Addition of rituximab to fludarabine may prolong progression-free survival and overall survival in patients with previously untreated chronic lymphocytic leukemia: an updated retrospective comparative analysis of CALBG 9712 and CALBG 9011. Blood 105: 49-53, 2005.

- 8. Hillmen P. Advancing therapy for chronic lymphocytic leukemia--the role of rituximab (Review). Semin Oncol 31 (Suppl 2): 22-26, 2004.

  Reference ID: 24767
- 9. Gregory R, Ewing PL, Duff-White V, Thomas ED. Effect of sodium pyruvate on the rate of metabolism of ethyl alcohol. Proc Soc Exp Biol Med 54: 209-211, 1943.

  Reference ID: 3
- Keating MJ, O'Brien S, Lerner S, Koller C, Beran M, Robertson LE, Freireich EJ, Estey E, Kantarjian H. Long-term follow-up of patients with chronic lymphocytic leukemia FHCRC Current Version 1/13/2016

(CLL) receiving fludarabine regimens as initial therapy. Blood 92: 1165-1171, 1998

Reference ID: 19933

11. Thomas ED. In vitro studies of erythropoiesis. II. The effect of anoxia on heme synthesis. Blood 6: 612-615, 1955.

Reference ID: 12

12. LaForet MT, Thomas ED. The effect of cobalt on heme synthesis by bone marrow in vitro. J Biol Chem 218: 595-598, 1956.

Reference ID: 14

- 13. Ferrebee JW, Thomas ED. Radiation injury and marrow replacement: Factors affecting survival of the host and the homograft. Ann Intern Med 49: 987-1003, 1958.

  Reference ID: 21
- Lochte HL, Jr., Ferrebee JW, Thomas ED. In vitro studies on the preservation of marrow cells in glycerol at low temperatures. J Lab Clin Med 53: 117-126, 1959.
   Reference ID: 24
- 15. Thomas ED, Kasakura S, Cavins JA, Swisher SN, Ferrebee JW. Significance of blood groups in homotransplantation of marrow in the dog. Ann NY Acad Sci 120: 362-366, 1964.

**Reference ID: 71** 

16. Blumenstock DA, Collins JA, Hechtman HB, Hosbein DJ, Lempert N, Thomas ED, Ferrebee JW. Lung transplantation in the dog. Ann NY Acad Sci 120: 677-688, 1964.

Reference ID: 72

17. Thomas ED, Epstein RB. Bone marrow transplantation in acute leukemia. Cancer Res 25: 1521-1524, 1965.

Reference ID: 75

18. Byrd JC, Murphy T, Howard RS, Lucas MS, Goodrich A, Park K, Pearson M, Waselenko JK, Ling G, Grever MR, Grillo-Lopez AJ, Rosenberg J, Kunkel L, Flinn IW. Rituximab using a thrice weekly dosing schedule in B-cell chronic lymphocytic leukemia and small lymphocytic lymphoma demonstrates clinical activity and acceptable toxicity. J Clin Oncol 19: 2153-2164, 2001.

Reference ID: 19937

19. Esteve J, Montserrat E, Dreger P, Meloni G, Pavletic S, Catovsky D, Dearden C, Scimè R, Sutton L, Michallet M, Desablens B, Kimby E, Coiffier B, Brunet S, Sanz MA, Besalduch J, Caballero D, Juliusson G, Conde E, del Potro E, Schmitz N. Stem cell transplantation (SCT) for chronic lymphocytic leukemia (CLL): outcome and prognostic factors after autologous and allogeneic transplants. Blood 98 (Part 1):

FHCRC Current Version 1/13/2016

482a, #2013, 2001.(Abstract)

Reference ID: 24525

20. Anasetti C, Etzioni R, Petersdorf EW, Martin PJ, Hansen JA. Marrow transplantation from unrelated volunteer donors. Annu Rev Med 46: 169-179, 1995.

**Reference ID: 9760** 

21. Anasetti C, Howe C, Petersdorf EW, Martin PJ, Hansen JA. Marrow transplants from HLA-matched unrelated donors: an NMDP update and the Seattle experience. Bone Marrow Transplant 13: 693-695, 1994.

Reference ID: 8994

22. Small TN, Papadopoulos EB, Boulad F, Black P, Castro-Malaspina H, Childs BH, Collins N, Gillio A, George D, Jakubowski A, Heller G, Fazzari M, Kernan N, Mackinnon S, Szabolcs P, Young JW, O'Reilly RJ. Comparison of immune reconstitution after unrelated and related T-cell-depleted bone marrow transplantation: effect of patient age and donor leukocyte infusions. Blood 93: 467-480, 1999.

Reference ID: 18623

- 23. Sorror ML, Maris MB, Sandmaier BM, Storer BE, Stuart MJ, Hegenbart U, Agura E, Chauncey TR, Leis J, Pulsipher M, McSweeney P, Radich JP, Bredeson C, Bruno B, Langston A, Loken MR, Al-Ali H, Blume KG, Storb R, Maloney DG. Hematopoietic cell transplantation after nonmyeloablative conditioning for advanced chronic lymphocytic leukemia. J Clin Oncol 23: 3819-3829, 2005.

  Reference ID: 26766
- 24. Sorror ML, Storer BE, Sandmaier BM, Maris M, Shizuru J, Maziarz R, Agura E, Chauncey TR, Pulsipher MA, McSweeney PA, Wade JC, Bruno B, Langston A, Radich J, Niederwieser D, Blume KG, Storb R, Maloney DG. Five-year follow-up of patients with advanced chronic lymphocytic leukemia treated with allogeneic hematopoietic cell transplantation after nonmyeloablative conditioning. J Clin Oncol 26: 4912-4920, 2008.

**Reference ID:** 34579

25. Thomas ED, Ferrebee JW. Transplantation of marrow and whole organs: Experiences and comments. Can Med Assoc J 86: 435-444, 1962.

Reference ID: 50

- 26. Thomas ED, Collins JA, Herman EC, Jr., Ferrebee JW. Marrow transplants in lethally irradiated dogs given methotrexate. Blood 19: 217-228, 1962.

  Reference ID: 49
- 27. Thomas ED, Ferrebee JW. Prolonged storage of marrow and its use in the treatment of radiation injury. (Short Communication). Transfusion 2: 115-117, 1962.

28. Lochte HL, Thomas ED, Truitt P. The nitrogen compounds in petroleum distillates. XXV. Isolation and identification of 3- and 4-cyclopentylpyridines from California petroleum. J Am Chem Soc 66: 550-552, 1944.

Reference ID: 4

29. Ferrebee JW, Thomas ED. Present status of bone marrow transplantation. Pediatr Clin North Am 9: 851-853, 1962.

**Reference ID: 55** 

- 30. Blumenstock DA, Collins JA, Hechtman HB, Thomas ED, Ferrebee JW. Functioning homografts of lung in dogs. Ann NY Acad Sci 99: 882-890, 1962.

  Reference ID: 56
- 31. Lochte HL, Jr., Levy AS, Guenther DM, Thomas ED, Ferrebee JW. Prevention of delayed foreign marrow reaction in lethally irradiated mice by early administration of methotrexate. Nature 196: 1110-1111, 1962.

  Reference ID: 57
- 32. Cavins JA, Kasakura S, Thomas ED, Ferrebee JW. Recovery of lethally irradiated dogs following infusion of autologous marrow stored at low temperature in dimethyl-sulphoxide. Blood 20: 730-734, 1962.

  Reference ID: 58
- 33. Thomas ED, Baker JA, Ferrebee JW. The effect of methotrexate on the production of antibodies against attenuated distemper virus in the dog. J Immunol 90: 324-328, 1963.

- 34. Hechtman HB, Blumenstock DA, Thomas ED, Ferrebee JW. Organ transplants in dogs after cross-circulation, chemotherapy and radiation. Surgery 52: 810-818, 1962.

  Reference ID: 60
- 35. Hechtman HB, Blumenstock DA, Thomas ED, Ferrebee JW. Prolongation of canine skin homografts by antimetabolites. Surg Forum 13: 55-57, 1962.

  Reference ID: 59
- 36. Thomas ED, Lochte HL, Jr., Stohlman F, Jr. Attempts to develop an in vitro system for the assay of erythropoietin. J Lab Clin Med 55: 311-318, 1960.

  Reference ID: 34
- 37. Thomas ED, Lochte HL, Jr., Greenough WB, III, Wales M. <u>In vitro</u> synthesis of foetal and adult haemoglobin by foetal haematopoietic tissues. Nature 185: 396-397, 1960. **Reference ID:** 36

- 38. Lochte HL, Jr., Kasakura S, Karetzky M, Ferrebee JW, Thomas ED. Infusion of marrow in the mouse and dog after Thio-TEPA. Blood 21: 424-428, 1963.

  Reference ID: 62
- 39. Ferrebee JW, Thomas ED. Transplantation of marrow in man. Arch Intern Med 106: 523-531, 1960.

**Reference ID: 39** 

40. Lochte HL, Crouch WW, Thomas ED. The nitrogen compounds in petroleum distillates. XXIV. Isolation and identification of  $C_{11}H_{17}N$  base from California petroleum. J Am Chem Soc 64: 2753-2755, 1942.

Reference ID: 1

- 41. Finch CA, Hegsted M, Kinney TD, Thomas ED, Rath CE, Haskins D, Finch S, Fluharty RG. Iron metabolism. The pathophysiology of iron storage. Blood 5: 983-1008, 1950. **Reference ID:** 7
- 42. Thomas ED. Transplantation of bone marrow. In: Proc. N.Y. State Assoc. Public Health Lab., p. 11-14, 1958.

  Reference ID: 22
- 43. Cavins JA, Scheer SC, Thomas ED, Ferrebee JW. The recovery of lethally irradiated dogs given infusions of autologous leukocytes preserved at -80 C. Blood 23: 38-43, 1964. **Reference ID:** 69
- 44. Thomas ED, Plain GL, Cavins JA, Blumenstock DA. Leukokinetics in dogs given supralethal irradiation with or without a graft of marrow. Ann NY Acad Sci 113: 1020-1032, 1964.

Reference ID: 68

- 45. Thomas ED, Plain GL, Graham TC, Ferrebee JW. Long-term survival of lethally irradiated dogs given homografts of bone marrow. (Brief Note). Blood 23: 488-493, 1964. **Reference ID:** 70
- 46. Thomas ED, Hershey FB, Abbate AM, Loofbourow JR. Chromatographic determination of nucleotides in the suspending medium from irradiated yeast. J Biol Chem 196: 575-582, 1952.

- 47. Blumenstock DA, Collins JA, Thomas ED, Ferrebee JW. Homotransplantation of the lung in dogs treated with methotrexate. Surg Forum 12: 121-122, 1961.

  Reference ID: 47
- 48. Garcia Manero G, O'Brien S, Cortes J, Faderl S, Giles F, Albitar M, Lerner S, Kantarjian H, Keating M. Update of results of the combination of fludarabine, cyclophosphamide and rituximab for previously treated patients with chronic lymphocytic leukemia.

Blood 98 (Part 1): 633a, #2650, 2001.(Abstract) **Reference ID:** 24547

- 49. Horn PA, Neff T, Peterson LJ, Morris JC, Thomasson BM, Sandmaier BM, Kiem H-P. Efficient lentiviral gene transfer to canine hematopoietic repopulating cells using an overnight transduction protocol. Blood 100 (Part 1): 184a, #687, 2002.(Abstract) **Reference ID:** 23068
- 50. Miller AD. PA317 retrovirus packaging cells. Mol Ther 6: 572-575, 2002. **Reference ID:** 23069
- 51. Mehal WZ, Azzaroli F, Crispe IN. Immunology of the healthy liver: old questions and new insights (Review). Gastroenterology 120: 250-260, 2001.

  Reference ID: 23079
- 52. Thomas ED, Motulsky AG, Walters DH. Homozygous hemoglobin C disease. Report of a case with studies on the pathophysiology and neonatal formation of hemoglobin C. Am J Med 18: 832-838, 1955.

  Reference ID: 10
- 53. Gopal AK, Gooley TA, Maloney DG, Petersdorf SH, Eary JF, Rajendran JG, Bush SA, Durack LD, Golden J, Martin PJ, Matthews DC, Appelbaum FR, Bernstein ID, Press OW. High-dose radioimmunotherapy versus conventional high-dose therapy and autologous hematopoietic stem cell transplantation for relapsed follicular non-Hodgkin lymphoma: a multivariable cohort analysis. Blood 102: 2351-2357, 2003. **Reference ID:** 23071
- 54. Ormo M, Cubitt AB, Kallio K, Gross LA, Tsien RY, Remington SJ. Crystal structure of the Aequorea victoria green fluorescent protein. Science 273: 1392-1395, 1996.

  Reference ID: 23073
- 55. Hegenbart U, Lange T, Leiblein S, Poenisch W, Deininger MW, Edelmann J, Kamprath F, Holler E, Forman S, Niederwieser D, Storb R. Successful treatment of severe paroxysmal nocturnal hemoglobinuria (PNH) with allogeneic hematopoietic stem cell transplantation (HSCT) from unrelated donors after minimal conditioning. Blood 98 (Suppl. 1): 675a, #2827, 2001.(Abstract)

  Reference ID: 23072
- 56. Stewart AK, Vescio R, Schiller G, Ballester O, Noga S, Rugo H, Freytes C, Stadtmauer E, Tarantolo S, Sahebi F, Stiff P, Meharchard J, Schlossman R, Brown R, Tully H, Benyunes M, Jacobs C, Berenson R, White M, DiPersio J, Anderson KC, Berenson J. Purging of autologous peripheral-blood stem cells using CD34 selection does not improve overall or progression-free survival after high-dose chemotherapy for multiple myeloma: results of a multicenter randomized controlled trial. J Clin Oncol 19: 3771-3779, 2001.

- 57. Crippa F, Holmberg L, Carter RA, Hooper H, Marr KA, Bensinger W, Chauncey T, Corey L, Boeckh M. Infectious complications after autologous CD34-selected peripheral blood stem cell transplantation. Biol Blood Marrow Transplant 8: 281-289, 2002. Reference ID: 20274
- 58. Korbling M, Katz RL, Khanna A, Ruifrok AC, Rondon G, Albitar M, Champlin RE, Estrov Z. Hepatocytes and epithelial cells of donor origin in recipients of peripheral-blood stem cells. N Engl J Med 346: 738-746, 2002. Reference ID: 23075
- 59. Ferrebee JW, Lochte HL, Jr., Jaretzki A, III, Sahler OD, Thomas ED. Successful marrow homograft in the dog after radiation. Surgery 43: 516-520, 1958. Reference ID: 19
- 60. Storb R. Non-myeloablative allogeneic transplantation state-of-the-art. Pediatr Transplant 8 (Suppl. 5): 12-18, 2004. Reference ID: 23083
- 61. Michallet M, Archimbaud E, Bandini G, Rowlings PA, Deeg HJ, Gahrton G, Montserrat E, Rozman C, Gratwohl A, Gale RP. HLA-identical sibling bone marrow transplantation in younger patients with chronic lymphocytic leukemia. European Group for Blood and Marrow Transplantation and the International Bone Marrow Transplant Registry. Ann Intern Med 124: 311-315, 1996. Reference ID: 11325
- 62. Thomas ED, Ashley CA, Lochte HL, Jr., Jaretzki A, III, Sahler OD, Ferrebee JW. Homografts of bone marrow in dogs after lethal total-body radiation. Blood 14: 720-736, 1959. Reference ID: 26
- 63. Thomas ED, Lochte HL, Jr., Ferrebee JW. Irradiation of the entire body and marrow transplantation: Some observations and comments. Blood 14: 1-23, 1959. Reference ID: 23
- 64. Storb R. History of pediatric stem cell transplantation. Pediatr Transplant 8 (Suppl. 5): 5-11, 2004. Reference ID: 23084
- 65. Schetelig J, Thiede C, Bornhauser M, Schwerdtfeger R, Kiehl M, Beyer J, Sayer HG, Kroger N, Hensel M, Scheffold C, Held TK, Hoffken K, Ho AD, Kienast J, Neubauer A, Zander AR, Fauser AA, Ehninger G, Siegert W. Evidence of a graftversus-leukemia effect in chronic lymphocytic leukemia after reduced-intensity conditioning and allogeneic stem-cell transplantation: the Cooperative German Transplant Study Group. J Clin Oncol 21: 2747-2753, 2003. Reference ID: 24027

FHCRC Current Version 1/13/2016

- 66. Dreger P, Brand R, Hansz J, Milligan D, Corradini P, Finke J, Deliliers GL, Martino R, Russell N, van Biezen A, Michallet M, Niederwieser D, Chronic Leukemia Working Party of the EBMT. Treatment-related mortality and graft-versus-leukemia activity after allogeneic stem cell transplantation for chronic lymphocytic leukemia using intensity-reduced conditioning (Review). Leukemia 17: 841-848, 2003.

  Reference ID: 24025
- 67. Storb R, Yu C, Wagner JL, Deeg HJ, Nash RA, Kiem H-P, Leisenring W, Shulman H. Stable mixed hematopoietic chimerism in DLA-identical littermate dogs given sublethal total body irradiation before and pharmacological immunosuppression after marrow transplantation. Blood 89: 3048-3054, 1997.

  Reference ID: 12941
- 68. McSweeney PA, Niederwieser D, Shizuru JA, Sandmaier BM, Molina AJ, Maloney DG, Chauncey TR, Gooley TA, Hegenbart U, Nash RA, Radich J, Wagner JL, Minor S, Appelbaum FR, Bensinger WI, Bryant E, Flowers MED, Georges GE, Grumet FC, Kiem H-P, Torok-Storb B, Yu C, Blume KG, Storb RF. Hematopoietic cell transplantation in older patients with hematologic malignancies: replacing high-dose cytotoxic therapy with graft-versus-tumor effects. Blood 97: 3390-3400, 2001. **Reference ID:** 18428
- 69. Niederwieser D, Maris M, Shizuru JA, Petersdorf E, Hegenbart U, Sandmaier BM, Maloney DG, Storer B, Lange T, Chauncey T, Deininger M, Pönisch W, Anasetti C, Woolfrey A, Little M-T, Blume KG, McSweeney PA, Storb RF. Low-dose total body irradiation (TBI) and fludarabine followed by hematopoietic cell transplantation (HCT) from HLA-matched or mismatched unrelated donors and postgrafting immunosuppression with cyclosporine and mycophenolate mofetil (MMF) can induce durable complete chimerism and sustained remissions in patients with hematological diseases. Blood 101: 1620-1629, 2003.

  Reference ID: 21841
- 70. Maris MB, Niederwieser D, Sandmaier BM, Storer B, Stuart M, Maloney D, Petersdorf E, McSweeney P, Pulsipher M, Woolfrey A, Chauncey T, Agura E, Heimfeld S, Slattery J, Hegenbart U, Anasetti C, Blume K, Storb R. HLA-matched unrelated donor hematopoietic cell transplantation after nonmyeloablative conditioning for patients with hematologic malignancies. Blood 102: 2021-2030, 2003. **Reference ID:** 23067
- 71. Plosker GL, Figgitt DP. Rituximab: a review of its use in non-Hodgkin's lymphoma and chronic lymphocytic leukaemia (Review). Drugs 63: 803-843, 2003. **Reference ID:** 35693
- 72. Hainsworth JD, Litchy S, Barton JH, Houston GA, Hermann RC, Bradof JE, Greco FA. Single-agent rituximab as first-line and maintenance treatment for patients with chronic lymphocytic leukemia or small lymphocytic lymphoma: a phase II trial of

the Minnie Pearl Cancer Research Network. J Clin Oncol 21: 1746-1751, 2003. **Reference ID:** 35692

73. Tam CS, Wolf M, Prince HM, Januszewicz EH, Westerman D, Lin KI, Carney D, Seymour JF. Fludarabine, cyclophosphamide, and rituximab for the treatment of patients with chronic lymphocytic leukemia or indolent non-Hodgkin lymphoma. Cancer 106: 2412-2420, 2006.

**Reference ID:** 35688

74. Vega MI, Huerta-Yepez S, Jazirehi AR, Garban H, Bonavida B. Rituximab (chimeric anti-CD20) sensitizes B-NHL cell lines to Fas-induced apoptosis. Oncogene 24: 8114-8127, 2005.

Reference ID: 35689

75. Zhang N, Khawli LA, Hu P, Epstein AL. Generation of rituximab polymer may cause hyper-cross-linking-induced apoptosis in non-Hodgkin's lymphomas. Clin Cancer Res 11: 5971-5980, 2005.

Reference ID: 35690

- 76. Skvortsova I, Popper BA, Skvortsov S, Saurer M, Auer T, Moser R, Kamleitner H, Zwierzina H, Lukas P. Pretreatment with rituximab enhances radiosensitivity of non-Hodgkin's lymphoma cells. Journal of Radiation Research 46: 241-248, 2005. **Reference ID:** 35691
- 77. Hsu FJ, Komarovskaya M. CTLA4 blockade maximizes antitumor T-cell activation by dendritic cells presenting idiotype protein or opsonized anti-CD20 antibody-coated lymphoma cells. J Immunotherapy 25: 455-468, 2002.

  Reference ID: 24719
- 78. Selenko N, Maidic O, Draxier S, Berer A, Jager U, Knapp W, Stockl J. CD20 antibody (C2B8)-induced apoptosis of lymphoma cells promotes phagocytosis by dendritic cells and cross-priming of CD8<sup>+</sup> cytotoxic T cells. Leukemia 15: 1619-1626, 2001. **Reference ID:** 24054
- 79. Selenko N, Majdic O, Jager U, Sillaber C, Stockl J, Knapp W. Cross-priming of cytotoxic T cells promoted by apoptosis-inducing tumor cell reactive antibodies? (Review). J Clin Immunol 22: 124-130, 2002.

Reference ID: 24093

80. Wierda W, O'Brien S, Wen S, Faderl S, Garcia-Manero G, Thomas D, Do KA, Cortes J, Koller C, Beran M, Ferrajoli A, Giles F, Lerner S, Albitar M, Kantarjian H, Keating M. Chemoimmunotherapy with fludarabine, cyclophosphamide, and rituximab for relapsed and refractory chronic lymphocytic leukemia. J Clin Oncol 23: 4070-4078, 2005.

81. Keating MJ, O'Brien S, Albitar M, Lerner S, Plunkett W, Giles F, Andreeff M, Cortes J, Faderl S, Thomas D, Koller C, Wierda W, Detry MA, Lynn A, Kantarjian H. Early results of a chemoimmunotherapy regimen of fludarabine, cyclophosphamide, and rituximab as initial therapy for chronic lymphocytic leukemia. J Clin Oncol 23: 4079-4088, 2005.

Reference ID: 35694

82. Byrd JC, Peterson BL, Morrison VA, Park K, Jacobson R, Hoke E, Vardiman JW, Rai K, Schiffer CA, Larson RA. Randomized phase 2 study of fludarabine with concurrent versus sequential treatment with rituximab in symptomatic, untreated patients with B-cell chronic lymphocytic leukemia: results from Cancer and Leukemia Group B 9712 (CALGB 9712). Blood 101: 6-14, 2003.

- 83. Berinstein NL, Grillo-López AJ, White CA, Bence-Bruckler I, Maloney D, Czuczman M, Green D, Rosenberg J, McLaughlin P, Shen D. Association of serum Rituximab (IDEC-C2B8) concentration and anti-tumor response in the treatment of recurrent low-grade or follicular non-Hodgkin's lymphoma. Ann Oncol 9: 995-1001, 1998. **Reference ID:** 17126
- 84. McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol 16: 2825-2833, 1998.

  Reference ID: 33375
- 85. Cartron G, Dacheux L, Salles G, Solal-Celigny P, Bardos P, Colombat P, Watier H. Therapeutic activity of humanized anti-CD20 monoclonal antibody and polymorphism in IgG Fc receptor FcgammaRIIIa gene. Blood 99: 754-758, 2002. **Reference ID:** 33371
- 86. Farag SS, Flinn IW, Modali R, Lehman TA, Young D, Byrd JC. Fc gamma RIIIa and Fc gamma RIIa polymorphisms do not predict response to rituximab in B-cell chronic lymphocytic leukemia. Blood 103: 1472-1474, 2004.

  Reference ID: 35695
- 87. Weng WK, Levy R. Two immunoglobulin G fragment C receptor polymorphisms independently predict response to rituximab in patients with follicular lymphoma. J Clin Oncol 21: 3940-3947, 2003.

  Reference ID: 35696
- 88. Carella AM, Biasco S, Nati S, Congiu A, Lerma E. Rituximab is effective for extensive steroid-refractory chronic graft-vs.-host-disease. Leuk Lymphoma 48: 623-624,

2007.

Reference ID: 33483

89. Cutler C, Miklos D, Kim HT, Treister N, Woo SB, Bienfang D, Klickstein LB, Levin J, Miller K, Reynolds C, Macdonell R, Pasek M, Lee SJ, Ho V, Soiffer R, Antin JH, Ritz J, Alyea E. Rituximab for steroid-refractory chronic graft-versus-host disease. Blood 108: 756-762, 2006.

Reference ID: 30214

- 90. Zaja F, Bacigalupo A, Patriarca F, Stanzani M, van Lint MT, Fili C, Scime R, Milone G, Falda M, Vener C, Laszlo D, Alessandrino PE, Narni F, Sica S, Olivieri A, Sperotto A, Bosi A, Bonifazi F, Fanin R. Treatment of refractory chronic GVHD with rituximab: a GITMO study. Bone Marrow Transplant 40: 273-277, 2007. **Reference ID:** 33392
- 91. Ratanatharathorn V, Horowitz MM, Logan B, Arora M, Wang D, Uberti JP, Gale RP, Antin JH, Bornhaeuser M, Hale GA, Ringden O, Cairo MS, Gupta V, Cutler C, Anasetti C, Pavletic SZ. Prior therapy with rituximab correlates with less acute graft-versus-host disease and better survival in B-cell lymphoma patients who received allogeneic peripheral blood stem cell transplantation (PBSCT). Blood 110 (Part 1): 322a, #1063, 2007.(Abstract)

Reference ID: 34194

- 92. Ratanatharathorn V, Ayash L, Reynolds C, Silver S, Reddy P, Becker M, Ferrara JL, Uberti JP. Treatment of chronic graft-versus-host disease with anti-CD20 chimeric monoclonal antibody. Biol Blood Marrow Transplant 9: 505-511, 2003.

  Reference ID: 28825
- 93. Mohty M, Marchetti N, El-Cheikh J, Faucher C, Furst S, Blaise D. Rituximab (RTX) as salvage therapy for refractory chronic graft-versus-host disease (cGVHD). Blood 110 (Part 1): 873A, #2972, 2007.(Abstract)

  Reference ID: 34198
- 94. Miklos DB, Kim HT, Miller KH, Guo L, Zorn E, Lee SJ, Hochberg EP, Wu CJ, Alyea EP, Cutler C, Ho V, Soiffer RJ, Antin JH, Ritz J. Antibody responses to H-Y minor histocompatibility antigens correlate with chronic graft-versus-host disease and disease remission. Blood 105: 2973-2978, 2005.

Reference ID: 30959

95. Stasi R, Del Poeta G, Stipa E, Evangelista ML, Trawinska MM, Cooper N, Amadori S. Response to B-cell depleting therapy with rituximab reverts the abnormalities of T-cell subsets in patients with idiopathic thrombocytopenic purpura. Blood 110: 2924-2930, 2007.

96. Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis 40: 373-383, 1987.

Reference ID: 22434

- 97. Sorror ML, Maris MB, Storer B, Sandmaier BM, Diaconescu R, Flowers C, Maloney DG, Storb R. Comparing morbidity and mortality of HLA-matched unrelated donor hematopoietic cell transplantation after nonmyeloablative and myeloablative conditioning: influence of pretransplant comorbidities. Blood 104: 961-968, 2004. **Reference ID:** 24482
- 98. Diaconescu R, Flowers CR, Storer B, Sorror ML, Maris MB, Maloney DG, Sandmaier BM, Storb R. Morbidity and mortality with nonmyeloablative compared to myeloablative conditioning before hematopoietic cell transplantation from HLA matched related donors. Blood 104: 1550-1558, 2004.

  Reference ID: 24498
- 99. Sorror ML, Maris MB, Storb R, Baron F, Sandmaier BM, Maloney DG, Storer B. Hematopoietic cell transplantation (HCT)-specific comorbidity index: a new tool for risk assessment before allogeneic HCT. Blood 106: 2912-2919, 2005.

  Reference ID: 28079
- 100. Sorror ML, Storer BE, Maloney DG, Sandmaier BM, Martin PJ, Storb R. Outcomes after allogeneic hematopoietic cell transplantation with nonmyeloablative or myeloablative regimens for treatment of lymphoma and chronic lymphocytic leukemia. Blood 111: 446-452, 2008.
  Reference ID: 33209
- 101. Ferrebee JW, Thomas ED. Infusions of marrow in the treatment of radiation casualty. Cincinnati J Med 41: 515-524, 1960.

  Reference ID: 40
- 102. Thomas ED, Herman EC, Jr., Greenough WB, III, Hager EB, Cannon JH, Sahler OD, Ferrebee JW. Irradiation and marrow infusion in leukemia. Arch Intern Med 107: 829-845, 1961.

### <u>APPENDICES – TABLE OF CONTENTS</u>

| APPENDIX A | ELIGIBILITY GUIDELINES FOR DONOR PBSC APHERESIS FOR TRANSFUSION |
|---|---|
| APPENDIX B | THE KARNOFSKY PERFORMANCE STATUS SCALE |
| APPENDIX C | ABO INCOMPATIBILITY |
| APPENDIX D | INFECTIOUS DISEASE GUIDELINES |
| APPENDIX E | GRAFT-VERSUS-HOST DISEASE DATA COLLECTION FORM |
| APPENDIX F | ACUTE GRAFT-VERSUS-HOST DISEASE GRADING |
| APPENDIX G | CHRONIC GRAFT-VERSUS-HOST DISEASE GRADING |
| APPENDIX H | EVALUATION OF DISEASE RESPONSE FOR CLL |
| APPENDIX I | STUDY COORDINATOR'S MANUAL INCLUDING PROCEDURE FOR REPORTING ADVERSE EVENTS |
| APPENDIX J | ADVERSE EVENT REPORT |
| APPENDIX K | NOTICE OF DEATH FORM |
| APPENDIX L | PATIENT DEMOGRAPHICS AND REGISTRATION FORM |
| APPENDIX M | CORE CASE REPORT FORM |
| APPENDIX N | INTRATHECAL THERAPY ADMINISTRATION |
| APPENDIX O | HLA MATCHING REQUIREMENTS FOR UNRELATED DONORS AT THE SCCA/FRED HUTCHINSON ALLIED SYSTEM |
| APPENDIX P | ADAPTED COMMON TOXICITY CRITERIA |
| APPENDIX Q | HCT COMORBIDITY INDEX |
| APPENDIX R | STAGING OF CLL |
| APPENDIX S | WEIGHT/ ADJUSTED BODY WEIGHT FOR DRUG DOSING |
| ADDENDIV T | COODDINATING CENTED FUNCTIONS |

#### **APPENDIX A**

## ELIGIBILITY GUIDELINES FOR DONOR PBSC APHERESIS FOR TRANSFUSION

IMMUNIZATION DONOR ELIGIBILITY

Cholera No wait

Diphtheria No wait

Flu 24 hour wait

Gamma globulin No wait unless for hepatitis

(Immune serum globulin)

Hepatitis B vaccine No wait unless given for hepatitis exposure

Measles (Rubella) 1 month wait

Mumps 2 week wait

Polio - Sabin (inj) No wait

Plague No wait

Rabies 1 year wait if given as treatment for bite. 2

week wait if given as prophylaxis (DMV's or

zoo workers)

Smallpox 2 week wait

Tetanus toxoid No wait

Typhoid No wait

Typhus No wait

Yellow Fever 2 week wait

### APPENDIX B

### THE KARNOFSKY PERFORMANCE STATUS SCALE

| General | Index | Specific criteria |
|---|---|---|
| Able to carry on normal activity; no special care needed. | 100 | Normal, no complaints, no evidence of disease. |
| | 90 | Able to carry on normal activity, minor signs or symptoms of disease. |
| | 80 | Normal activity with effort, some signs or symptoms of disease. |
| Unable to work, able to live at home and care for most personal needs, varying amount of | 70 | Care for self, unable to carry on normal activity or to do work. |
| assistance needed. | 60 | Requires occasional assistance from others but able to care for most needs. |
| | 50 | Requires considerable assistance from others and frequent medical care. |
| Unable to care for self, requires institutional or hospital care or equivalent, disease may be | 40 | Disabled, requires special care and assistance. |
| rapidly progressing. | 30 | Severely disabled, hospitalization indicated, death not imminent. |
| | 20 | Very sick, hospitalization necessary, active supportive treatment necessary. |
| | 10 | Moribund |
| | 0 | Dead |

# APPENDIX C ABO INCOMPATIBILITY

#### **Red Blood Cell - Incompatibility (Major):**

Occasional patients may have antibodies directed against red blood cell antigens found on the donor's cells. These are generally ABO or Rh antigens, although incompatibility with other red cell antigens identified by donor-recipient crossmatch may occur. Although the volume of red blood cells (RBC) in most PBMC products will only be 2-5% of the product volume before infusion, the small quantity may cause a hemolytic transfusion reaction. According to the FHCRC policy it is generally acceptable to infuse a volume of about 10ml RBCs per product. If the recipient shows an anti-donor titer of  $\geq 1:32$  or the RBC volume is greater than 10ml (or > 20ml in two products combined) the PBMC components should be RBC depleted by Starch Sedimentation (flowsheet below). Refer to the Clinical Coordinator's Patient Information Sheet for instructions regarding management of a specific patient.

Post transplant blood component support will be according to Standard Practice Guidelines.

**Timing:** Every attempt should be made to infuse red cell depleted PBMC products within 2 hours of depletion.

**Expected Results:** Red blood cell depleted PBMC products will contain < 10ml of red blood cells and  $\ge 90\%$  nucleated cell recovery.

#### **Red Blood Cell - Incompatibility (Minor):**

Occasional donors may have antibodies directed against red blood cell antigens (ABO, Rh, or other antigen system) found on the recipient's cells. The risk of hemolysis of recipient red cells immediately after transplant is not of very much clinical import. Due to the high number of lymphocytes in the PBMC inoculum, recipients may be at much greater risk for a delayed type of hemolysis that can be severe. PBMC products contain < 200ml of plasma according to FHCRC policy and no deleterious effects have been observed so far. However, if donors show an antirecipient titer  $\ge 1:256$ , the PBMC component should be plasma depleted (see flowsheet below). Refer to the Clinical Coordinator's Patient Information Sheet for instructions regarding management of a specific patient.

Post transplant blood component support will be according to Standard Practice Guidelines.

**Timing:** Every attempt should be made to infuse plasma-depleted PBMC within 2 hours of depletion.

**Expected Results:** The plasma depletion should not affect the nucleated cell recovery.

#### **Red Blood Cell – Bidirectional Incompatibility:**

Patients undergoing transplants for bidirectional RBC incompatibility should be managed according to both algorithms shown below. Most red cell depletion techniques also deplete plasma from the PBMC component with no additional cell loss. *Refer to the Clinical Coordinator's Patient Information Sheet for instructions regarding management of a specific patient.* 

Post transplant blood component support will be according to Standard Practice Guidelines.

## **Appendix C (continued)**

| MAJOR ABO INCOMPATIBLE | | | | |
|---|---|---|---|---|
| | ≥ 1:32 | <20ml RBC total | | Infuse without modification |
| Recipient anti-<br>Donor titer | ≥ 1.32 | >20ml RBC total | $\Rightarrow$ | RBC depletion of component |
| | ≤ 1:16 | $\Rightarrow$ | | Infuse without modification |
| MINOR ABO | MINOR ABO INCOMPATIBLE | | | |
| Donor anti- | ≥ 1:256 | Plasma depletion of component | | |
| Recipient titer | ≤ 1:128 | Infuse without modification | | |

## APPENDIX D INFECTIOUS DISEASE GUIDELINES

Please note that the content of these PDFs is from the Fred Hutchinson Clinical Research Division Standard Practice Manual and does not contain research related procedures.

Herpes Simplex and Varicella Zoster Virus Prevention and Treatment



**CMV Prevention: Surveillance and Preemptive Therapy** 



**CMV Disease: Diagnosis and Treatment** 



**Antifungal Therapy Guidelines** 



Pneumonia / Pneumocystis Jiroveci Prophylaxis



pneumocystisjiroveci

Antibiotic Prophylaxis for Encapsulated Bacteria in Allogeneic Patients with Chronic GvHD Requiring Immunosuppressive Therapy



Vaccinations



**Foscarnet** 



FHCRC Current Version 1/13/2016
## **APPENDIX E**

## GRAFT-VERSUS-HOST DISEASE DATA COLLECTION FORM

## **GVHD TREATMENT:**

| Check each agent used to treat GVHD: | Date Treatment Started None |
|---|---|
| Cyclosporine Systemic Corticosteroids Topical Corticosteroids Beclomethasone Rapamycin MMF ATG In Vivo anti-T lymphocyte McAb Blinded Randomized Trial Specify Other, specify | |
| Date of Death:/ | _/ |
| Was an autopsy done? | s 🗌 No |
| Was GVHD found at autopsy? ☐ Ye | s No N/A |
| If yes:<br>☐ Skin<br>☐ Liver<br>☐ Gut | |
| | HD SUMMARY |
| Date of onset:// | Day |
| Overall Grade | |
| Skin Liver | Gut |
| Comments | |

| | BIOPSIES |
|---|---|
| Was skin biopsy done? Date of skin biopsy: Results: Negative Positive GVHD Positive Other | ☐ Yes ☐ No<br>// |
| Was liver biopsy done? Date of liver biopsy: Results: Negative Positive GVHD Positive Other Did patient have any GI Biopsy? Date of biopsy: Results: Negative Positive GVHD Positive Other | ☐ Yes No // |
| | <u>CLINICAL SKIN</u> |
| Did patient ever have rash after trar | nsplant? |
| Was rash thought to be due to GVH | ID? |
| Date of onset of rash: | |
| Extent of rash on date of first treatment of maximum severity of rash: 0 – No rash 1 – Maculopapular rash 2 – Maculopapular rash 3 – Generalized erythrod 4 – Generalized erythrod | <25% BSA<br>25-50% BSA |
| Date of maximum rash seve | rity:/ |
| | CLINICAL LIVER |
| Bilirubin level on date of first treatme | ent for GVHD: |
| Maximum Bilirubin Date | |
| <ul> <li>□ 0 – Bilirubin &lt; 2.0 mg/dl</li> <li>□ 1 – Bilirubin 2.0 – 3.0 mg/dl</li> <li>□ 2 – Bilirubin 3.1 – 6.0 mg/dl</li> </ul> | |

FHCRC Current Version 1/13/2016

| ☐ 3 – Bilirubin 6.1 – 15.0 mg/dl<br>☐ 4 – Bilirubin >15.0 mg/dl |
|---|
| Did patient have other liver process? VOD Cyclosporine Toxicity Sepsis Other liver complication |
| CLINICAL GUT |
| GI consult? |
| Stool volume on date of first treatment for GVHD: |
| Maximum Daily Stool Output after day 21 |
| <ul> <li>□ 0 - 0 - ≤200 ml</li> <li>□ 1 - &gt;200 but ≤1000 ml</li> <li>□ 2 - &gt;1000 but ≤1500 ml</li> <li>□ 3 - &gt;1500 ml</li> <li>□ 4 - Severe abdominal pain with or without ileus</li> </ul> Date of maximum stool output:// |
| Was stool mixed with urine on day of Maximum Stool Output? Yes No If stool volume not measurable, what was maximum number of stools/day? Date of maximum number of stools/day:// Did patient have the following process? Frank blood in stool attributed to GVHD CMV infection of GI tract at time of maximum stool volume Narcotic withdrawal at time of maximum stool volume C. difficile infection at time of maximum stool volume Other GI process Specify |
| Date Completed/ Completed by: |

## APPENDIX F ACUTE GRAFT-VERSUS-HOST DISEASE GRADING<sup>a</sup>

#### Severity of Individual Organ Involvement

| Skin | <ul> <li>a maculopapular eruption involving less than 25% of the body surface</li> <li>a maculopapular eruption involving 25-50% of the body surface</li> <li>generalized erythroderma</li> <li>generalized erythroderma with bullous formation and often with desquamation</li> </ul> |
|---|---|
| <u>Liver</u> | +1 bilirubin (2.0-3.0 mg/100 ml)<br>+2 bilirubin (3-5.9 mg/100 ml)<br>+3 bilirubin (6-14.9 mg/100 ml)<br>+4 bilirubin > 15 mg/100 ml |
| <u>Gut</u> | rrhea is graded +1 to +4 in severity. Nausea and vomiting and/or anorexia sed by GVHD is assigned as +1 in severity severity of gut involvement is assigned to the most severe involvement noted. ents with visible bloody diarrhea are at least stage +2 gut and grade +3 overall |
| <u>Diarrhea</u> | +1 $\leq 1000 \text{ ml of liquid stool/day}^* (\leq 15\text{ml of stool/kg/day})^{\dagger}$<br>+2 $\geq 1,000 \text{ ml of stool/day}^* (\geq 15\text{ml of stool/kg/day})^{\dagger}$ |

<sup>\*</sup>In the absence of infectious/medical cause

+2 +3

+4

#### Severity of GVHD

>1,500 ml of stool/day\* (> 20ml of stool/kg/day)<sup>†</sup> 2,000 ml of stool/day\* (> 25ml of stool/kg/day)<sup>†</sup>

Grade I +1 to +2 skin rash

No gut or liver involvement

Grade II +1 to +3 skin rash

+1 gastrointestinal involvement and/or +1 liver involvement

Grade III +2 to +4 gastrointestinal involvement and/or

+2 to +4 liver involvement with or without a rash

<u>Grade IV</u> Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms

or death

<sup>&</sup>lt;sup>†</sup>For pediatric patients

a From "Graft-vs-host disease" Sullivan, Keith M. *Hematopoietic Cell Transplantation* Ed: D. Thomas, K. Blume, S. Forman, Blackwell Sciences; 1999, pages 518-519

#### APPENDIX G

#### CHRONIC GRAFT-VERSUS-HOST DISEASE GRADING <sup>a</sup>

In all cases, concomitant processes (i.e. infections or drug reactions) must be ruled out. Karnofsky or Lansky Clinical Performance scores, 60%, > 15% weight loss, and recurrent infections are usually signs of clinical extensive chronic GVHD. Abnormalities that could indicate chronic GVHD are categorized by organ systems as listed below.

Skin Erythema, dryness, pruritus, pigmentary changes (i.e. hyperpigmentation,

vitiligo), mottling, papulosquamous plaques, nodules, exfoliation, macular-papular or urticarial rash, scleroderma, morphea (one or several circumscribed,

indurated and shiny lesions)

Nails Ridging, onychodystrophy, onycholysis

Hair Premature graying, (scalp hair, eyelashes, eyebrows), thinning scalp hair,

alopecia, decreased body hair

Mouth Dryness, burning, gingivitis, mucositis, striae, atrophy, erythema, lichenoid

changes, ulcers, labial atrophy or pigmentary changes, tooth decay, tightness

around the mouth

Eyes Dryness, burning, blurring, gritty eyes, photophobia, pain

Vagina/vulva Dryness, dyspareunia, stricture or stenosis, erythema, atrophy or lichenoid

changes not included

Liver Elevated liver function tests not due to other causes (alkaline phosphatase  $\geq 3x$ 

upper limit of normal, AST or ALT  $\geq$ 4x upper limit of normal or total serum bilirubin  $\geq$  2.5; in the absence of chronic GVHD involving other organs, liver

biopsy is required to confirm diagnosis)

Lung Bronchiolitis obliterans (see diagnostic indicators), cough, wheezing, dyspnea on

exertion, history of recurrent bronchitis or sinusitis

GI Anorexia, nausea, vomiting, weight loss, dysphasia, odynophagia, malabsorption

Fasciitis Stiffness and tightness with restriction of movement, occasionally with swelling

pain, cramping, erythema and induration, most commonly affecting forearms, wrists and hands, ankles, legs, and feet, inability to extend wrists without flexing

the fingers or the elbows, contractures

Serositis Chest pain or cardiopulmonary comprise due to pericarditis or pleuritis

Muscle Proximal muscle weakness, cramping

Skeletal Arthralgia of large proximal girdle joints and sometimes smaller joints

### Laboratory testing sand diagnostic indicators of chronic GVHD<sup>a</sup>

Eye Schirmer's test with a mean value  $\leq 5$ mm at 5 minutes, or symptomatic with

values of 6-10mm or keratitis detected by slit lamp examination

Liver Elevated liver function tests not due to other causes (see definition of clinical

limited and extensive chronic GVHD)

Lung New obstructive lung defect defined as  $FEV_1 \le 80\%$  of predicted with either an

FEF  $_{25-75}$  <65% of predicted or RV >120% of predicted, or a decrease of FEV<sub>1</sub>/FVC by > 12% within a period of less than 1 year. A diagnosis of bronchiolitis obliterans requires negative microbiological tests from

bronchoalveolar lavage and evidence of air trapping by high resolution endexpiratory and end-inspiratory CAT scans o the chest. A thoracoscopic lung biopsy may be necessary in order to confirm the diagnosis of bronchiolitis

obliterans in patients who have obstructive lung disease without air trapping when

chronic GVHD involving other organs is absent

Esophagus Esophageal web formation, stricture or dysmotility demonstrated by barium

swallow, endoscopy or manometry

Muscle Elevated CPK or aldolase, EMG findings consistent with myositis

Blood Thrombocytopenia (usually 20,000-100,000/µl), eosinophilia,

hypogammaglobulinemia, hypergammaglobulinemia, and autoantibodies occur in

some cases

<sup>&</sup>lt;sup>a</sup> From Standard Practice Guidelines for "Chronic Graft-versus-Host Disease Classification at the time of presentation" developed by Long Term Follow-Up at the FHCRC

### GRADING OF CHRONIC GRAFT-VERSUS-HOST DISEASE

#### A Clinical limited chronic GVHD

- 1. Oral abnormalities consistent with chronic GVHD, a positive skin or lip biopsy, and no other manifestations of chronic GVHD
- 2. Mild liver test abnormalities (alkaline phosphatase  $\leq 2x$  upper limit of normal, AST or ALT  $\leq 3x$  upper limit of normal and total bilirubin  $\leq 1.6$ ) with positive skin or lip biopsy, and no other manifestation of chronic GVHD
- 3. Less than six papulosquamous plaques or limited skin rash or dyspigmentation (< 20% of the body surface), positive skin biopsy, and no other manifestations of chronic GVHD
- 4. Ocular sicca (Schirmer's test ≤ 5mm), positive skin or lip biopsy, and no other manifestations of chronic GVHD
- 5. Vaginal or vulvar abnormalities with positive biopsy, and no other manifestations of chronic GVHD

#### B. Clinical extensive chronic GVHD

- 1. Involvement of two or more organs with symptoms or signs of chronic GVHD, with biopsy documentation of chronic GVHD in any organ
- 2. > 15% base line body weight loss not due to other causes, with biopsy documentation of chronic GVHD in any organ
- 3. Skin involvement more extensive than defined for limited chronic GVHD, confirmed by biopsy
- 4. Scleroderma or morphea
- 5. Onycholysis or onychodystrophy thought to represent chronic GVHD, with documentation of chronic GVHD in any organ
- 6. Decreased range of motion in wrist of ankle extension due to fasciitis caused by chronic GVHD
- 7. Contractures thought to represent chronic GVHD
- 8. Bronchiolitis obliterans
- 9. Positive liver biopsy; abnormal liver function tests not due to other causes with alkaline phosphatase > 2x upper limit of normal, AST or ALT > 3x upper limit of normal, or total bilirubin > 1.6, and documentation of chronic GVHD in any organ
- 10. Pericarditis or pleuritis not due to other causes
- 11. Positive upper or lower GI biopsy

<sup>&</sup>lt;sup>a</sup> From Standard Practice Guidelines for "Chronic Graft-versus-Host Disease Classification at the time of presentation" developed by Long Term Follow-Up at the FHCRC

#### APPENDIX H

#### EVALUATION OF DISEASE RESPONSE FOR CLL

CLL: Modified response criteria based on the NCI-Working Group and the International Workshop Group Joint Formal Criteria for evaluating disease response for CLL. [1-3]

| Complete Remission (CR) | |
|---|---|
| Imaging studies (Xray, CT, MRI) (nodes, liver, and spleen) | Normal |
| Peripheral blood by flow cytometry | No clonal lymphocytes |
| Bone marrow by morphology | No nodules; or if present, nodules are free |
| | from CLL cells by immunohistochemistry |
| Duration | ≥2 months |
| CR with minimal residual disease | |
| Peripheral blood or bone marrow by flow cytometry | >0 - <1 CLL cells/1000 leukocytes (0.1%) |
| Partial Remission (PR): | |
| Both criteria: | |
| Absolute lymphocyte count in peripheral blood | ≥50% decrease³ |
| Physical exam/Imaging studies (nodes, liver, and/or spleen) | ≥50% decrease <sup>3,4</sup> |
| Duration | ≥2 months |
| Progressive disease: ≥1 of | |
| Physical exam/Imaging studies (nodes, liver, and/or spleen) | ≥50% increase or new |
| Circulating lymphocytes by morphology and/or flow cytometry | ≥50% increase |
| Lymph node Biopsy | Richter's transformation |
| Stable disease | |
| Did not meet any of the above criteria for complete or partial remissi | on or progression. |
| Relapsed disease | |

Criteria of progression occurring 6 months after achievement of complete or partial remission.

- 1. Cheson BD, Bennett JM, Grever M, Kay N, Keating MJ, O'Brien S, Rai KR. National Cancer Institute-sponsored Working Group guidelines for chronic lymphocytic leukemia: revised guidelines for diagnosis and treatment. Blood 87: 4990-4997, 1996.
- 2. Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ, International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the

Without granulocyte colony stimulating factor support.

<sup>&</sup>lt;sup>2</sup> Without red blood cell transfusions or erythropoietin support.

<sup>&</sup>lt;sup>3</sup> Compared to before starting therapy.

<sup>&</sup>lt;sup>4</sup> Defined by the sum of the products of up to 6 lymph nodes with no increase in the size of any single lymph node (ie, an increase of <25 percent in a lymph node <2cm is not considered significant) and no new enlarged lymph nodes.

International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines [Erratum appears in Blood. 2008 Dec 15;112(13):5259]. Blood 111: 5446-5456, 2008.

3. Chronic lymphocytic leukemia: recommendations for diagnosis, staging, and response criteria. International Workshop on Chronic Lymphocytic Leukemia. Ann Intern Med 110: 236-238, 1989.

#### **APPENDIX I**

## STUDY COORDINATOR'S MANUAL INCLUDING PROCEDURE FOR REPORTING ADVERSE EVENTS

#### I. Introduction

The mixed chimerism protocols have been opened to multiple sites to increase the referral base and accrual. Because of this expansion of collaborators, the data collection procedures are being revised. The procedure manual was created to assure consistency of data reporting across the centers and to assure compliance with regulations. General expectations of collaborators are that they will comply with appropriate regulatory requirements, specified protocol requirements, and provide outcome data.

The manual translates working procedures for study coordination. Its goal is to describe the procedures with sufficient clarity to ensure that all study centers will use the same procedures and follow-up schedules for participant data management and reporting. Changes to the manual and relevant forms will be made as soon as practical and will become effective on receipt of the revised procedures at the study centers, unless otherwise noticed.

#### II. Institutional Review Board Review of Protocols and Modifications

All research protocols proposed for use that involves human subjects must be reviewed and approved by the Institutional Review Board (IRB) prior to implementation. New protocols will undergo review at the FHCRC IRB and then will be distributed to sites that wish to participate for their IRB's review. For Centers that have a Federal Wide Assurance (FWA), formal collaboration includes submission of a form 310 and a copy of the IRB approved protocol and consent forms to the FHCRC. For sites without a FWA, an FWA form needs to be filed. Once the paperwork is submitted to the Office for Human Research Protection, the approval process can take up to a couple of months, and must be <u>completed</u> before collaboration on a protocol can begin.

In addition, all amendments and/or revisions to on-going, approved activities must be submitted for review and approved prior to implementation at an institution. No revisions may be implemented at outside institutions without the prior approval of the FHCRC Principal Investigator. The FHCRC and the local site's IRB must review all protocol activities at least once annually. This must be done within 365 days of the last review regardless of the policies of the institution. A copy of annual renewal approvals must be received for collaboration to continue for the next year.

## III. Registrations

<u>Collaborating Institutions</u>: The principal investigator of the collaborating institution who will register the patient with the FHCRC will identify eligible patients. Registration will include completion of the eligibility checklist/demographic form. This form and a copy of the signed informed consent will be faxed (206-667-5378) prior to treatment initiation. Patients must be registered prior to treatment initiation for valid registration

## **Appendix I (continued)**

## IV. Reporting Adverse Events

The following guidelines are the minimum serious adverse event (SAE) reporting guidelines for Category 1 and 2 studies conducted at the Fred Hutchinson Cancer Research Center.

Expedited Reporting Requirements

All unexpected and serious adverse events which may be due to study treatment or intervention must be reported to the FHCRC Institutional Review Office as soon as possible but within at least 10 calendar days of the investigator learning of the event.

**Definitions** 

**Adverse Event** - Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, medical treatment or procedure and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, medical treatment or procedure whether or not considered related to the medicinal product.

**Life-threatening Adverse Event** – Any adverse event that places the patient or subject, in view of the investigator, at immediate risk of death from the reaction. Study toxicities are graded using the NCI Common Toxicity Criteria (where appropriate use the criteria for transplant patients.) All Grade 4 (life-threatening) toxicities occurring between start of conditioning to day 200 that meet expedited reporting requirements must be reported as soon as possible but within at least 10 calendar days of the investigator learning of the event.

**Unexpected Adverse Event** – An adverse event, the nature or severity of which is not consistent with the applicable product information (e.g., Investigator's Brochure for an unapproved investigational product or package insert/summary of product characteristics for an approved product). If applicable product information is not available, such as for studies that do not involve pharmaceutical products or devices, an unexpected adverse event is an adverse event that was not described in the study protocol or informed consent.

**Serious Adverse Event (SAE)** – Any adverse event occurring that results in any of the following outcomes:

- ➤ Death start of conditioning to day 200, regardless of cause,
- ➤ A life-threatening adverse event (see above)
- ➤ A persistent or significant disability/incapacity,
- > A congenital anomaly
- > Requires intervention to prevent permanent impairment or damage.

### **Appendix I (continued)**

Hospitalization, in general, will not be considered a serious adverse event as approximately half of evaluable MRD patients AND the majority of evaluable URD patients receiving nonmyeloablative transplants were hospitalized. Hospitalization will be considered a serious adverse event if it fulfills the criteria for a serious and unexpected adverse event as described above.

To ensure no confusion or misunderstanding exist of the differences between the terms "serious" and "severe," which are not synonymous the following note of clarification is provided:

The term "severe" is often used to describe the intensity (severity) or a specific event (as in mild, moderate or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe headache). This is *not* the same as "serious," which is based on patient/event *outcome or action* criteria usually associated with events that pose a threat to a patient's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory obligations.

**Attribution** - The FHCRC designation for the determination of whether an adverse event is related to a medical product, treatment or procedure will be as follows:

- ➤ Related includes adverse events that are definitely, probably, or possibly related to the medical treatment or procedure.
- ➤ Not Related includes adverse events are doubtfully related or clearly not related to the medical treatment or procedure.

The FHCRC Serious Adverse Event (SAE) Report Form should be completed for all adverse events that meet the expedited reporting requirements. All available information should be submitted but it is acceptable to fax an incomplete report form at the initial report. A completed report should be faxed as soon as possible but must be received within 10 calendar days.

It is the responsibility of the FHCRC Principal Investigator to notify the sponsor, NIH, FDA or other agencies of serious adverse events as required in the protocol.

Serious adverse events that do not meet the requirement for expedited reporting (not related to study treatment or expected) will be reported to the IRB as part of the annual renewal of the protocol.

FHCRC is acting as the Coordinating Center for this multi-institutional study, and it is the responsibility of the FHCRC Principal Investigator (or designee) to complete the FHCRC Serious Adverse Event Report for all serious adverse events that meet the expedited reporting requirements that are received from the participating sites.

### **Appendix I (continued)**

Procedure for Reporting Serious and Unexpected Adverse Events from Participating Sites Regulations defining the responsibilities for reporting serious and unexpected adverse reactions are defined above. Serious and unexpected adverse events must be reported to the FHCRC Investigator within 10 days of learning of the event. This includes patient deaths (serious, unexpected, and related/possibly related), regardless of cause, occurring start of condition to day 200 post-transplant procedure. The immediate telephone report must be followed by faxed comments to the Trial Coordinator at (206) 667-5378. This will be followed by detailed written report (See Appendix J) within 10 working days. The report must include the date and time of onset, severity and duration of the event, the relationship to the study, the treatment given and eventual outcome. Follow-up information to a SAE report must be submitted as soon as the relevant information is available.

#### **Obligation of Investigators**

All grade 3 or 4 adverse events (or highly unusual grade 2 adverse events), which occur between start of conditioning to day 100 during the study will be recorded on the Case Report Form (**Appendix M**). These adverse events which are observed by the Investigator or reported by the patient, whether or not attributed to the study, will be reported on the Case Report Form using the modified (for HSCT) NCI Common Toxicity Criteria (**Appendix P**). Attributes will include a description, date of onset, maximum severity, and assessment of relationship to the study agent or other suspect agent(s).

Adverse events will be graded accordingly: 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening or debilitating, and 5 = fatal. All Grade 4 (life-threatening) or Grade 5 (fatal) events on the NCI scale meet expedited reporting requirements.

Association or relatedness to the study agent will be graded as follows: 1 = unrelated, 2 = unlikely, 3 = possibly, 4 = probably, and 5 = definitely related.

#### V. Case Report Forms

Case report forms must be completed for all patients registered onto the protocol and submitted to the FHCRC data coordinating center. The first case report form (day 28) is due on day 50. For outside centers a Staging Form must accompany the form with the patient staging at registration, day 28, day 56, day 84 and day 100. Staging forms should also be completed with each Follow Up Form completed on day 180, 1 year, 1.5 years, 2 years, 3 years, and yearly thereafter. For Outside Centers, case report forms are expected to be submitted no later than 30 days following the scheduled follow up date.

## VI. Protocol Monitoring

As the coordinating center, FHCRC will monitor accrual at the outside institutions. The guidelines below are intended to guide the reviewers in their assessment of items that significantly alter the clinical effectiveness of the treatment or the evaluation of its toxicity.

### Appendix I (continued)

#### A. Registration/Randomization

- 1. Patient was registered prior to treatment and approval by FHCRC PI occurs prior to randomization.
- 2. Information given at registration represents actual data in medical records (stage, diagnosis, cell type, etc.)

## B. Informed Consent/IRB Approval Dates

- 1. The consent was signed prior to registration
- 2. The consent is in language was approved by the institution's IRB. IRB approval and reapproval are documented including appropriate use of full-board review and proper review of appropriate amendments or revisions
- 3. Consent was dated and has written witness signature. IRB approval was obtained prior to the patient signing the consent form and start of treatment.

## C. Patient Eligibility

- 1. Eligibility criteria and exclusion criteria were met
- 2. Treatment/Intervention Administration
- 3. Doses were modified according to protocol
- 4. Accurate documentation of drug administration

#### D. Study Tests/Evaluation

- 1. Protocol specified laboratory tests or diagnostic studies are available
- 2. Appropriate record of protocol intervention is documented.

#### E. Study Events/Adverse Drug Experience

1. Serious Adverse Evens reported according to protocol specifications

#### F. Follow-Up

- 1. Disease status assessed according to the required protocol guidelines documenting response to treatment.
- 2. Accurate determination of cancer progression

## **APPENDIX J**

## Fred Hutchinson Cancer Research Center SERIOUS ADVERSE EVENT REPORT (SAE) Form IRO-08

| FHCRC IR File Number: | FHCRC Protocol Number: |
|---|---|
| FHCRC Unique Patient # | ☐ FHCRC/SCCA ☐ Other |
| Gender: Male Female | Age: |
| FHCRC Principal Investigator: | |
| Phone Number: | Mailstop: |
| Date study staff became aware of event: | |
| Date of Report: Initial Report Follow-Up | Report # Other |
| Date Serious Adverse Event Started: | |
| Date Ended: Or Ongoing (if | ongoing – must submit follow up report) |
| Adverse Event: | |
| Describe the Serious Adverse Event including a summar (Or attach a MedWatch Form or other SAE reporting for Outcomes Attributed to adverse event: (Check all that a Death / Life-Threatening Hospitalization (initial or prolonged) Specify Agent(s) and/or Procedure(s) involved in this present Pharmaceutical product/medical treatment/procedure Not Related (Unrelated, Unlikely) Related (Possible, Probable, Definite) | pply) Disability Congenital Anomaly Required intervention to prevent permanent impairment/damage |
| ☐ Follow-up Report Required | Final Report (PI must sign final report) |
| Report Completed by: | Date: |
| The PI has determined that the consent form must be rev | rised: Yes No |
| Does this study involve the deliberate transfer of recomb DNA, into human subjects (human gene transfer)? ye outpatient clinic, a copy of this Protocol Modification For approved, will be forwarded to the FHCRC's Institutions (Mailstop: LM-230). | es no If yes and the activity involves the SCCA orm and any supporting documents to be reviewed and |
| Signature of Principal Investigator | Date: |

Page 2

## Fred Hutchinson Cancer Research Center SERIOUS ADVERSE EVENT REPORT (SAE) Form IRO-08

| FHCRC IR File Number: | FHCRC Protocol Number: |
|---|---|
| FHCRC Unique Patient # | Date of Report: |
| Describe the Serious Adverse Event including a summary of all relevant clinical information. | |

## APPENDIX K NOTICE OF DEATH

| Patient ID: | Date of Death: |
|---|---|
| Place of Event: | |
| Apparent cause of death (Please be possible): | specific. Attach hospital summary or death summary when |
| Form completed by: | Date: |

## APPENDIX L

## **Patient Demographics and Eligibility Form**

## 1840

Please Fax this completed form to (206)-667-5378 for patient registration. Questions regarding eligibility should go to Mohamed Sorror, M.D., 206-667-2765.

| UPN# | | |
|---|---|---|
| Patient Name: (Last) | (First) | |
| Date of Birth:// | Gender (choose one): Male Female | Unknown |
| Patient Diagnosis: | Planned Day 0: ${(Mo)} / {(Do)}$ | ay) / (Year) |
| Ethnicity (choose one): Instruct the research subject to select one of the following. Hispanic (A person of Cuban, Mexican, Puerto Rican, South or Central American, or other Spanish culture or origin, regardless of race. Term "Spanish Origin" can also be used in addition to "Hispanic" or "Latino". Not Hispanic or Latino Declined to report | | |
| Race (check all that apply): Instruct the research subject to select one or more of the following. American Indian/Alaska Native (A person having origins in any of the original peoples of North, Central, or South America, and who maintains tribal affiliations or community attachment). Asian (A person having origins in any of the original peoples of the Far East, Southeast, Asia, or the Indian subcontinent including, for example, Cambodia, China, India, Japan, Korea, Malaysia, Pakistan, the Philippine Islands, Thailand and Vietnam). Native Hawaiian/Pacific Islander (A person having origins in any of the original peoples of Hawaii, Guam, Samoa or other Pacific Islands). Black/African American (A person having origins in any of the black racial groups of Africa). White (A person having origins in any of the original peoples of Europe, the Middle East or North Africa). Research subject does not know race Declined to report | | |
| Protocol 1840 Eligibility | | |
| Inclusion Criteria: All of the following questions must be marked "Yes" for t | he patient to enter the stud | dy. |
| 1. Yes No Patient signed IRB approved cons | | |

| 2. | ☐ Yes ☐ No | Patient has a diagnosis of CLL (or small lymphocytic lymphoma) or Diagnosis of CLL that progresses to prolymphocytic leukemia (PLL). | | | | | |
|---|---|---|---|---|---|---|---|
| 3. | ☐ Yes ☐ No | Patient has at le | east one of t | he following: | | | |
| | | a. 🗌 Yes 🗀 | W<br>or<br>re<br>ni<br>di<br>th | Has B-Cell CLL or P<br>Vorking Group criter<br>r partial response after<br>egimen containing fluctures and the<br>ucleoside analog, e.g<br>isease relapse within<br>herapy with a fludara<br>malog) containing reg | ia (Appendix er 2 cycles of udarabine (or g. 2-CDA, pen 12 months af bine (or anoth | H) for complete therapy with a another atostatin) or effect completing | |
| | | b. Yes | _ | as B-Cell CLL or PI<br>ombination chemother | | | |
| | | c. Yes | ao<br>P | las B-Cell CLL or PI<br>cquired "17p deletion<br>atients should have r<br>ut could be transplan | n" cytogenetic<br>received induc | e abnormality. | |
| 4. | ☐ Yes ☐ No | Related don | or who is g | enetically phenotypi | cally HLA-id | entical | |
| | | OR | | | | | |
| | | i) Matc<br>resolu<br>ii) Only | hed for HLaution typing<br>a single all<br>d by high re | are prospectively: A-A,B,C, DRB1 and g <u>AND</u> ele disparity will be esolution typing (See | allowed for H | ILA-A, B, or C | |
| | Patient | | | | | | |
| | | | | C: | | B: | |
| | DRB1: | DRB1: | DQB1: | DQB1: | _ | | _ |
| | Donor | Δ. | C. | C. | D. | D. | |
| | | | | C: | | D | |
| | DRB1: | DKRI: | ndri: | DQB1: | _ | | |

| iii) | Have a negative anti-donor cytotoxic crossmatch. Cytotoxic crossmatch <b>not done as patient and donor are phenotypically identical by molecular methods.</b> |
|---|---|
| iv) 🗌 Yes 🗌 No | Patient and donor pairs must not be homozygous at a mismatched allele. |
| 5. Yes No F | Patient is 18 years of age or older. |
| Exclusion criteria: Each of the following quest | tions must be marked "No" Or "NA" for the patient to enroll in the study. |
| 6. Yes No | Has active CNS involvement with CLL. For LP requirement, see Appendix N. |
| | Patients with active non-hematologic malignancies (except non-melanoma skin cancers). This exclusion does not apply to patients with non-hematologic malignancies that do not require therapy |
| 8. Yes No | Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a >20% risk of disease recurrence. This exclusion does not apply to patients with non-hematologic malignancies that do not require therapy |
| 9. Yes No NA | Fertile man or woman unwilling to use contraceptive techniques during and for 12 months following treatment. |
| 10. | Female who is pregnant or breastfeeding. |
| 11. Yes No | The addition of cytotoxic agents for "cytoreduction" with the exception of tyrosine kinase inhibitors (such as imatinib mesylate), cytokine therapy, hydroxyurea, low dose cytarabine, chlorambucil, or rituxan within three weeks of the initiation of conditioning. |
| | function as described below. Please check <b>YES</b> if patient has any of following. |
| a. Cardiovascula | <u>nr:</u> |
| Y | es No Cardiac Ejection Fraction <40%. Ejection fraction is required if age >50 years or there is a history of prior transplant, anthracycline exposure or history of cardiac disease. |

FHCRC Current Version 1/13/2016

| | ∐ Yes ∐ No | multiple antihypertensives. |
|---|---|---|
| b. <u><b>Pulmo</b></u> | onary:<br>☐ Yes ☐ No | DLCO < 40%, TLC <40%, FEV1 <40% and/or is requiring supplementary continuous oxygen, or severe deficits in pulmonary function testing as defined by pulmonary consultant service. The FHCRC PI of the study must approve of enrollment of all patients with pulmonary nodules. |
| c. <u>Hepat</u> | PI Signature: | Date: |
| с. перас | Yes No | Patients with clinical or laboratory evidence of liver diseas would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension. Patients will be excluded if they ar found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, hepatic damage with bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombir time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin >3 mg/dl, or symptomatic biliary disease. |
| 13. | Performance stat<br>a. Karnofsk | tus: ty score < 60 (see <b>Appendix B</b> ) for adult patients |
| 14. Yes No | Infection with | h HIV |
| 15. | Active bacterial therapy. | or fungal infections unresponsive to medical |
| Note: The HCT-C (fax HCT-CI wor | CI score is:_<br>ksheet with regis | tration—see Appendix Q) |
| Signature of person | completing form: | Date: |
| Signature of Princip | al Investigator: | Date: |

## APPENDIX M CORE CASE REPORT FORMS



## APPENDIX N

## INTRATHECAL THERAPY ADMINISTRATION



## **Appendix O**

## **HLA Matching Requirements For Unrelated Donors At The SCCA/Fred Hutchinson Allied System**

Human Leukocyte Antigen (HLA) Terminology. The HLA region consists of genes that encode two classes of HLA molecules. HLA class I molecules, HLA-A, -B, and -C, are composed of a single glycoprotein chain that is expressed in association with ®2-microglobulin on most tissue cells. HLA class II molecules, HLA-DR, -DQ, and -DP, are heterodimers consisting of  $\langle$  and  $\otimes$  glycoprotein chains. HLA class I and HLA class II molecules are highly polymorphic.

HLA Typing Methods. At the Seattle Cancer Care Alliance Clinical Immunogenetics Laboratory (CIL) DNA-based methods of HLA-A, B, C, DRB1, DQB1 typing are now performed routinely. High resolution typing is required to define individual alleles and the level of mismatching between donor and recipient. High resolution data are reported with four or more digits (e.g., A\*0201, A\*0205, B\*1504, or DRB1\*0401). A current listing of recognized HLA alleles and their sequences can be found at the Immunogenetics/HLA sequence database website at www.anthonynolan.org.uk/HIG/data.html.

Initial typing reports obtained through the international marrow donor registries may consist of **intermediate resolution** typing. **Intermediate resolution** defines alleles in groups of related families historically defined as *antigens* by alloantisera. **Intermediate resolution** typing results are reported as two digits (e.g., A\*02, B\*15, or DRB1\*04). In cases where the HLA-A, B and C loci are typed at intermediate resolution and high resolution data are not available, it should be understood that unidentified allele disparity might be present.

**Donor Selection.** Final selection of an unrelated donor should be based upon results of **high resolution** typing of HLA-A, B, C, DRB1, DQB1 alleles. Cross match assay is not required when high resolution typing indicates matching for HLA-A, B, C, DRB1 and DQB1 AND the platelet reactive antibody (PRA) screen is not elevated (defined as  $\leq$ 10%). A negative cross match test result is required for final donor selection in the following situations: 1) PRA screen is positive (>10%), or 2) high resolution typing indicates mismatching for one or more HLA-A, B, C, DRB1 and DQB1 alleles. A positive anti-donor cytotoxic crossmatch absolutely excludes the donor.

**Donor Selection Criteria.** Protocols and treatment plans must specify donor inclusion and exclusion criteria, using terminology indicated below.

Donor inclusion criteria **must specify** 1) the allowable genetic relationship between the patient and donor (related and/or unrelated), 2) the allowable limits of mismatch, and if applicable 3) any modification of mismatch criteria according to type of disease or patient characteristics.

## **HLA Matching Requirements For Unrelated Donors At The SCCA/Fred Hutchinson Allied System**

Acceptable levels of recipient-donor mismatch for research related treatment protocols or standard treatment plans include the following:

Allele-match for HLA-A, B, C, DRB1 and DQB1.

Single allele disparity for HLA-A, B, C, or DRB1 or DQB1

Two allele disparities for HLA-A, B, or C.

Single allele disparity for HLA-DRB1 and/or a single DQB1 antigen or allele disparity.

Single antigen plus single allele disparity for HLA-A, B, or C.

The following levels of patient-donor mismatch should be restricted to research protocols:

Two antigen disparity, either HLA-A plus C or HLA-B plus C.

*Single antigen disparity* for HLA-DRB1 with or without DQB1 allele or antigen disparity *Combined disparity of class I and class II loci*, i.e. disparity for HLA-A, or B, or C, and any additional disparity for DRB1 or DQB1

Donor Exclusion Criteria to be considered for protocols or standard treatment plans include:

**Double locus disparity.** Two disparities are not allowed when they both involve the same locus, i.e., the patient is A\*0101, A\*0201 and the donor is A\*0102 and A\*0205.

**Recipient and donor homozygous at mismatched locus.** Patient and donor pairs homozygous at the mismatched locus are considered a two-locus mismatch, i.e., the patient is A\*0101 and the donor is A\*0201, and this type of mismatch is not allowed.

**Recipient homozygous at mismatched locus.** If the recipient is homozygous at HLA-A, B, or C and the donor is mismatched at that locus, i.e., patient is A\*0101 and donor is A\*0101 and A\*0201, the risk of rejection is increased. Such a donor should be avoided if there is already an appreciable risk of rejection, i.e., in patients with CML/MDS/Severe Aplastic Anemia (SAA) or those receiving reduced conditioning.

#### Relevance of HLA matching for transplantation of unrelated hematopoietic cells:

Human Leukocyte Antigen (HLA) typing of patients and prospective hematopoietic stem cell (HSC) donors is carried out to identify and match for HLA determinants associated with successful HSC transplant outcome. While several preliminary studies (1, 2, 3) suggested the importance of allele level matching in hematopoietic cell transplantation (HCT), recent comprehensive studies confirmed that allele-level typing and matching is necessary to optimize clinical outcome in hematopoietic cell transplantation (4, 5, 6, 7).

The pervasiveness of occult HLA mismatch was shown by Petersdorf, et al in an analysis of 300 CML/CP unrelated donor-recipient pairs matched for HLA-A and B by serologic typing, and matched for the DRB1 alleles.(4) The percent of patient-donor pairs found to be matched at the allele level for all 5 loci (HLA-A, B, C, DRB1, DQB1) was only 47% (n=142). High resolution typing demonstrated previously undetected mismatches in 53% (158), indeed 26% (79) pairs were mismatched for multiple alleles. Mismatch of class I HLA was found at one locus in 55 pairs (18%) and at two or more loci in 35 pairs (12%). A single mismatch of class II HLA was

detected in 24 pairs (8%), whereas 7 pairs (2%) had multiple class II mismatches, and 37 pairs (12%) had multiple mismatches involving both class I and class II. These data show the

## **HLA Matching Requirements For Unrelated Donors At The SCCA/Fred Hutchinson Allied System**

importance of high resolution typing for defining the degree of mismatching between potential unrelated patient-donor pairs.

The degree of HLA mismatch, as well as the locus of mismatch, influence the development of alloimmune reactions and have significant implications for the outcome of HSC transplants. Studies of patient-donor pairs have shown an increased risk for graft failure with multiple mismatches that involve at least one class I allele. The incidence of graft failure was 29% in pairs where the mismatch involved more than one class I allele mismatch and 12% for mismatches involving both class I and class II alleles, compared with 2% or less for pairs with either no mismatch or mismatch confined to a single HLA-A, B, C, DRB1 and DQB1 allele. The risk of developing grades III-IV acute GVHD also has been shown to be influenced by the number and class of mismatched alleles. In studies involving primarily Caucasian patient-donor pairs, the highest risk for severe acute GVHD was observed for multiple mismatches involving both class I and class II alleles (2.0 hazard ratio and p=0.02). Pairs with a single class I mismatch did not have a significant increase in acute GVHD compared with matched recipients, but a single class II mismatch or multiple class I mismatches both appeared to confer a higher (though not significant) hazard of severe GVHD. As results of future studies further define risks of mismatches, particularly in nonCaucasian populations, we may be able to delineate more precisely "low risk" from "high risk" mismatches. Until then, the donor selection process should endeavor to identify the best matched donor within the time allowed by the clinical situation.

#### References:

- 1. Petersdorf EW, Longton GM, Anasetti C, Martin PJ, Mickelson EM, Smith AG, Hansen JA. The significance of HLA-DRB1 matching on clinical outcome after HLA-A, B, DR identical unrelated donor marrow transplantation. Blood 1995: 86:1606-1613.
- 2. Petersdorf EW, Longton GM, Anasetti C, Mickelson EM, Smith AG, Martin PJ, Hansen JA. Definition of HLA-DQ as a transplantation antigen. Proc. Natl. Acad. Sci. USA 1996; 93: 15358.
- 3. Petersdorf EW, Longton GM, Anasetti C, Mickelson EM, McKinney SK, Smith AG, Martin PJ, Hansen JA. Association of HLA-C disparity with graft failure after marrow transplantation from unrelated donors. Blood 1997: 89: 1818
- 4. Petersdorf EW, Gooley TA, Anasetti C, Martin PJ, Smith AG, Mickelson EM, Woolfrey AE, Hansen JA. Optimizing outcome after unrelated marrow transplantation by comprehensive matching of HLA class I and II alleles in the donor and recipient. Blood 1998: 92: 3515.
- 5. Sasazuki T, Juji T, Morishima Y, Kinukawa N, Kashiwabara H, Inoko H, Yoshida T, Kimura A, Akaza T, Kamikawaji N, Kodera Y, Takaku F. Importance of HLA-class I allele matching for clinical outcome after unrelated donor hematopoietic stem cell transplantation. New Engl J Med 1998: 339: 1177.
- 6. Hansen JA, Yamamoto K, Petersdorf E, Sasazuki T. The role of HLA matching in hematopoietic cell transplantation. Reviews in Immunogenetics 1999: 1: 359.
- 7. Petersdorf EW, Hansen JA, Martin PJ, Woolfrey A, Malkki M, Gooley T, Storer B, Mickelson E, Smith A, Anasetti C. Major-histocompatibility-complex class I alleles and antigens in hematopoietic-cell transplantation. New Engl J Med 2001: 345: 1794.

- 8. Bodmer JG, Marsh SGE, Albert ED, Bodmer WF, Bontrop RE, Dupont B, Erlich HA, Hansen JA, Mach B, Mayr WR, Parham P, Petersdorf EW, Sasazuki T, Schreuder GMTh, Strominger JL, Svejgaard A, Terasaki PI. Nomenclature for factors of the HLA system, 1998. Tissue Antigens 1999: 53: 407.
- 9. List of known HLA allele sequences: www.anthonynolan.org.uk/HIG/data.html.
- 10. Information on HLA complex: http://www.ebi.ac.uk/imgt/hla/intro.html.

## **HLA Matching Requirements For Unrelated Donors At The SCCA/Fred Hutchinson Allied System**

#### References continued:

- 11. Little AM and Parham P. Polymorphism and evolution of HLA class I and II genes and molecules. Reviews in Immunogenetics 1999: 1: 105.
- 12. Schreuder GMTh, Hurley CK, Marsh SGE, Lau M, Maiers M, Kollman C, Noreen H. The HLA Dictionary 2001: A summary of HLA-A, B, C, DRB1/3/4/5, DQB1 alleles and their association with serologically defined HLA-A, B, C, DR, and DQ antigens. Tissue Antigens 2001: 58: 109-140.
- 13. Smith A, McKinney S, Menninger O, Warnock S, Hansen JA. Detection of a novel "nonexpression" HLA-B\*15 allele adds to data on the frequency of class I expression variants in a hematopoietic transplant population. Human Immunology 29th Annual ASHI Meeting Abstracts 2003: 64: S159.
- 14. Hurley CK, Baxter Lowe LA, Logan B, Karanes C, Anasetti C, Weisdorf D, Confer DL. National marrow donor program HLA-matching guidelines for unrelated marrow transplants. Biology of Blood and Marrow Transplantation 2003: 9.
- 15. Petersdorf, E.W., Anasetti, C., Martin, P.J., Gooley, T., Radich, J., Malkki, M., Woolfrey, A., Smith, A., Mickelson, E., Hansen, J.A. Limits of HLA mismatching in unrelated hematopoietic cell transplantation. Blood, (in press).

Approved by the Standard Practice Committee January 16, 2002 (Donor Selection Matching Requirements.doc) HLA\_matching\_for\_URD\_selection.doc
Approved by the Medical Advisory Committee (Medical Exec. Comm.) April 9, 2002
Approved by the Clinical Sectional Meeting April 16, 2002
Revised by the Standard Practice Committee June 15, 2005

Minor wording change approved by SPC chairperson March 13, 2006

# APPENDIX P Adapted from COMMON TOXICITY CRITERIA (CTC)

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| ALLERGY/IMMUNOLOGY | | |
| Allergic | Symptomatic bronchospasm, requiring | Anaphylaxis |
| reaction/hypersensitivity | parenteral medication(s), with or | |
| (including drug fever) | without urticaria; allergy-related | |
| | edema/angioedema | |
| Vasculitis | Requiring steroids | Ischemic changes or requiring amputation |
| Allergy/Immunology – Other | Severe | Life-threatening or disabling |
| (Specify,) | | 8 |
| BLOOD/BONE MARROW | | |
| Bone marrow cellularity | | |
| Hemolysis (e.g., immune | Requiring transfusion and/or medical | Catastrophic consequences of hemolysis |
| hemolytic anemia, drug-related | intervention (e.g., steroids) | (e.g., renal failure, hypotension, |
| hemolysis, other) | | bronchospasm, emergency splenectomy) |
| For BMT studies, if specified in | >4 u pRBC in 24 hours | Hemorrhage or hemolysis associated with |
| the protocol. | z + u prede in 2+ nours | life-threatening anemia; medical |
| the protocol. | | intervention required to improve |
| | | hemoglobin |
| For pediatric BMT studies, if | >30mL/kg in 24 hours | nemogloom |
| | /30IIIL/kg III 24 IIOUIS | Hansamhana an hansalania anna siatad seith |
| specified in the protocol. | | Hemorrhage or hemolysis associated with |
| | | life-threatening anemia; medical |
| | | intervention required to improve |
| | Grade | hemoglobin |
| Adverse Event | 3 | 4 |
| Auverse Event | ] 3 | 7 |
| CARDIOVASCULAR (ARRHY | YTHMIA) | |
| Cardiovascular/Arrhythmia | Symptomatic, and requiring | Life-threatening (e.g., arrhythmia |
| -Other (Specify, | treatment of underlying cause | associated with CHF, hypotension, |
| other (Speerly, | deather of anderlying eadse | |
| ) | | syncope, shock) |
| CARDIOVASCULAR (GENER | RAL) | |
| Acute vascular leak | Respiratory compromise or | Life-threatening; requiring pressor |
| syndrome | requiring fluids | support and/or ventilatory/support |
| 5,116101110 | requiring marao | support and/or ventuatory/support |
| Cardiac- | Angina without evidence of | Acute myocardial infarction |
| ischemia/infarction | infarction | |

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| CARDIOVASCULAR (GENER | CARDIOVASCULAR (GENERAL) continued. | |
| | Lave | |
| Cardiac left ventricular | CHF responsive to treatment | Severe or refractory CHF or |
| function | | requiring intubation |
| Cardiac troponin I (cTnI) | Levels consistent with unstable | Levels consistent with myocardial |
| | angina as defined by the | infarction as defined by the |
| | manufacturer | manufacturer |
| Cardiac troponin T (cTnT) | $\geq 0.1 - <0.2 \text{ ng/mL}$ | $\geq 0.2 \text{ ng/mL}$ |
| Hypotension | Requiring therapy and sustained | Shock (associated with acidemia and |
| | medical attention, but resolves | impairing vital organ function due to |
| | without persisting physiologic | tissue hypoperfusion) |
| | consequences | |
| Myocarditis | CHF responsive to treatment | Severe or refractory CHF |
| Pericardial effusion/ | With physiologic consequences | Tamponade (drainage or pericardial |
| pericarditis | | window required) |
| Syncope (fainting) is | - | - |
| graded in the | | |
| NEUROLOGY category. | | |
| Thrombosis/embolism | Deep vein thrombosis, requiring | Embolic event including pulmonary |
| | anticoagulant therapy | embolism |
| Vein/artery operative | | |
| injury is graded as | | |
| Operative injury of | | |
| vein/artery in the | | |
| CARDIOVASCULAR | | |
| (GENEARL) category. | | |
| Cardiovascular/General – | Severe | Life-threatening or disabling |
| Other | | |
| (Specify,) | | |

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| COAGULATION | | |
| DIC (disseminated intravascular coagulation) Also consider Platelets. Note: Must have increased fibrin split products or D-dimer in order to grade as DIC. | Laboratory findings present with <u>no</u> bleeding | Laboratory findings <u>and</u> bleeding |
| Coagulation - Other (Specify,) | Severe | Life-threatening or disabling |
| CONSTITUTIONAL SYMPTOMS | | |
| Weight gain associated with<br>Veno-Occlusive Disease<br>(VOD) for BMT studies, if<br>specified in the protocol.<br>Also consider Ascites Edema,<br>Pleural effusion (non-<br>malignant). | >10% or as ascites | >10% or fluid retention resulting in pulmonary failure |
| DERMATOLOGY/SKIN | | |
| Erythema multiforme (e.g.,<br>Stevens-Johnson syndrome,<br>toxic epidermal necrolysis) | Severe or requiring IV fluids (e.g., generalized rash or painful stomatitis) | Life-threatening (e.g., exfoliative or ulcerating dermatitis or requiring enteral or parenteral nutritional support) |

| APPENDIX P (continued) Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| DERMATOLOGY/SKIN continued | | |
| Rash/desquamation associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol. | Symptomatic generalized erythroderma or symptomatic macular, papular or vesicular eruption, with bullous formation, or desquamation covering ≥50% of body surface area | Generalized exfoliative dermatitis or ulcerative dermatitis or bullous formation |
| GASTROINTESTINAL | | |
| Ascites(none-malignant) | Symptomatic, requiring therapeutic paracentesis | Life-threatening physiologic consequences |
| Also consider Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia, Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia, Melena/GI bleeding, Rectal bleeding/hematochezia, Hypotension. | Abdominal pain, fever, change in bowel habits with ileus or peritoneal signs, and radiographic or biopsy documentation | Perforation or requiring surgery or toxic megacolon |
| Diarrhea associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol. | >1500mL of diarrhea/day | Severe abdominal pain with or without ileus |
| For pediatric BMT studies, if specified in the protocol. | >15mL/kg of diarrhea/day | |
| Also consider Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia, Hemorrhage/bleeding without | | |

| grade 3 or 4 thrombocytopenia,<br>Pain, Dehydration, |
|------------------------------------------------------|
| Hypotension. |

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| GASTROINTESTINAL (continued). | | |
| Duodenal ulcer (requires radiographic or endoscopic documentation) | Uncontrolled by outpatient medical management; requiring hospitalization | Perforation or bleeding, requiring emergency surgery |
| Gastric ulcer<br>(requires radiographic or<br>endoscopic documentation) | Bleeding without perforation,<br>uncontrolled by outpatient<br>medical management; requiring<br>hospitalization or surgery | Perforation or bleeding, requiring emergency surgery |
| Also consider Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia, Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia. | | |
| Gastritis | Uncontrolled by out-patient medical management; requiring hospitalization or surgery | Life-threatening bleeding, requiring emergency surgery |
| Also consider Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia, Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia. | | |
| Pancreatitis Also consider Hypotension. | Abdominal pain with pancreatic enzyme elevation | Complicated by shock (acute circulatory failure) |
| Note: Amylase is graded in the METABOLIC/LABORATOR Y category. | | |

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| GASTROINTESTINAL (continued). | | |
| Mucositis Note: Radiation-related mucositis is graded as Mucositis due to radiation. | Painless erythema, edema, or ulcers preventing swallowing or requiring hydration or parenteral (or enteral) nutritional support | Severe ulceration requiring prophylactic intubation or resulting in documented aspiration pneumonia |
| Typhlitis (inflammation of the cecum) Also consider Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia, Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia, Hypotension, Febrile neutropenia. | Abdominal pain, diarrhea, fever, and radiographic or biopsy documentation | Perforation, bleeding or necrosis or other life-threatening complication requiring surgical intervention (e.g., colostomy) |

## APPENDIX P cont'd

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| HEMORRHAGE | | |
| Notes: Trans | sfusion in this section refers to pRI | 3C infusion. |
| For <u>any</u> bleeding with grade 3 or 4 ple<br>thrombocytopenia. Also consider Platele<br>severit | | sfusion: platelets in addition to grading |
| If the site or type of Hemorrhage/bleeding is listed, also use the grading that incorporates the site of bleeding: NS Hemorrhage/bleeding, Hematuria, Hematemesis, Hemoptysis, Hemorrhage/bleeding with surgery, Melena/lower GI bleeding, Petechiae/purpura (Hemorrhage/bleeding into skin), Rectal bleeding/hematochezia, Vaginal bleeding. | | |
| Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia | Requiring transfusion | Catastrophic bleeding, requiring major non-elective intervention |
| Also consider Platelets, Hemoglobin, Transfusion: platelets, Transfusion: pRBCs, site or type of bleeding. If the site is not listed, grade as Hemorrhage – Other (Specify site,). Note: This adverse event must be | | |
| graded for any bleeding with grade 3 or 4 thrombocytopenia. | | |
| Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia Also consider Platelets, Hemoglobin, | Requiring transfusion | Catastrophic bleeding requiring major non-elective intervention |
| Transfusion: platelets, Transfusion: pRBCs, Hemorrhage – Other (Specify site,). | | |
| Note: Bleeding in the absence of grade 3 or 4 thrombocytopenia is graded here only if the specific site or type of bleeding is not listed elsewhere in the HEMORRHAGE category. Also grade as Other in the HEMORRHAGE category. | | |

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| HEMORRHAGE (continued) | HEMORRHAGE (continued) | |
| CNS hemorrhage/bleeding | Bleeding noted on CT or other scan with no clinical consequences | Hemorrhagic stroke or<br>hemorrhagic vascular event<br>(CVA) with neurologic signs<br>and symptoms |
| Hemoptysis | Requiring transfusion | Catastrophic bleeding, requiring major non-elective intervention |
| Melena/GI bleeding | Requiring transfusion | Catastrophic bleeding, requiring major non-elective intervention |
| Rectal bleeding/hematochezia | Requiring transfusion | Catastrophic bleeding, requiring major non-elective intervention |
| Vaginal bleeding | Requiring transfusion | Catastrophic bleeding, requiring major non-elective intervention |
| Hemorrhage – Other (Specify site,) | Requiring transfusion | Catastrophic bleeding, requiring major non-elective intervention |
| | Grade | |
| Adverse Event | 3 | 4 |
| HEPATIC | | |
| Bilirubin | >3.0 – 10.0 x ULN | >10.0 x ULN |
| Bilirubin associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol. | >6 - <15 mg/100mL | >15 mg/100mL |

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| INFECTION/FEBRILE NEUTROPENIA | | |
| Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection) | Present | Life-threatening sepsis (e.g., septic shock) |
| Infection/Febrile Neutropenia – Other (Specify, ) | Severe | Life-threatening or disabling |

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| NEUROLOGY | | |
| Aphasia, receptive and/or expres category. | sive, is graded under Speech impair | rment in the NEUROLOGY |
| CNS cerebrovascular ischemia | Transient ischemic event or attack (TIA) | Permanent event (e.g., cerebral vascular accident) |
| Leukoencephalopathy associated radiological findings | Severe increase in SAS; severe ventriculomegaly; near total white matter T2 hyperintensities or diffuse low attenuation (CT); focal white matter necrosis (cystic) | Severe increase in SAS; severe ventriculomegaly; diffuse low attenuation with calcification (CT); diffuse white matter necrosis (MRI) |
| Seizure(s) | Seizure(s) in which consciousness is altered | Seizures of any type which are prolonged, repetitive, or difficult to control (e.g., status epilepticus, intractable epilepsy) |
| | Grade | , |
| Adverse Event | 3 | 4 |
| PULMONARY Adult Respiratory Distress | - | Present |
| Syndrome (ARDS) | | |
| Apnea | Present | Requiring intubation |
| Carbon monoxide diffusion capacity (DLCO) FEV1 | >25 - <50% of pretreatment or<br>normal value<br>>25 - <50% of pretreatment or | <25% of pretreatment or normal value <25% of pretreatment or normal |
| Hypoxia | normal value Decreased O2 saturation at rest, requiring supplemental oxygen | value Decreased O2 saturation, requiring pressure support (CPAP) or assisted ventilation |

| Grade | | |
|---|---|---|
| Adverse Event | 3 | 4 |
| RENAL/GENITOURINARY | | |
| Creatinine | >3.0- 6.0 x ULN | >6.0 x ULN |
| Note: Adjust to age-appropriate | | |
| levels for pediatric patients. | | |
| Renal failure | Requiring dialysis, but | Requiring dialysis and |
| | reversible | irreversible |
| SECONDARY MALIGNANCY | | |
| Secondary Malignancy – Other | - | Present |
| (Specify type,) | | |
| excludes metastasis from initial | | |
| primary | | |

APPENDIX Q
The Hematopoietic Cell Transplant-Comorbidity Index (HCT-CI) 9/7/10

## Assign scores appropriately if the patient has any of these comorbidities

| Patient | (name), | UPN | I | Date |
|---------|---------|-----|---|------|
| | ( // | | | |

| Comorbidities | Definitions | HCT-CI | Actual Lab |
|---|---|---|---|
| <b>Comorbidities</b> | Definitions | scores | Values/Comments |
| Arrhythmia | ventricular arrhythmias requiring treatment in the patient's past history | | |
| Cardiac | Coronary artery disease†, congestive heart failure, myocardial infarction <i>in patient's past history</i> or EF of ≤50% at time of HCT | 1 | |
| Inflammatory bowel disease | Crohn's disease or ulcerative colitis requiring treatment in the patient's past history | 1 | |
| Diabetes | Requiring treatment with insulin or oral hypoglycemic, but not diet alone, at time of HCT | 1 | |
| Cerebro-vascular disease | Transient ischemic attack or cerebro-vascular accident in patient's past history | 1 | |
| Psychiatric disturbance | Depression/anxiety requiring psychiatric consult or treatment at time of HCT | 1 | |
| Hepatic – mild | Chronic hepatitis, Bilirubin >ULN- 1.5 X ULN, or AST/ALT >ULN-2.5XULN at time of HCT | 1 | |
| Obesity | Patients with a BMI of >35 for adults or with BMI-for-age percentile of ≥ 95th percentile for children <i>at time of HCT</i> | 1 | |
| Infection | nfection Documented infection or fever of unknown etiology requiring anti-microbial treatment before, during and after the start of conditioning regimen | | |
| Rheumatologic SLE, RA, polymyositis, mixed CTD, polymyalgia rheumatica <i>in patient's past history</i> | | 2 | |
| Peptic ulcer | Requiring treatment in patient's past history | 2 | |
| Renal | Serum creatinine >2 mg/dl, on dialysis, or prior renal transplantation <i>at time of HCT</i> | 2 | |
| Moderate pulmonary | Moderate pulmonary DLco and/or FEV <sub>1</sub> >65%-80% or Dyspnea on slight activity at time of HCT | | |
| Prior solid tumor | Treated at any time point in the patient's past history, excluding non-melanoma skin cancer | 3 | |
| Heart valve disease | At time of HCT excluding mitral valve prolapse | 3 | |
| Severe pulmonary | DLco and/or FEV <sub>1</sub> $\leq$ 65% or<br>Dyspnea at rest or requiring oxygen <i>at time of HCT</i> | 3 | |
| Moderate/severe Liver cirrhosis, Bilirubin >1.5 X ULN, or AST/ALT epatic >2.5XULN at time of HCT | | 3 | |
| Please provide (KPS): | Karnofsky Performance Score =% | Total | Signature of Provider: |

†One or more vessel-coronary artery stenosis, requiring medical treatment, stent, or bypass graft.

EF indicates ejection fraction; ULN, upper limit of normal; SLE, systemic lupus erythmatosis; RA, rheumatoid arthritis; CTD, connective tissue disease; DLco, diffusion capacity of carbon monoxide; FEV<sub>1</sub>, forced expiratory volume in one second; AST, aspartate aminotransferase; ALT, alanine aminotransferase.

EF indicates ejection fraction; ULN, upper limit of normal; SLE, systemic lupus erythmatosis; RA, rheumatoid arthritis; CTD, connective tissue disease; DLco, diffusion capacity of carbon monoxide; FEV<sub>1</sub>, forced expiratory volume in one second; AST, aspartate aminotransferase; ALT, alanine aminotransferase.

## APPENDIX R STAGING OF CLL

## **Binet staging**

| Binet stage | Lymph node areas | Hemoglobin Platelet | | Survival |
|---|---|---|---|---|
| | | <11 g/dl | $< 100 \times 10^{9}/L$ | (years) |
| A | < 3 | No | No | 12 |
| В | 3 or > | No | No | 7 |
| С | ± | Yes (or low platelet) | Yes (or low hemoglobin) | 2 |
| | | (or low platelet) | (or low hemoglobin) | |

**Modified Rai staging** 

| | TIOU I LUI SUUGII | <b>B</b> | | | | | |
|---|---|---|---|---|---|---|---|
| Rai | Risk category | Lymphocytosis | Lymph node | Spleen/liver | Hemoglobin | Platelet | Survival |
| stage | | | enlargement | enlargement | < 11 g/dl | $<100\times10^{9}/L$ | (years) |
| 0 | Low | Yes | No | No | No | No | > 10 |
| I | Intermediate | Yes | Yes | No | No | No | > 7 |
| II | Intermediate | Yes | <u>±</u> | $\pm$ | No | No | > 7 |
| III | High | Yes | <u>±</u> | <u>±</u> | Yes | No | 1.5 |
| IV | High | Yes | ± | <u>±</u> | ± | Yes | 1.5 |

## Appendix S

Weight / Adjusted Body Weight for Drug Dosing



Weight for Drug Dosing

#### **APPENDIX T**

#### COORDINATING CENTER FUNCTIONS

Outside Center – PI Communication in Hematologic Malignancies

### I. Study Management, data analysis, and Data and Safety Monitoring

- a. Study Management:
  - i. Each local PI is responsible for selection, training and oversight of local study coordinators
  - ii. The Coordinating Center registers subjects on the study and assigns study IDs
  - iii. One copy of the research data is retained by the site. Another data set (identified only by study IDs) is transmitted to the Coordinating Center to create the master data file. All data are kept in locked areas and password protected databases accessible only to study staff
  - iv. The quality of data is monitored in an ongoing fashion with the study team and corrective action plans instituted as necessary

#### b. Data Analysis:

- i. Study staff review data for completeness as it is submitted by the sites
- ii. The study statistician is responsible for data cleaning and the conduct of analyses as outlined in the protocol and grant
- c. Data Safety and Monitoring:
  - i. The trial coordinators at collaborating centers or the local PIs will fax an official report of an SAE (as defined by the protocol) to the Coordinating Center within ten days
  - ii. The SAE report is reviewed by the Overall PI. If the SAE meets the FHCRC criteria for reporting then an official signed report is submitted to the IRB
  - iii. An independent DSMB will meet at six-month intervals and all outcome data is reviewed including all adverse events and SAEs reported to the Coordinating Center along with those officially reported to the IRB
  - iv. A report from the DSMB is submitted to the IRB as well as the trial coordinators/local PIs participating in the protocol

## II. Protocol and informed consent document management

- a. A master protocol is maintained by the Coordinating Center and distributed to the sites for customization and local IRB review
- b. All protocol and consent modifications initiated by the Coordinating Center are sent to the Collaborating Sites following approval by the Coordinating Center IRB, for review and approval by the local IRB
- c. Changes required by local IRBs are reviewed by the Coordinating Center and approved prior to implementation at local sites

## III. Assurance of local IRB OHRP-approved assurance

- a. Each site provides their OHRP assurance number and evidence of IRB certification
- b. Study staff monitor maintenance of institutional assurance and IRB certification

#### IV. Assurance of local IRB approvals

- a. The Coordinating Center maintains copies of the most current collaborating site Consent Forms and IRB approval documentation
- b. No site may enroll subjects until the Coordinating Center has received confirmation of local IRB approval
- Each site is responsible for preparation and submission of their continuing reviews.
   Any changes to the protocol or consent form will be communicated to the Coordinating Center
- d. Sites are required to have active IRB approvals to participate in any study related activities

## V. Any substantive modification by the Collaborating Institution related to risks or alternative procedures is appropriately justified

a. The Coordinating Center reviews any modifications to consent forms to ensure that site consents do not delete or change the basic or additional elements or alternatives required in the sample consent form

## VI. Informed consent is obtained from each subject in compliance with HHS regulations

- a. Subjects must provide written informed consent prior to study participation
- b. The Coordinating Center verifies eligibility and signed consent prior to assigning a study ID number